# N-DOSE: A randomized, double blind, dose optimization trial of nicotinamide riboside in Parkinson's disease.

**Protocol Identification Number:** v3.1, 5<sup>th</sup> June 2025

SPONSOR: Haukeland University Hospital

Address: Jonas Lies 65

Tel: 55975000

PRINCIPAL INVESTIGATOR (PI): Charalampos Tzoulis

Tel: 55975061

E-mail: <a href="mailto:charalampos.tzoulis@helse-bergen.no">charalampos.tzoulis@helse-bergen.no</a>

PROTOCOL VERSION NO. 3.1, -June 2025

# **CONTACT DETAILS**

| Sponsor: | Haukeland University Hospital Address: Jonas Lies 65 Tel: 55975000 |
|---|---|
| Study Director | Charalampos Tzoulis E-mail: <a href="mailto:charalampos.tzoulis@helse-bergen.no">charalampos.tzoulis@helse-bergen.no</a> |
| Coordinating Investigator Principal investigator (at each participating site or if single site study): | Haakon Berven cand.med Haukeland university hospital Tel: 48495197 E-mail: haakonberven@outlook.com Haukeland university hospital Charalampos Tzoulis E-mail: charalampos.tzoulis@helse-bergen.no |
| Participating Departments: | Haukeland university hospital, Department of Neurology Department of Clinical Medicine, University of Bergen |
| Monitor: | Section of Innovation and Research Haukeland University Hospital, department of Research and Development |

# **SIGNATURE PAGE**

| Title | N-DOSE: A randomized, double blind, dose optimization trial on nicotinamide riboside in Parkinson's disease. | of |
|---|---|---|
| Protocol ID no: | | |

I hereby declare that I will conduct the study in compliance with the Protocol, ICH GCP and the applicable regulatory requirements:

To be signed by sponsor's representative, Coordinating Investigator, Principal Investigator, statistician etc. This section and table above should be completed as appropriate for the type of study conducted and the parties involved.

| Name | Title | Role | Signature | Date |
|---------------|------------------|------------------------|-----------|------|
| Torhild Næss | Neurology clinic | Sponsor | | |
| Vedeler | Director | representative | | |
| Charalampos | Professor of | Principal Investigator | | |
| Tzoulis | Neurology | / Study Director | | |
| Haakon Berven | Neurology | Coordinating | | |
| | resident | Investigator | | |

# **PROTOCOL SYNOPSIS**

# N-DOSE: A randomized, double blind, dose optimization trial of nicotinamide riboside in Parkinson's disease.

Sponsor: Haukeland University Hospital

Phase and study type: Phase II, Dose-Optimization study

Investigational Product (IP) (including active comparator and placebo):

Nicotinamide Riboside, Placebo

Centers: Haukeland University Hospital

Study Period: Estimated date of first patient enrolled: 28.11.2022

Anticipated recruitment period: 01.10.2022 - 20.01.2025.

Estimated date of last patient completed: 22.04.2025.

Treatment Duration: 12 weeks

#### **Objectives and endpoints**

| Objective | | Endpoint |
|---|---|---|
| Primary | To compare the effect of orally administered nicotinamide riboside (NR), escalated to 1500 mg twice per day (3000 mg/day) in the dose-escalation group (DE-group) - versus stable dosing of 500 mg twice per day (1000 mg/day) in the dose-stable group (DS-group) on cerebral NAD-levels, at week 12. | Change in cerebral NAD/ATP-α ratio measured by 31 Phosphorus magnetic resonance spectroscopy (31P-MRS) in the posterior brain (encompassing the occipital, parietooccipital and posterior parts of the temporal cortex). |
| Secondary | To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in cerebral NAD levels from baseline to weeks 4, 8 and 12. | Change in cerebral NAD/ATP- $\alpha$ ratio measured by 31 Phosphorus magnetic resonance spectroscopy (31P-MRS) in the posterior brain (encompassing the occipital, parietooccipital and posterior parts of the temporal cortex). |
| | To compare the effectiveness of orally administered nicotinamide riboside (NR) 1500 mg twice per day versus 500 mg twice per day in augmenting the NAD-metabolome in the central nervous system (CNS) at week 12. | Change in the cerebrospinal fluid (CSF) levels of NAD or other metabolites of the NAD metabolome*, measured by LC-MS. |

| Exploratory | Neuroimaging | |
|---|---|---|
| , | To compare the effect of orally administered NR | Change in NRRP expression, measured by FDG- |
| | in the DE-group versus DS-group on the NR | PET. |
| | related metabolic pattern (NRRP) expression at | |
| | week 12. | |
| | To assess the dose-response relationship | |
| | between NR dose (1000 mg, 2000 mg, 3000 mg | Change in NRRP expression, measured by FDG- |
| | per day) and changes in NRRP expression from | PET. |
| | baseline to weeks 4, 8 and 12. | |
| | To compare the effect of orally administered NR | Change in PDRP expression, measured by FDG- |
| | DE-group versus DS-group on the PD-related | PET. |
| | pattern (PDRP) expression at week 12. | FLI. |
| | To assess the dose-response relationship | |
| | between NR dose (1000 mg, 2000 mg, 3000 mg | Change in PDRP expression, measured by FDG- |
| | per day) and changes in PDRP expression from | PET. |
| | baseline to weeks 4, 8 and 12. | |
| | Metabolism & molecular markers | |
| | To compare the effect of orally administered NR | Change in levels of NAD metabolites in blood, |
| | in the DE-group versus DS-group on the NAD | urine and CSF, measured by HPLC-MS and/or the |
| | metabolome* in the blood, urine and central | NADMed method. |
| | nervous system (CNS) at week 12. | |
| | To assess the dose-response relationship | |
| | between NR dose (1000 mg, 2000 mg, 3000 mg | Change in levels of NAD metabolites in blood and |
| | per day) and changes in the NAD metabolome* in | urine, measured by HPLC-MS and/or the NADMed |
| | blood and urine from baseline to weeks 4, 8 and | method. |
| | 12. | |
| | To compare the effect of orally administered NR | Change in inflammatory cytokines in serum and |
| | in the DE-group versus DS-group on serum and | CSF, measured by ELISA. |
| | CSF inflammatory markers at week 12. | |
| | To assess the dose-response relationship | Change in inflammatory sytalines in serum |
| | between NR dose (1000 mg, 2000 mg, 3000 mg | Change in inflammatory cytokines in serum, |
| | per day) and changes in serum inflammatory markers from baseline to weeks 4, 8 and 12. | measured by ELISA. |
| | Clinical – motor & non motor symptom severity, c | nuality of life |
| | To compare the effect of orally administered NR | quanty of me |
| | in the DE-group versus DS-group on clinical | Change in the total MDS-UPDRS score in the ON- |
| | severity of PD symptoms at week 12. | medication state. |
| | To assess the dose-response relationship | |
| | between NR dose (1000 mg, 2000 mg, 3000 mg | Change in total MDS-UPDRS score in the ON- |
| | per day) and change in clinical severity of PD | medication state. |
| | symptoms from baseline to weeks 4, 8 and 12. | |
| | To compare the effect of orally administered NR | |
| | in the DE-group versus DS-group on severity of | Change in the MDS-UPDRS part I score in the ON- |
| | non-motor symptoms of daily living in PD at week | medication state. |
| | 12. | |
| | To assess the dose-response relationship | |
| | between NR dose (1000 mg, 2000 mg, 3000 mg | |
| | per day) and change in severity of non-motor | Change in the MDS-UPDRS part I score in the ON- |
| | symptoms of daily living in PD from baseline to | medication state. |
| | weeks 4, 8 and 12. | |
| | To compare the effect of orally administered NR | Change in the MDS-UPDRS part II score in the ON- |
| | • | |

| in the DE-group versus DS-group on severity of motor aspects of experiences of daily living in PD | medication state. |
|---|---|
| at week 12. | |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | |
| per day) and changes in severity of motor aspects | Change in the MDS-UPDRS part II score in the ON- |
| of experiences of daily living in PD from baseline | medication state. |
| to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | Change in the MDS-UPDRS part III score in the ON- |
| in the DE-group versus DS-group on severity of PD | medication state. |
| motor symptoms at week 12. | medication state. |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in the MDS-UPDRS part III score in the ON- |
| per day) and changes in severity of PD motor | medication state. |
| symptoms from baseline to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | Change in the MDS-UPDRS part IV score in the |
| in the DE-group versus DS-group on severity PD | ON-medication state. |
| motor complications at week 12. | |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in the MDS-UPDRS part IV score in the |
| per day) and changes in severity of PD motor | ON-medication state. |
| complications from baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on clinical | Change in the total MDS-NMS score. |
| severity of PD non-motor symptoms at week 12. | Change in the total MD3-MM3 Score. |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | |
| per day) and changes in clinical severity of PD | Change in the total MDS-NMS score. |
| non-motor symptoms from baseline to weeks 4, 8 | |
| and 12. | |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on clinical | Change in the modified CIDS DD coors |
| severity of gastrointestinal non-motor | Change in the modified GIDS-PD score. |
| dysfunction in PD at week 12. | |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | |
| per day) and changes in clinical severity of | Change in the modified GIDS-PD score. |
| gastrointestinal non-motor dysfunction in PD | |
| from baseline to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on cognition at | Change in the MoCA score. |
| week 12. | |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in cognition from baseline | Change in the MoCA score. |
| to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on quality of life | Change in the EQ-5D-5L score. |
| in PD at week 12. | 5 - 1 - |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in the EQ-5D-5L score. |
| ( 5, 111 6, 1110 116 | |

| per day) and changes in quality of life in PD from | |
|---|---|
| baseline to weeks 4, 8 and 12. | |
| | endpoints (may be reported in follow-up or |
| secondary publications). | |
| To compare the effect of orally administered NR | Change in gene expression, measured by RNA |
| in the DE-group versus DS-group on gene | sequencing (RNAseq). |
| expression at week 12. | 3.4.5.5.00 |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in gene expression, measured by RNA |
| per day) and changes in gene expression from | sequencing (RNAseq). |
| baseline to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on protein | Change in protein levels, measured by LC-MS. |
| expression at week 12. | |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in protein levels, measured by LC-MS. |
| per day) and changes in protein expression from | |
| baseline to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | Change in inflammatory cytokines in serum and |
| in the DE-group versus DS-group on serum and | CSF, measured by ELISA. |
| CSF inflammatory markers at week 12. | · |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in inflammatory cytokines in serum, |
| per day) and changes in serum inflammatory | measured by ELISA. |
| markers from baseline to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | Change in histone panacetylation, measured by |
| in the DE-group versus DS-group on histone | immunoblotting. |
| acetylation in PD at week 12. | |
| To assess the dose-response relationship | Change in history representation reserved by |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in histone panacetylation, measured by |
| per day) and changes in histone acetylation in PD from baseline to weeks 4, 8 and 12. | immunoblotting. |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on H3K27 and | Changes in levels of H3K27 and H4K16 |
| H4K16 histone acetylation in PD at week 12. | acetylation, measured by immunoblotting. |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg | |
| per day) and changes in on H3K27 and H4K16 | Changes in levels of H3K27 and H4K16 |
| histone acetylation in PD from baseline to weeks | acetylation, measured by immunoblotting. |
| 4, 8 and 12. | |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on the genomic | Change in the genomic distribution of H3K27 and |
| distribution of H3K27 and H4K16 histone | H4K16 acetylation, measured by chromatin |
| acetylation in PD at week 12. | immunoprecipitation sequencing (ChIPseq). |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in the genomic distribution of H3K27 and |
| per day) and changes in the genomic distribution | H4K16 acetylation, measured by chromatin |
| of H3K27 and H4K16 histone acetylation in PD | immunoprecipitation sequencing (ChIPseq). |
| from baseline to weeks 4, 8 and 12. | minumoprecipitation sequencing (citil seq). |
| To compare the effect of orally administered NR | Change in folate and one-carbon metabolites in |
| in the DE-group versus DS-group on folate and | blood and CSF, measured by HPLC-MS. |
| and 22 or one reliand to broad our locate and | and and act, maddica by the Lo 1910. |

| | one-carbon metabolism in PD at week 12. | |
|---|---|---|
| | To assess the dose-response relationship | |
| | between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in folate and one-carbon metabolism in PD from baseline to weeks 4, 8 and 12. | Change in folate and one-carbon metabolites in blood, measured by HPLC-MS. |
| | To compare the effect of orally administered NR in the DE-group versus DS-group on methyl donors in PD at week 12. | Change in methyl-donors (e.g., SAM), measured by HPLC-MS, in the blood and/or CSF. |
| | To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in methyl-donors in PD from baseline to weeks 4, 8 and 12. | Change in methyl-donors (e.g., SAM), measured by HPLC-MS, in the blood. |
| | To compare the effect of orally administered NR in the DE-group versus DS-group on DNA methylation at week 12. | Change in level and genomic distribution of DNA methylation, measured by Illumina Infinium MethylationEpic kit. |
| | To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in methyl-donors in PD from baseline to weeks 4, 8 and 12. | Change in level and genomic distribution of DNA methylation, measured by Illumina Infinium MethylationEpic kit. |
| | To compare the effect of orally administered NR in the DE-group versus DS-group on synthesis of neurotransmitters in PD at week 12. | Change in neurotransmitters in CSF, measured by HPLC-MS. |
| | Determine whether NR-therapy affects the gut microbiome in a dose-responsive manner at week 12. | Change in gut microbiome composition, measured by metagenomics in fecal samples. |
| | To compare the effect of orally administered NR in the DE-group versus DS-group on the gut metabolome at week 12. | Change in fecal metabolomics, measured by LC-MS in fecal samples. |
| | To compare the effect of orally administered NR in the DE-group versus DS-group on the sense of smell at week 12. | Change in sense of smell, measured by B-SIT score. |
| Safety | To determine the safety and tolerability of NR at a dose of 1000 mg, 2000 mg, and 3000 mg per day in PD. | Number and severity of adverse events from baseline to week 12 across treatment groups and NR dose levels. |

\*The NAD metabolome is comprised of: Nicotinamide adenine dinucleotide oxidized (NAD+), Nicotinamide adenine dinucleotide reduced (NADH), NAD+/NADH ratio, total NAD (sum of NAD+ and NADH), Nicotinamide adenine dinucleotide phosphate oxidized (NADP+), Nicotinamide adenine dinucleotide phosphate reduced (NADPH), NADP+/NADPH ratio, total NADP (sum of NADP+ and NADPH, 1-methyl nicotinamide (Me-Nam), nicotinic acid-adenine dinucleotide (NAAD), N1-methyl-2-pyridone-5-carboxamide (Me-2-PY), Nicotinamide (Nam), Nicotinamide N-oxide (Nam N-oxide), ADP-ribose (ADPR), Nicotinic acid riboside (NAR), Nicotinamide riboside (NR), Nicotinamide mononucleotide (NMN), Nicotinic acid (NA).

Study Design: Single-center, double-blinded, randomized, placebo controlled, dose-optimization

#### Inclusion Criteria:

- Clinically established diagnosis of idiopathic PD according to the MDS criteria.
- 123I-Ioflupane dopamine transporter imaging (DAT-scan) or 18-F-FDOPA positron emission tomography imaging (18F-FDOPA PET) confirming nigrostriatal degeneration.
- Hoehn and Yahr score < 4 at enrollment.
- Age ≥ 40 years at the time of enrollment.
- Able to undergo lumbar punction.
- Able to undergo MRI

#### **Exclusion Criteria:**

- Dementia or other neurodegenerative disorder at baseline visit.
- Diagnosed with atypical parkinsonism (PSP, MSA, CBD) or vascular parkinsonism.
- Any psychiatric disorder that would interfere with compliance in the study.
- Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.
- Use of high dose vitamin B3 supplementation within 30 days of enrollment

Sample Size:

80 patients (20 in placebo group, 60 in treatment groups)

Efficacy

Primary endpoint: Cerebral NAD levels as measured by <sup>31</sup>P-MRS (see details under

Assessments: Endpoints).

Safety

Biochemistry: Routine blood analysis (see Lab-manual).

Assessments:

Vital signs: pulse, blood pressure.

Registration of adverse events.

# **TABLE OF CONTENTS**

| C | CONTA | CT DETAILS | 2 |
|---|---|---|---|
| S | GNAT | TURE PAGE | 3 |
| P | ROTO | COL SYNOPSIS | 4 |
| T | ABLE | OF CONTENTS | 10 |
| 1 | IN | TRODUCTION | 15 |
| | 1.1 | Background – Disease | 15 |
| | 1.1<br>1.2 | .1 Parkinson's disease (PD) is a major societal challenge | |
| | 1.2<br>1.2<br>1.3 | 1 17 1 17 | 15 |
| | 1.3<br>1.3<br>1.4 | .1 Preclinical evidence for NR-therapy | 16<br>16 |
| 2 | | UDY OBJECTIVES AND RELATED ENDPOINTS | |
| | 2.1 | Primary Endpoint Measure | |
| | 2.2 | Secondary Endpoint Measure | 25 |
| | 2.3 | Exploratory Endpoint Measures | 26 |
| 3 | OV | /ERALL STUDY DESIGN | 28 |
| | 3.1 | Study design | 28 |
| 4 | ST | UDY POPULATION | 29 |
| | 4.1 | Selection of Study Population | 29 |
| | 4.2 | Number of Patients | 29 |
| | 4.3 | Inclusion Criteria | 29 |
| | 4.4 | Exclusion Criteria | 29 |
| 5 | TR | EATMENT | 30 |
| | 5.1 | Drug Identity, Supply and Storage | 30 |
| | 5.2 | Dosage and Drug Administration | 30 |
| | 5.3 | Duration of Therapy | 30 |
| | 5.4 | Dopaminergic therapy during Screening and Treatment period | 31 |
| | 5.5 | Concomitant Medication | 31 |
| | 5.6 | Subject Compliance | 31 |
| | 5.7 | Drug Accountability | 32 |
| | 5.8 | Drug Labeling | 32 |
| | 5.9 | Subject Numbering | 32 |
| 6 | ST | UDY PROCEDURES | 32 |
| | 6.1 | Flow Chart | 32 |

| 6.2 | By Visit | 34 |
|---|---|---|
| 6 | S.2.1 Screening Visits/ Before start of Investigational Product (IP) | |
| _ | 5.2.2 Baseline/Week 0 | |
| | 5.2.3 During treatment (visits 2-4) | |
| 6.3 | | |
| 6.4 | Procedures for Discontinuation | 36 |
| 6 | S.4.1 Patient Discontinuation | 36 |
| _ | S.4.2 Trial Discontinuation | |
| | ASSESSMENTS | |
| 7.1 | , | |
| 7.2 | | |
| 7.3 | , | |
| 7.4 | Imaging studies | 38 |
| 7.5 | Molecular analyses | 39 |
| 8 9 | SAFETY MONITORING AND REPORTING | 39 |
| 8.1 | Definitions | 39 |
| | 3.1.1 Adverse Event (AE) | |
| | 3.1.2 Serious Adverse Event (SAE) | |
| 8.2 | , 3 | |
| 8.3 | • | |
| 8.4 | | |
| 8.5 | 3.4.1 AEs and SAEs Clinical Study Report | |
| | DATA MANAGEMENT AND MONITORING | |
| 9.1 | Electronic - Case Report Forms (e-CRFs) | |
| 9.2 | | |
| 9.2 | | |
| 9.4 | ů . | |
| | STATISTICAL METHODS AND DATA ANALYSIS | |
| 10.1 | ' | |
| 10.2 | | |
| | ndomization is done by e-CRF upon enrollment to the study. Participants will be randomized into | • |
| | acebo, NR 1000 mg for the duration of the study, NR dose escalation group) | |
| 10.3 | | |
| 10.4 | • | |
| 10.5 | • | |
| 11 \$ | STUDY MANAGEMENT | |
| 11.1 | 1 Investigator Delegation Procedure | 47 |
| 11.2 | 2 Protocol Adherence | 47 |

| 11 | .3 | Study Amendments | 47 |
|---|---|---|---|
| 11 | .4 | Audit and Inspections | 47 |
| 12 | ETH | IICAL AND REGULATORY REQUIREMENTS | 48 |
| 12 | .1 E | Ethics Committee Approval | 48 |
| 12 | .2 ( | Other Regulatory Approvals | 48 |
| 12 | .3 I | Informed Consent Procedure | 48 |
| 12 | .4 \$ | Subject Identification | 48 |
| 13 | TRIA | AL SPONSORSHIP AND FINANCING | 48 |
| 14 | TRIA | AL INSURANCE | 48 |
| 15 | PUB | BLICATION POLICY | 49 |
| 16 | REF | ERENCES | 49 |
| 17 | LIST | T OF APPENDICES | 53 |
| STA | NDAI | RD OPERATING PROCEDURE (SOP) FOR SAMPLING AND PREPARATION OF BIOLOGICAL | . MATERIAL |
| (LAE | 3 MA | NUAL) | 54 |
| 1 | GEN | NERAL INFORMATION | 55 |
| 2 | HEN | MATOLOGY, BIOCHEMISTRY, HORMONE, SEROLOGY AND SAFETY LABORATORY PARAMI | ETERS 56 |
| | 2.1.1 | | |
| 3 | | MPLING FOR BIOBANK AND RESEARCH | |
| 3.1 | | Mandatory research and biobank samples | |
| | 3.1.1<br>3.1.2 | | |
| | 3.1.2<br>3.1.3 | · | |
| ; | 3.1.4 | Whole blood for Serum | 58 |
| | 3.1.5 | | |
| | 3.1.6<br>3 1 7 | 6 Cerebrospinal fluid (CSF) | 58<br>58 |
| ` | 3.1.8 | 1 0000 | |
| 4 | | MPLE PROCESSING AND STORAGE | |
| 4.1 | 1 \ | Whole blood (EDTA): standard | 59 |
| 4.2 | 2 ١ | Whole blood (EDTA): snap-frozen | 60 |
| 4.3 | | RNA PAXgene tubes | |
| 4.4 | | Serum for biobanking | |
| 4.5 | 5 F | Platelet isolation and cryopreservation for mitochondrial research | 63 |
| 4.6 | 6 ( | Collection, of cerebrospinal fluid | 63 |
| | 4.6.1 | - I | |
| 4.7 | | 2 Processing and storage of cerebrospinal fluid Fecal sample for biobanking | |
| 4.7 | | Fecal sample for biobanking | |
| 4.6<br><b>5</b> | | VTACT PERSONS | |
| | | Helse Bergen | |
| 5.3 | | - | |
| | 5.1.1 | Biobank Haukeland | ნ8 |

| 5.1.2 | Laboratory Clinic | 68 |
|----------|----------------------------|-----|
| | Department of Neurology | |
| APPENDI | X B | 69 |
| MRI AND | FDG-PET – PROTOCOL, N-DOSE | 69 |
| APPENDI | X C | 73 |
| CLINICAL | RATING SCALES | 73 |
| 1 GEN | IERAL INFORMATION | 73 |
| 2 MRS | S-UPDRS | 74 |
| 3 MDS | S-NMS | 107 |
| 4 MOD | DIFIED GIDS-PD | 119 |
| | A | |
| 6 EQ-5 | 5D-EL | 136 |

# **List of Abbreviations and Definitions of Terms**

| Abbreviation or special term | Explanation |
|---|---|
| AE | Adverse Event |
| ChIPseq | Chromatin immunoprecipitation sequencing |
| CNS | Central Nervous System |
| CRF | Case Report Form (electronic/paper) |
| CSF | Cerebrospinal fluid |
| SAM | S-denosyl methionine |
| DS-group | Dose-stable group |
| DE-group | Dose-escalation group |
| CSA | Clinical Study Agreement |
| СТС | Common Toxicity Criteria |
| CTCAE | Common Terminology Criteria for Adverse Event |
| DAE | Discontinuation due to Adverse Event |
| EC | Ethics Committee, synonymous to Institutional Review Board (IRB) and |
| | Independent Ethics Committee (IEC) |
| EQ-5D-5L | A standardized measure of health-related quality of life |
| GCP | Good Clinical Practice |
| GIDS-PD | Gastrointestinal Dysfunction Scale for Parkinson's Disease |
| HPLC-MS | High pressure liquid chromatography-mass spectrometry |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IP | Investigational Product (includes active comparator and placebo) |
| IND | Investigational New Drug |
| LC-MS | Liquid chromatography-mass spectrometry |
| HPLC-MS | High performance liquid chromatography-mass spectrometry |
| MDS-CDC | Movement Disorders Society – Clinical Diagnosis Criteria for PD |
| MDS-NMS | Movement Disorders Society – Non-Motor rating Scale |
| MDS-UPDRS | Movement Disorders Society – Unified Parkinson's Disease Rating Scale |
| MDS-NMS | Movement Disorders Society – Non-Motor rating Scale |

| MoCA | Montreal Cognitive Assessment |
|---|---|
| MRS-responder | An individual susceptible to NR-induced increase in cerebral NAD levels, |
| | detectable by <sup>31</sup> P-MRS |
| MRS-non-responder | An individual showing no NR-induced increase in cerebral NAD levels |
| | detectable by <sup>31</sup> P-MRS |
| NAD | Nicotinamide adenine dinucleotide |
| NR | Nicotinamide Riboside |
| NRRP | NR-related metabolic pattern |
| PDRD | Parkinson's disease related pattern |
| OBD | Optimal biological dose |
| PBMC | Peripheral Blood Mononuclear Cells |
| PD | Parkinson's Disease |
| PDRP | Parkinson's Disease-Related Pattern |
| SAE | Serious Adverse Event |
| SOP | Standard Operating Procedure |

# 1 INTRODUCTION

# 1.1 Background – Disease

#### 1.1.1 Parkinson's disease (PD) is a major societal challenge

PD affects 1-2% of the population above the age of 65, and is a major cause of death and disability with a devastating global socioeconomic impact<sup>1,2</sup>. In Europe alone, PD affects an estimated 1.2 million people and has a cost of €14 billion per year<sup>3</sup>. Current treatments for PD are purely symptomatic and have no impact on disease progression. As a result, patients confront a future of progressive disability, early institutionalization, and premature death. Since demographic studies show that patient numbers will continue to grow, effectively doubling by 2040, our failure to make any significant impact to halt or delay disease progression means that PD is now a **major challenge** to health care and society.

# 1.2 Background - Therapeutic Information

#### 1.2.1 NAD-replenishment therapy shows promise as neuroprotective therapy for PD

Increasing evidence supports that boosting cellular levels of nicotinamide adenine dinucleotide (NAD) confers neuroprotective effects in both healthy aging and neurodegeneration<sup>4</sup>. NAD, which constantly shuttles between its oxidized (NAD<sup>+</sup>) and reduced (NADH) state, is an essential cofactor for metabolic redox reactions, including mitochondrial respiration. Furthermore, NAD<sup>+</sup> is substrate to vital signaling reactions involved in DNA repair, histone- and other protein deacylation, and second messenger generation<sup>5</sup>. These reactions consume NAD<sup>+</sup> at high rates, requiring constant replenishment via NAD biosynthesis. NAD levels have been shown to decline with age and this is believed to contribute to agerelated diseases<sup>5,6</sup>. Increasing the NAD replenishment rate (e.g., via supplementation of precursors), and/or enhancing the NAD<sup>+</sup>/NADH ratio (e.g., via caloric restriction) have shown beneficial effects on lifeand healthspan in multiple model systems, and evidence of neuroprotection in models of neurodegeneration and other age-related diseases<sup>5-7</sup>. Enhancing NAD replenishment could potentially help ameliorate several major processes implicated in the pathogenesis of PD, including mitochondrial respiratory dysfunction<sup>8-10</sup>, neuroinflammation<sup>11</sup>, epigenomic dysregulation<sup>12,13</sup> and increased neuronal DNA damage<sup>14</sup>.

NAD can be replenished via supplementation of nicotinamide riboside (NR), a vitamin B3 molecule and biosynthetic precursor of NAD<sup>5,15</sup>. NR has undergone extensive preclinical testing<sup>16</sup> and is well tolerated by adult humans, showing no evidence of toxicity with doses up to at least 2000 mg daily<sup>17</sup>.

#### 1.2.2 Investigational Product (IP)

NR (Niagen®, Chromadex) is fully approved for human use and no evidence of toxicity has been found. NR has undergone extensive preclinical testing¹6 and is Generally Recognized as Safe (GRAS) for use in food products by the United States Food and Drug Administration³¹ and by the European Food Safety Authority³². NR is well tolerated with no evidence of toxicity in adult humans with doses up to at least 3,000 mg daily¹6-2¹. This evidence includes our recently concluded safety and tolerability trial NR-SAFE (clinicaltrials.gov: NCT05344404), which revealed no adverse events of clinical relevance with 3000mg NR daily for 30 days (manuscript in preparation). We therefore propose that dosages up to 3000 mg is highly unlikely to cause evidence of toxicity. Niagen and placebo will be provided from Chromadex, <a href="https://chromadex.com/">https://chromadex.com/</a>. Active study drug capsules will contain 250 mg NR. Placebo will contain

microcrystalline cellulose, which will be identical in appearance and taste.

# 1.3 Pre-Clinical & Clinical Experience with Investigational Product (IP)

## 1.3.1 Preclinical evidence for NR-therapy

Trials in healthy individuals have shown that oral intake of 1000 mg NR daily substantially elevates total levels of NAD and related metabolites in blood and muscle, boosts mitochondrial bioenergetics and decreases circulating inflammatory cytokines<sup>19,22–24</sup>. Moreover, evidence from cell and animal studies suggests that NR supplementation promotes healthspan and has neuroprotective effects in models of Cockayne syndrome<sup>25</sup>, noise-induced injury<sup>26,27</sup>, amyotrophic lateral sclerosis<sup>28</sup>, Alzheimer's disease <sup>29,30</sup> and PD<sup>31</sup>.

#### 1.3.2 Phase I evidence for NR-therapy in PD

Two phase I studies of NR in PD have been completed, the **NADPARK**<sup>18,32</sup> study and the **NR-SAFE**<sup>21</sup> study. These are described briefly below.

- <u>I. The NADPARK study</u> (ClinicalTrials.gov: *NCT03816020*)<sup>32</sup> is a phase I randomized, double blinded trial, aiming to assess the tolerability, cerebral bioavailability and molecular effects of NR therapy in PD. A total of 30 individuals with newly diagnosed, drug-naïve PD were randomized to NR 500 mg x2/day or placebo for 30 days. The study showed promising results, which were published in 2022<sup>18</sup> and are briefly summarized below:
- **1) NR** is **well-tolerated**: NR 1000 mg per day has excellent compliance, tolerability and no signs of toxicity or adverse effects in PD.
- 2) NR achieves brain penetration: *In vivo* measurement of cerebral NAD levels using phosphorus magnetic resonance spectroscopy (31P-MRS) of the brain showed a highly significant (paired t-test: P = 0.016) increase in cerebral NAD levels in the NR group, while no change was observed in the placebo group (Fig 1A-C). Cerebral penetration was further validated by detecting the metabolite Me-2-PY in the CSF of participants receiving NR, but not placebo (Fig 1G). While a significant NR-induced increase in cerebral NAD levels was detected at the group level, this effect was not uniform at the individual level. The magnitude of the cerebral NAD-increase showed high interindividual variation (Fig 1C). Moreover, three participants showed no evidence of cerebral NAD response, despite a clear peripheral metabolic response, confirming treatment compliance and an impact on the NAD metabolome, in CSF, blood, and muscle. Thus, the variable cerebral NAD response observed by <sup>31</sup>P-MRS may reflect interindividual variability in cerebral penetration and/or cerebral NAD metabolism.
- 3) NR is associated with clinical improvement of PD: NR was associated with a significant decrease in the total MDS-UPDRS (I-III) score between visits (mean decrease:  $2.33 \pm 2.35$ ; paired t-test: p = 0.017).
- **4)** NR has a major impact on cerebral metabolism: <sup>18</sup>F-fluorodeoxyglucose positron emission tomography (FDG-PET), performed at baseline and 30 days of treatment, revealed that NR altered cerebral metabolic activity. The analysis revealed a significant ordinal trend pattern (i.e., metabolic network), which was represented by the first principal component (PC1), accounting for 20.6% of the variance in the paired data. This novel **NR-related metabolic pattern (NRRP)** was characterized by multiple regional metabolic changes, including bilateral metabolic reductions in the caudate and putamen, extending into the adjacent globus pallidus, and in the thalamus (**Fig 1D-E**). Interestingly, the NRRP overlapped spatially with the Parkinson's Disease-Related Pattern (PDRP)<sup>33</sup>, and changes in NRRP expression in the NR group resulted in partial normalization of the striatal and thalamic hypermetabolism (**Fig 1D**), typically

characterizing the PD brain<sup>33</sup>. Furthermore, changes in NRRP expression in the NR group correlated significantly (r=-0.59, p = 0.026) with a decrease of the UPDRS ratings recorded at the time of PET (**Fig 1F**). These results indicate that NR ameliorates the cerebral metabolic pattern of PD, and this is associated with significant clinical improvement.

5) NR has widespread metabolic and regulatory effects: Metabolomics revealed highly significant increase in NAD-related metabolites in blood, muscle and CSF (Fig 1G), indicating that NR supplementation boosts NAD metabolism across tissues. Intriguingly, RNA-sequencing in blood and muscle biopsy showed a highly significant (FDR  $< 10^{-8}$ ) upregulation of the mitochondrial, proteasomal and lysosomal pathways in the NR group. These findings indicate that NR supplementation increases both mitochondrial respiration and proteostasis – two hallmark pathogenic processes involved in PD<sup>34</sup>



**Fig 1. Results of the NADPARK trial. A-C: 31P-MRS** was performed at baseline (v1) and after 30 days of treatment (v2). **A:** exemplary data from one subject showing voxel position. Spectra were acquired for each grid position. **B** (top): average processed spectra from multiple voxels (black) and the model fit (red). **B (bottom):** the model fit is composed of the convolution of all spectral contributions of a simulated dataset fitted to the experimental data. Arrow shows the NAD<sup>+</sup>/NADH spectral peaks. PCr: phosphocreatine. **C:** comparison of cerebral NAD levels in the placebo (PL) and NR groups at baseline (v1) and visit-2 (v2). The Y-axis shows measured levels of NAD normalized to α-ATP (which remain unchanged and stable by the intervention). Individual subjects are indicated by dots. Connecting lines show the change between v1 and v2. The black points and lines show the mean of each group. The treatment group shows a highly significant increase in cerebral NAD levels (\*paired t-test p = 0.016), whereas no difference is observed in the placebo group (paired t-test p = 0.75). **D:** FDG-PET data from all subjects in the NR-group, showing the mean NR-Related Pattern (NRRP, top panel), PD-related pattern (PRDP, middle panel), and the overlap of the two (bottom panel). NR partially ameliorates the striatal and thalamic hypermetabolism of PD. **E:** Between visit changes showing increased NRRP expression in the NR versus the placebo group. The red line indicates mean values before and after the treatment, black lines indicate individuals with a positive NAD response in the

MRS analysis, grey lines indicate individuals without an NAD response in the MRS (\*p =0.027, permutation test, 1000 iterations). **F:** the NR-induced change in metabolic pattern (delta NRRP) shows a strong negative correlation (P<0.01) with the decrease in the UPDRS score (delta UPDRS). **G: Metabolomics in PBMCs, muscle, and CSF.** NR-induced metabolic changes include highly significant (p<<0.001 for all tests) increases in the acid form of NAD (NAAD), and nicotinamide (Nam) degradation products: methyl-Nam (Me-Nam) and the methyl pyridone (Me-2-PY).

- <u>II. The NR-SAFE study</u> (ClinicalTrials.gov: NCT05344404)<sup>21</sup> is a phase I randomized, double blinded trial, aiming to assess the safety, tolerability, and bioavailability of NR in PD at an oral dose of 3000 mg daily. A total of 20 individuals with PD were randomized, in a 1:1 ratio, to NR 1500 mg x2/day or placebo for 30 days. The study was concluded in July 2022 and is currently in preparation. The main results are summarized below:
- 1) NR at a dose of 3000 mg daily is safe and well-tolerated: the treatment had excellent compliance, tolerability, and no signs of toxicity or clinically significant adverse effects in PD.
- **2)** NR, **3000** mg daily, augments NAD-metabolism: oral NR intake at a dose of 3000 mg daily induced a potent (up to 5-fold) and highly significant augmentation of NAD<sup>+</sup> and NADP<sup>+</sup> levels, as well as a clear increase of the redox ratio (NAD<sup>+</sup>/NADH) and the NADP<sup>+</sup>/NADPH ratio (Fig. 2A).
- 3) NR, 3000 mg daily, is associated with clinical improvement of PD: the treatment was associated with a significant and substantial decrease in the total MDS-UPDRS (I-IV) score between visits (mean decrease  $14 \pm 13.7$ ; paired t-test: P = 0.01). No significant change was seen in the placebo group (Fig. 2B). The UPDRS change (delta) in the NR-group was significantly higher than that of the placebo (t-test, P = 0.02) (Fig. 2C).



Fig 2. Results of the NR-SAFE trial. A: Metabolomics were performed in snap-frozen blood from the NR-SAFE participants at baseline (V2) and after 30 days of treatment (V9). Oral NR intake at a dose of 3000 mg daily induced a potent (up to 5-fold) and highly significant augmentation of NAD+ and NADP+ levels, as well as a clear increase of the redox ratio (NAD+/NADH) and the NADP+/NADPH ratio. P-values indicate the results of paired t-tests in the NR-group. There were no significant changes in the placebo group. B: Oral NR intake at a dose of 3000 mg daily was associated with a significant and substantial decrease in total MDS-UPDRS in the NR (mean decrease  $14 \pm 13.7$ ; paired t-test: p = 0.01), but not in the placebo (mean decrease  $1 \pm 12.7$ ; paired t-test: p = 0.81). C: At the group level, the change (delta) in total MDS-UPDRS in the NR group was significantly (t-test, P = 0.02) larger than that of the placebo group (B).

**Key:** V2: baseline; V9: after 30 days of treatment; NR: the group receiving NR 3000 mg daily; PL: the placebo group.

# 1.4 Rationale for the Study and Purpose

Our phase I trials (see section 1.3) showed that NR holds promise as a potential neuroprotective, disease-modifying therapy for PD, and that its effects are likely to be dose-dependent. Encouraged by these findings, this project aims to determine the optimal biological dose of NR in PD and to further explore its neuroprotective potential. The outcomes of this project will take us several steps closer to developing NR into a PD-drug, so that we may harness its full therapeutic potential and maximize its clinical benefit and impact. Specifically, the following knowledge gaps (KG) will be addressed by the N-DOSE study:

**KG1** – **Determine the Optimal Biological Dose (OBD) of NR in PD.** We define the OBD of NR as the dose required to achieve maximal cerebral NAD increase (measured by 31P-MRS or CSF metabolomics), <u>or</u> maximal expression increase in the NRRP (measured by FDG-PET), <u>or</u> maximal proportion of MRS-responders, <u>in the absence of</u> unacceptable toxicity.

While our trials show that the treatment responses to NR in PD are clearly dose-dependent, the OBD of NR in PD remains undetermined. Based on the results of NR-SAFE, it is likely that improved biological and clinical responses can be achieved by escalating the dose. Moreover, the NR OBD may not be universal. NADPARK showed that the NR-mediated increase in cerebral NAD-levels, and accompanying metabolic and clinical response, are not universal and vary across individuals. The fact that all NR-recipients showed a robust metabolic response in blood, muscle and CSF, suggests that the variable cerebral NAD response may reflect interindividual variability in cerebral NAD metabolism (i.e., variation in the rate of NAD-synthesis or consumption). It is likely that such differences can be modulated by varying the substrate concentration (i.e., the intake dose of NR). This question is critical to address, so that NR-therapy can be correctly dosed and tailored to individual patients to achieve an optimal neurometabolic response.

KG2 – Confirm whether NR has a symptomatic clinical effect and assess its dose responsiveness. The NADPARK and NR-SAFE studies showed that NR was associated with a clinical improvement, in the form of UPDRS decrease, and this correlated significantly with the increase in cerebral NAD levels and change in the brain metabolic network (NRRP). Furthermore, the clinical improvement was more pronounced with 3000 mg NR in the NR-SAFE study, compared to 1000 mg in the NADPARK study. These findings suggest that NR may be ameliorating neuronal function in PD, resulting in symptom improvement. Confirming this effect and assessing its dose-dependence will allow us to: 1) determine the optimal clinical dose of NR in PD, and 2) account for symptomatic effects in neuroprotection trials.

**KG3** – **Determine the dose-dependence of the metabolic response to NR therapy.** The NADPARK study showed that a dose of 1000 mg NR daily augmented the NAD metabolome in PBMC, muscle and CSF. The NR-SAFE study suggested that a dose of 3000 mg NR daily leads to a more potent augmentation of the NAD metabolome in blood. The relationship between NR dose and metabolic response needs to be further explored in order to determine optimal dosing regimens.

KG4 – Determine whether NR therapy enhance proteostasis in PD and characterize the dose dependence of this effect. Impaired proteostasis plays a central role in PD and other neurodegenerative disorders, including Alzheimer's disease (AD) and amyotrophic lateral sclerosis (ALS). Our transcriptomic analyses in the NADPARK study indicated that NR therapy may enhance proteostasis by inducing the expression of both proteasomal and lysosomal pathways. If confirmed, this would suggest that NR targets

multiple major processes implicated in the pathophysiology of PD, including mitochondrial respiratory dysfunction, oxidative damage, lysosomal and proteasomal impairment, and neuroinflammation. Moreover, it is not known whether higher NR doses can induce stronger induction of proteostasis in PD.

**KG5** – Determine whether NR therapy influences histone acetylation status and characterize the dose dependence of this effect. We have recently shown that genome-wide histone hyperacetylation and altered transcriptional regulation occur in the brain of individuals with PD<sup>12</sup>. Increasing neuronal NAD levels would boost the activity of the NAD-dependent histone deacetylases of the sirtuin family, potentially, ameliorating histone hyperacetylation in PD. It is currently unknown whether NR-therapy influences histone acetylation status in PD, and whether this effect is dose-dependent.

**KG6 – Confirm that NR therapy decrease neuroinflammation and characterize the dose dependence of this effect.** While it is known that NR has anti-inflammatory properties in peripheral tissues<sup>24</sup>, the results of the NADPARK trial suggest it also downregulates multiple inflammatory cytokines in the central nervous system. If confirmed this would be of importance for PD and other neurodegenerative and neuroinflammatory disorders. Moreover, it is not known whether higher NR doses can induce stronger anti-inflammatory effects in PD.

**KG7 – Determine whether NR therapy alter methylation metabolism and characterize any dose dependence of such an effect.** In theory, NAD replenishment via NR administration could decrease/deplete the cellular methylation capacity. NR boosts the NAD-metabolome, leading to increased production of the degradation product nicotinamide (NAM), which is eliminated via methylation to MeNAM, Me-2-PY, and Me-4-PY, and excreted in the urine. Synthesis of Me-Nam requires the methyl-donor *S*-adenosylmethionine (SAM). This, in turn, could limit SAM availability for other essential methylation reactions, such as DNA and histone methylation, and neurotransmitter synthesis, including dopamine<sup>35</sup>. Thus, in theory, NR would cause an increased consumption of SAM, limiting methylation reactions and generating higher levels of homocystein. Such a phenomenon would be a particular concern for the ~60% of the population that carries MTHFR variants that reduce the efficiency of methylation. The NADPARK study showed no change in serum homocystein levels, or any other evidence of methylation depletion associated with NR 1000 mg daily. It is, however, unknown whether such effects may occur with higher NR doses.

**KG8** – **Determine how orally ingested NR interacts with the microbiome in PD.** Current evidence suggests that the gut microbiome is involved in the pathogenesis of PD and that individuals with PD host a different microbiome composition compared to neurologically healthy individuals<sup>36</sup>. It is possible that NR therapy may beneficially affect the gut microbiome in PD restoring normal patterns. On the other hand, it is also possible that variation in the gut microbiome may affect local metabolism of NR and absorption in the bloodstream. These effects have not been studied.

To address these pertinent questions, we will conduct N-DOSE, a single-center randomized double-blinded placebo-controlled trial to assess the optimal biological dose for NR.

# 2 STUDY OBJECTIVES AND RELATED ENDPOINTS

DS-group refers to the dose-stable group, i.e. participants receiving NR 1000 mg daily for 3 months. DE-group refers to the dose-escalation group, i.e. participants receiving NR 1000 mg in an escalating dose with 1000 mg from baseline to week 4, 2000 mg from week 4 to week 8 and 3000 mg from week 8 to week 12. PL-group refers to the placebo group.

| Objective | | Endpoint |
|---|---|---|
| Primary | To compare the effect of orally administered nicotinamide riboside (NR), escalated to 1500 mg twice per day (3000 mg/day) in the dose-escalation group (DE-group) - versus stable dosing of 500 mg twice per day (1000 mg/day) in the dose-stable group (DS-group) on cerebral NAD-levels, at week 12. | Change in cerebral NAD/ATP- $\alpha$ ratio measured by 31 Phosphorus magnetic resonance spectroscopy (31P-MRS) in the posterior brain (encompassing the occipital, parietooccipital and posterior parts of the temporal cortex). |
| Secondary | To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in cerebral NAD levels from baseline to weeks 4, 8 and 12. | Change in cerebral NAD/ATP-α ratio measured by 31 Phosphorus magnetic resonance spectroscopy (31P-MRS) in the posterior brain (encompassing the occipital, parietooccipital and posterior parts of the temporal cortex). |
| | To compare the effectiveness of orally administered nicotinamide riboside (NR) 1500 mg twice per day versus 500 mg twice per day in augmenting the NAD-metabolome in the central nervous system (CNS) at week 12. | Change in the cerebrospinal fluid (CSF) levels of NAD or other metabolites of the NAD metabolome*, measured by LC-MS. |
| Exploratory | Neuroimaging | |
| | To compare the effect of orally administered NR in the DE-group versus DS-group on the NR related metabolic pattern (NRRP) expression at week 12. | Change in NRRP expression, measured by FDG-PET. |
| | To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in NRRP expression from baseline to weeks 4, 8 and 12. | Change in NRRP expression, measured by FDG-PET. |
| | To compare the effect of orally administered NR DE-group versus DS-group on the PD-related pattern (PDRP) expression at week 12. | Change in PDRP expression, measured by FDG-PET. |
| | To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in PDRP expression from baseline to weeks 4, 8 and 12. | Change in PDRP expression, measured by FDG-PET. |
| | Metabolism & molecular markers | |
| | To compare the effect of orally administered NR in the DE-group versus DS-group on the NAD metabolome* in the blood, urine and central | Change in levels of NAD metabolites in blood, urine and CSF, measured by HPLC-MS and/or the NADMed method. |
| | metabolome in the blood, drine and telltral | the Nadivica method. |

| nervous system (CNS) at week 12. | |
|---|---|
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in levels of NAD metabolites in bloo |
| per day) and changes in the NAD metabolome* | and urine, measured by HPLC-MS and/or th |
| in blood and urine from baseline to weeks 4, 8 | NADMed method. |
| and 12. | |
| To compare the effect of orally administered NR | Change in inflammatory cytokines in serum an |
| in the DE-group versus DS-group on serum and | Change in inflammatory cytokines in serum ar |
| CSF inflammatory markers at week 12. | CSF, measured by ELISA. |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in inflammatory cytokines in serur |
| per day) and changes in serum inflammatory | measured by ELISA. |
| markers from baseline to weeks 4, 8 and 12. | |
| Clinical – motor & non motor symptom severity, | quality of life |
| To compare the effect of orally administered NR | , quanty of me |
| · | Change in the total MDS-UPDRS score in the |
| in the DE-group versus DS-group on clinical | ON-medication state. |
| severity of PD symptoms at week 12. | |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in total MDS-UPDRS score in the O |
| per day) and change in clinical severity of PD | medication state. |
| symptoms from baseline to weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on severity of | Change in the MDS-UPDRS part I score in t |
| non-motor symptoms of daily living in PD at | ON-medication state. |
| week 12. | |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | Change in the MDC LIDDDC next I seems in t |
| per day) and change in severity of non-motor | Change in the MDS-UPDRS part I score in t |
| symptoms of daily living in PD from baseline to | ON-medication state. |
| weeks 4, 8 and 12. | |
| To compare the effect of orally administered NR | |
| in the DE-group versus DS-group on severity of | Change in the MDS-UPDRS part II score in t |
| motor aspects of experiences of daily living in | ON-medication state. |
| PD at week 12. | - 25 |
| To assess the dose-response relationship | |
| between NR dose (1000 mg, 2000 mg, 3000 mg | |
| per day) and changes in severity of motor | Change in the MDS-UPDRS part II score in t |
| aspects of symposius and delications in DD f | ON-medication state. |
| aspects of experiences of daily living in PD from | ON-medication state. |
| baseline to weeks 4, 8 and 12. | ON-medication state. |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR | |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of | Change in the MDS-UPDRS part III score in t |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of PD motor symptoms at week 12. | |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of | Change in the MDS-UPDRS part III score in t |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of PD motor symptoms at week 12. | Change in the MDS-UPDRS part III score in t<br>ON-medication state. |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of PD motor symptoms at week 12. To assess the dose-response relationship | Change in the MDS-UPDRS part III score in t ON-medication state. |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of PD motor symptoms at week 12. To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg | Change in the MDS-UPDRS part III score in to ON-medication state. Change in the MDS-UPDRS part III score in to the MDS-UPDRS part III score in to the MDS-UPDRS part III score in the MDS-UPD |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of PD motor symptoms at week 12. To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in severity of PD motor | Change in the MDS-UPDRS part III score in to ON-medication state. Change in the MDS-UPDRS part III score in to ON-medication state. |
| baseline to weeks 4, 8 and 12. To compare the effect of orally administered NR in the DE-group versus DS-group on severity of PD motor symptoms at week 12. To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in severity of PD motor symptoms from baseline to weeks 4, 8 and 12. | Change in the MDS-UPDRS part III score in to ON-medication state. Change in the MDS-UPDRS part III score in to the MDS-UPDRS part III score in to the MDS-UPDRS part III score in the MDS-UPD |

| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in severity of PD motor complications from baseline to weeks 4, 8 and 12. | Change in the MDS-UPDRS part IV score in the ON-medication state. |
|---|---|
| To compare the effect of orally administered NR in the DE-group versus DS-group on clinical severity of PD non-motor symptoms at week 12. | Change in the total MDS-NMS score. |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in clinical severity of PD non-motor symptoms from baseline to weeks 4, 8 and 12. | Change in the total MDS-NMS score. |
| To compare the effect of orally administered NR in the DE-group versus DS-group on clinical severity of gastrointestinal non-motor dysfunction in PD at week 12. | Change in the modified GIDS-PD score. |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in clinical severity of gastrointestinal non-motor dysfunction in PD from baseline to weeks 4, 8 and 12. | Change in the modified GIDS-PD score. |
| To compare the effect of orally administered NR in the DE-group versus DS-group on cognition at week 12. | Change in the MoCA score. |
| To assess the dose-response relationship<br>between NR dose (1000 mg, 2000 mg, 3000 mg<br>per day) and changes in cognition from baseline<br>to weeks 4, 8 and 12. | Change in the MoCA score. |
| To compare the effect of orally administered NR in the DE-group versus DS-group on quality of life in PD at week 12. | Change in the EQ-5D-5L score. |
| To assess the dose-response relationship<br>between NR dose (1000 mg, 2000 mg, 3000 mg<br>per day) and changes in quality of life in PD from<br>baseline to weeks 4, 8 and 12. | Change in the EQ-5D-5L score. |
| Hypothesis-generating or resource-dependent endpoints (may be reported in follow-up or secondary publications). | |
| To compare the effect of orally administered NR in the DE-group versus DS-group on gene expression at week 12. | Change in gene expression, measured by RNA sequencing (RNAseq). |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in gene expression from baseline to weeks 4, 8 and 12. | Change in gene expression, measured by RNA sequencing (RNAseq). |
| To compare the effect of orally administered NR in the DE-group versus DS-group on protein expression at week 12. | Change in protein levels, measured by LC-MS. |

| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in protein expression from baseline to weeks 4, 8 and 12. | Change in protein levels, measured by LC-MS. |
|---|---|
| To compare the effect of orally administered NR in the DE-group versus DS-group on serum and CSF inflammatory markers at week 12. | Change in inflammatory cytokines in serum and CSF, measured by ELISA. |
| To assess the dose-response relationship<br>between NR dose (1000 mg, 2000 mg, 3000 mg<br>per day) and changes in serum inflammatory<br>markers from baseline to weeks 4, 8 and 12. | Change in inflammatory cytokines in serum, measured by ELISA. |
| To compare the effect of orally administered NR in the DE-group versus DS-group on histone acetylation in PD at week 12. | Change in histone panacetylation, measured by immunoblotting. |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in histone acetylation in PD from baseline to weeks 4, 8 and 12. | Change in histone panacetylation, measured by immunoblotting. |
| To compare the effect of orally administered NR in the DE-group versus DS-group on H3K27 and H4K16 histone acetylation in PD at week 12. | Changes in levels of H3K27 and H4K16 acetylation, measured by immunoblotting. |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in on H3K27 and H4K16 histone acetylation in PD from baseline to weeks 4, 8 and 12. | Changes in levels of H3K27 and H4K16 acetylation, measured by immunoblotting. |
| To compare the effect of orally administered NR in the DE-group versus DS-group on the genomic distribution of H3K27 and H4K16 histone acetylation in PD at week 12. | Change in the genomic distribution of H3K27 and H4K16 acetylation, measured by chromatin immunoprecipitation sequencing (ChIPseq). |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in the genomic distribution of H3K27 and H4K16 histone acetylation in PD from baseline to weeks 4, 8 and 12. | Change in the genomic distribution of H3K27 and H4K16 acetylation, measured by chromatin immunoprecipitation sequencing (ChIPseq). |
| To compare the effect of orally administered NR in the DE-group versus DS-group on folate and one-carbon metabolism in PD at week 12. | Change in folate and one-carbon metabolites in blood and CSF, measured by HPLC-MS. |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in folate and one-carbon metabolism in PD from baseline to weeks 4, 8 and 12. | Change in folate and one-carbon metabolites in blood, measured by HPLC-MS. |
| To compare the effect of orally administered NR in the DE-group versus DS-group on methyl donors in PD at week 12. | Change in methyl-donors (e.g., SAM), measured by HPLC-MS, in the blood and/or CSF. |
| To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg | Change in methyl-donors (e.g., SAM), measured by HPLC-MS, in the blood. |

| | per day) and changes in methyl-donors in PD | |
|---|---|---|
| | from baseline to weeks 4, 8 and 12. | |
| | To compare the effect of orally administered NR | Change in level and genomic distribution of DNA |
| | in the DE-group versus DS-group on DNA | methylation, measured by Illumina Infinium |
| | methylation at week 12. | MethylationEpic kit. |
| | To assess the dose-response relationship | Change in level and consumindictable with the of DNA |
| | between NR dose (1000 mg, 2000 mg, 3000 mg | Change in level and genomic distribution of DNA |
| | per day) and changes in methyl-donors in PD | methylation, measured by Illumina Infinium |
| | from baseline to weeks 4, 8 and 12. | MethylationEpic kit. |
| | To compare the effect of orally administered NR | Change in neurotransmitters in CSE measured |
| | in the DE-group versus DS-group on synthesis of | Change in neurotransmitters in CSF, measured |
| | neurotransmitters in PD at week 12. | by HPLC-MS. |
| | Determine whether NR-therapy affects the gut | Change in gut microbiome composition, measured by metagenomics in fecal samples. |
| | microbiome in a dose-responsive manner at | |
| | week 12. | measured by metagenomics in recar samples. |
| | To compare the effect of orally administered NR | Change in fecal metabolomics, measured by LC- |
| | in the DE-group versus DS-group on the gut | MS in fecal samples. |
| | metabolome at week 12. | ivis in recar samples. |
| | To compare the effect of orally administered NR | Change in conce of small measured by D.CIT. |
| | in the DE-group versus DS-group on the sense | Change in sense of smell, measured by B-SIT |
| | of smell at week 12. | score. |
| Safety | To determine the safety and tolerability of NR | Number and severity of adverse events from |
| | at a dose of 1000 mg, 2000 mg, and 3000 mg | baseline to week 12 across treatment groups |
| | per day in PD. | and NR dose levels. |

\*The NAD metabolome is comprised of: Nicotinamide adenine dinucleotide oxidized (NAD+), Nicotinamide adenine dinucleotide reduced (NADH), NAD+/NADH ratio, total NAD (sum of NAD+ and NADH), Nicotinamide adenine dinucleotide phosphate oxidized (NADP+), Nicotinamide adenine dinucleotide phosphate reduced (NADPH), NADP+/NADPH ratio, total NADP (sum of NADP+ and NADPH, 1-methyl nicotinamide (Me-Nam), nicotinic acidadenine dinucleotide (NAAD), N1-methyl-2-pyridone-5-carboxamide (Me-2-PY), Nicotinamide (Nam), Nicotinamide N-oxide (Nam N-oxide), ADP-ribose (ADPR), Nicotinic acid riboside (NAR), Nicotinamide riboside (NR), Nicotinamide mononucleotide (NMN), Nicotinic acid (NA).

# 2.1 Primary Endpoint Measure

Change in cerebral NAD level, measured by <sup>31</sup>P-MRS.

<sup>31</sup>P-MRS assesses the levels of key-energy metabolites in the brain, including NAD, ATP, free inorganic phosphate (Pi), and phosphocreatine, and others, as previously shown<sup>18,37</sup>. Using this method, we will assess total brain NAD levels normalized to ATP- $\alpha$  levels (i.e., the NAD/ATP- $\alpha$  ratio) in the posterior brain - encompassing the occipital, parietooccipital and posterior parts of the temporal cortex.

## 2.2 Secondary Endpoint Measure

Change in the CSF level of NAD or other metabolites of the NAD metabolome in CSF, measured by HPLC-MS.

Using **high performance liquid chromatography mass spectrometry (HPLC-MS)**, we will measure the NAD metabolome in CSF, including the following specific measures: Nicotinamide adenine dinucleotide oxidized (NAD+), Nicotinamide adenine dinucleotide reduced (NADH), NAD+/NADH ratio, total NAD (sum

of NAD<sup>+</sup> and NADH), Nicotinamide adenine dinucleotide phosphate oxidized (NADP<sup>+</sup>), Nicotinamide adenine dinucleotide phosphate reduced (NADPH), NADP<sup>+</sup>/NADPH ratio, total NADP (sum of NADP<sup>+</sup> and NADPH, 1-methyl nicotinamide (Me-Nam), nicotinic acid-adenine dinucleotide (NAAD), N1-methyl-2-pyridone-5-carboxamide (Me-2-PY), Nicotinamide (Nam), Nicotinamide N-oxide (Nam N-oxide), ADP-ribose (ADPR), Nicotinic acid riboside (NAR), Nicotinamide riboside (NR), Nicotinamide mononucleotide (NMN), Nicotinic acid (NA).

# 2.3 Exploratory Endpoint Measures

Change in the following parameters listed below:

**NR** related pattern (NRRP), an ordinal trend pattern (i.e., metabolic network), associated with NR treatment identified in the NADPARK study<sup>18</sup>, measured by <sup>18</sup>F-fluorodeoxyglucose positron emission tomography (FDG-PET).

**PD** related pattern (PDRP), an ordinal trend pattern (i.e., metabolic network), associated with PD<sup>33</sup>, measured by <sup>18</sup>F-fluorodeoxyglucose positron emission tomography (FDG-PET).

The International Parkinson and Movement Disorder Society – Non-Motor Rating Scale (MDS-NMS)<sup>38</sup>, a 52 item scale that assesses the frequency and severity of non-motor symptoms in PD across 13 non-motor domains. The MDS-NMS consists of two parts: the Total MDSS-NMS (range 0-832) and the MDS-NMS Non-Motor Fluctuations (NMF) Subscale to assess changes in non-motor symptoms in relation to the timing of anti-parkinsonian medication (range 0-128). Each item in each scale is scored according to frequency from 0 to 4 and severity from 0 to 4. Each item's frequency is then multiplied by its severity to calcultate the item scorer. A low score indicates a good outcome, higher scores indicate a poorer outcome.

The International Parkinson's disease and movement disorders society unified Parkinson's disease rating scale (MDS-UPDRS)<sup>39</sup> is a scale assessing clinical impairment and disability in PD. It consists of 4 parts. Part I assesses non-motor experiences of daily living and has 2 components IA and IB (Range 0-52). Part IA comprises 6 questions assessed by the examiner (Range 0-24). Part IB comprises 7 questions completed by the participants (Range 0-28). Part II assesses motor experiences of daily living (Range 0-52). It comprises 13 questions completed by the participant. Part III evaluates motor severity and contains 33 scores based on 18 items, which are assessed by the rater during clinical examination (Range 0-132). Part IV assesses motor complications, which comprises 6 questions assessed by the examiner (Range 0-24). For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of parts I, II, III and IV (Range 0-260). A higher score indicates more severe symptoms of PD.

**MDS-UPDRS part I** is a scale assessing non-motor experiences of daily living and has 2 components (Range 0-52). Part IA comprises 6 questions assessed by the examiner (Range 0-24). Part IB comprises 7 questions completed by the participants (Range 0-28). A higher score indicated more severe symptoms. This will be assessed in the ON medication state.

**MDS-UPDRS part II** assesses motor experiences of daily living (Range 0-52). It comprises 13 questions completed by the participant. A higher score indicated more severe symptoms. This will be assessed in the ON medication state.

MDS-UPDRS part III evaluates motor severity and contains 33 scores based on 18 items, which are assessed by the rater during clinical examination (Range 0-132). For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score

indicated more severe symptoms. This will be assessed in the ON medication state.

MDS-UPDRS part IV evaluates motor complications and contains 6 questions assessed by the examiner (Range 0-24). For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms. This will be assessed in the ON medication state.

The International Parkinson and Movement Disorder Society Gastrointestinal Dysfunction Scale in Parkinson's Disease (mGIDS-PD) $^{40}$  modified\*. The following version of GIDS-PD has been modified by permission and license from MDS for use in the N-DOSE trial. The modifications in this version are that the timeframe for all questions has been reduced from six months to one month. Part 1b has also been omitted from the scale. A low score indicates a good outcome, higher scores indicate a poorer outcome. The range is 0 to 108 points. The scale consists of two main parts: Section 1 -12, which are counted as a scale. Section 1a, and sections A - F, which are anamnestic and do not count towards the scale score.

**MoCA**<sup>41</sup> is a validated global measure of cognitive ability. This will be assessed in the ON medication state.

**EQ-5D-5L**<sup>42</sup> is a 5 item questionnaire and visual analogue scale that allows calculation of quality adjusted life years (QALY) to enable health economic analyses to be performed. The questionnaire covers 5 domains with scores 0 to 4. A low score indicates a good outcome, higher scores indicate a poorer outcome. The EQ VAS score in mm is a general assessment from the participants perspective of how good their health is, from 0 to 100. A low score indicates a poor outcome, a high value indicates a better outcome.

NAD metabolome. Using liquid chromatography mass spectrometry (HPLC-MS) and/or the NADMed method, we will measure the NAD metabolome in whole blood (and/or PBMCs), CSF and urine including the following specific measures: Nicotinamide adenine dinucleotide oxidized (NAD+), Nicotinamide adenine dinucleotide reduced (NADH), NAD+/NADH ratio, total NAD (sum of NAD+ and NADH), Nicotinamide adenine dinucleotide phosphate oxidized (NADP+), Nicotinamide adenine dinucleotide phosphate reduced (NADPH), NADP+/NADPH ratio, total NADP (sum of NADP+ and NADPH, 1-methyl nicotinamide (Me-Nam), nicotinic acid-adenine dinucleotide (NAAD), N1-methyl-2-pyridone-5-carboxamide (Me-2-PY), Nicotinamide (Nam), Nicotinamide N-oxide (Nam N-oxide), ADP-ribose (ADPR), Nicotinic acid riboside (NAR), Nicotinamide riboside (NR), Nicotinamide mononucleotide (NMN), Nicotinic acid (NA).

**Gene and protein expression levels in PBMC,** measured by RNA sequencing (RNAseq) and proteomics (HPLC-MS), respectively.

**Levels of inflammatory cytokines in serum and CSF**, measured using enzyme-linked immunosorbent essay (ELISA).

Levels of histone panacetylation, and levels and genomic distribution of H3K27 and H4K16 acetylation in PBMC, measured by immunoblotting and chromatin immunoprecipitation sequencing (ChIPseq).

Levels of methyl-donors (e.g., SAM) in blood and/or CSF, measured by HPLC-MS.

**Levels of neurotransmitters in CSF**, measured by HPLC-MS.

Levels of one carbon metabolism metabolites, measured by HPLC-MS metabolomics in PBMC and CSF.

Levels and genomic distribution of DNA methylation, measured by the Illumina Infinium

MethylationEPIC Kit.

**Gut microbiome composition**, assessed by metagenomics in fecal samples.

Fecal metabolomics, including fatty acid profiling, assessed by HPLC-MS in fecal samples.

**Brief Smell Identification Test (B-SIT)** assesses olfaction. It consists of 12 items with 4 alternatives, from which the participant attempts to identify the correct smell. It is performed by the participant under supervision of the investigator. Not available for all participants as this was added as an exploratory outcome during the trial. A low score indicates a poor outcome, higher scores indicate a better outcome. The range for the total score is 0 to 12 points.

## 3 OVERALL STUDY DESIGN

This is a single-center, phase II, double blinded, randomized, placebo-controlled dose-optimization study.

Study Period Estimated date of first patient enrolled: 28.11.2022

Anticipated recruitment period: 28.11.2022 - 20.01.2025B

Estimated date of last patient completed: 22.04.2025

Treatment Duration: 12 weeks.

# 3.1 Study design

N-DOSE is a single-center, phase II, double blinded, randomized, placebo-controlled dose-optimization clinical trial with a dose escalation design. Patients with PD (n = 80) who fulfil participation criteria (see section 4) will be randomized (1:1:2) into one of three groups: 1) The placebo group (PL-group, n = 20) will receive placebo for the duration of the study. 2) The NR 1000 mg group (DS-group, n=20) will receive NR 1000 mg (500 mg x 2) per day for the duration of the study. 3) The NR dose escalation group (DE-group, n=40) will receive first 1000 mg (500 mg x 2) NR per day for 30 days, then 2000 mg (1000 mg x 2) NR per day for 30 days (Fig. 3). The selected dose range is within safety limits for healthy humans (see section 1.3). After eligibility screening, eligible participants will be randomly assigned to one of three study groups and assessed at baseline (Visit-1, V1) and three more visits (Visit-2, Visit-3 and Visit-4; V2, V3, V4) spaced 30 days apart (Fig. 3). Participants and investigators will be blinded to treatment group. Participants will be followed for a total of 90 days. All participants will be recruited from the Neuro-SysMed Center, at the department of Neurology, Haukeland University Hospital (HUS).



**Figure 3.** N-DOSE design. A total of 80 patients will be recruited in three arms. Patients will be assessed at baseline (V1) and three additional visits, at 4 (V2), 8 (V3) and 12 (V4) weeks.

#### 4 STUDY POPULATION

# 4.1 Selection of Study Population

The study will include individuals  $\geq$  40 years with a clinically established diagnosis of PD according to the MDS criteria<sup>43</sup>, and Hoehn and Yahr score < 4 (see full list of eligibility criteria below). Participants from all of Norway will be recruited at the department of Neurology, Haukeland University Hospital.

#### 4.2 Number of Patients

A total of n=80 patients will be included in this study and randomized to placebo (PL-group, n=20), NR 500 mg twice per day (DS-group, n=20), or NR escalating dose (DE-group, n=40), starting at 500 mg twice per day, increasing to 1000 mg twice per day, and finally increasing to 1500 mg twice per day.

#### 4.3 Inclusion Criteria

The following condition must apply to the prospective patient at screening prior to receiving study agent:

- Clinically established diagnosis of PD according to the MDS criteria.
- 123I-Ioflupane dopamine transporter imaging (DAT-scan) or 18-F-FDOPA positron emission tomography imaging (18F-FDOPA PET) confirming nigrostriatal degeneration.
- Hoehn and Yahr score < 4 at enrolment.
- Age ≥ 40 years at the time of enrollment.
- Able to undergo lumbar punction.
- Able to undergo MRI

#### 4.4 Exclusion Criteria

Patients will be excluded from the study if they meet any of the following criteria:

- Dementia or other neurodegenerative disorder at baseline visit.
- Diagnosed with atypical parkinsonism (PSP, MSA, CBD) or vascular parkinsonism.
- Any psychiatric disorder that would interfere with compliance in the study.
- Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.
- Use of high dose vitamin B3 supplementation within 30 days of enrollment.

## 5 TREATMENT

For this study NR (Niagen®, Chromadex) is defined as the Investigational Product(s) (IP). IP includes also active comparator and placebo.

# 5.1 Drug Identity, Supply and Storage

NR (Niagen\*, Chromadex) and placebo will be manufactured and provided from Chromadex. Both NR and Placebo will be prepared as identical capsules. The drug has marketing consent in Norway but is not registered by Statens legemiddelverk (SLV)/Direktoratet for medisinske produkter (DMP) as medical drug but as a supplement. The NR and placebo have a 1-year expiry date. Both the NR and placebo will be stored in room temperature with temperature <25 degrees (according to instructions given by Chromadex).

# 5.2 Dosage and Drug Administration

Each NR capsule contains 250 mg. To keep the study fully blinded, all participants will receive the same number of daily capsules irrespective of which treatment group they belong to. To achieve this, NR capsules will be combined with placebo capsules as necessary (see below):

- Patients in the NR 1000mg group will administer orally [2 NR capsules (250mg) + 4 placebo capsules] x 2 times daily (1000mg NR daily in total).
- Patients in the NR dose escalation group will administer orally the following doses:
  - Weeks 0-4: [2 NR capsules (500mg) + 4 placebo capsules] x 2 times daily (1000mg NR daily in total).
  - Weeks 5-8: [4 NR capsules (1000mg) + 2 placebo capsules] x 2 times daily (2000mg daily total).
  - Weeks 9-12: [6 NR capsules (1500mg) + 0 placebo capsules] x 2 times daily (3000mg daily total).
- The placebo group will administer orally [6 placebo capsules] x 2 times daily.

There is no specified time of day the dosages should be taken, only that they should be taken with about 12 hours apart if possible. If a dose is missed, the patient can take the missed dose as soon as it is remembered, provided it is shorter time to the missed dose than the next scheduled dose. There are no restrictions with respect to combining the dose with other medication and/or food.

The study medication is to be taken every day during the treatment period, and must be taken prior to study visits.

# 5.3 **Duration of Therapy**

Therapy duration for the study is 3 months (12 weeks).

# 5.4 Dopaminergic therapy during Screening and Treatment period

Eligible and consenting men and women with PD will be given optimal dopaminergic therapy, as indicated by their clinical disease. All and any form of dopaminergic therapy formally approved in Norway may be used. Patients who do not use dopaminergic therapy are eligible, provided that they have a clinically established diagnosis of PD according to the MDS criteria. The treatment regimen will be optimized, if necessary, and will then be frozen and remain unchanged for the study period (3 months):

- For patients who are already on dopaminergic therapy, the regimen may be adjusted, if
  necessary, to optimal clinical effect. Adjustment may involve change in dose, formulation, or
  drug. When adjustment of the dopaminergic regimen is undertaken, treatment efficacy will be
  assessed upon reexamination by physical or telephone consultation, until optimal effect or
  exclusion. Once the treatment regimen is deemed optimal, it will be frozen and remain
  unchanged for the study period (3 months).
- Newly diagnosed and/or treatment naïve patients will be given dopaminergic treatment if- and
  as appropriate based on clinical indication. The treatment will be titrated to optimal effect.
  When adjustment of the dopaminergic regimen is undertaken, treatment efficacy will be
  assessed upon reexamination by physical or telephone consultation, until optimal effect or
  exclusion. Once the treatment regimen is deemed optimal, it will be frozen and remain
  unchanged for the study period (3 months).
- Patients who do not use dopaminergic therapy are eligible, provided that they have a clinically established diagnosis of PD according to the MDS criteria.

If adverse effects occur due to the dopaminergic therapy after enrollment, the treatment will be adjusted according to good clinical practice. All patients will be enrolled to the main study within 3 months after the last screening if inclusion/exclusion criteria are fulfilled.

At the end of study visit (month 3), the physician determines whether the patient is still adequately treated for his/her parkinsonism with their current dopaminergic treatment.

#### 5.5 Concomitant Medication

Dopaminergic therapy will be given as described in section 5.4. above.

In addition, the patient should not take any vitamin B3 supplements for the duration of the study.

There are no other restrictions on any other use of medications. All patients should use medications prescribed prior to enrollment in the study. There are no restrictions with respect to starting new medications that are necessary for the patient.

All concomitant medication (incl. vitamins with the exception of vitamin B3, herbal preparation and other "over-the-counter" drugs) used by the patient will be recorded in the patient's file and CRF.

# 5.6 Subject Compliance

Patient compliance will be determined based on self-report at study visits. A pill count of remaining medication will be performed when providing new study medication and at the end of the study.

# 5.7 Drug Accountability

The responsible site personnel will confirm receipt of study drug and will use the study drug only within the framework of this clinical study and in accordance with this protocol. Receipt, distribution, return, and destruction (if any) of the study drug must be properly documented according to the sponsor's agreed and specified procedures. Study drugs are stored locally at the study site and distributed by the study nurse upon registration in CRF. Remaining study drug is returned for pill count.

# 5.8 Drug Labeling

The investigational product will have a label permanently affixed to the outside and will be labeled according with ICH GCP and national regulations, stating that the material is for clinical trial / investigational use only and should be kept out of reach of children.

#### Label will include:

- Kit number
- Study number (CRF number)
- Expiration date

# 5.9 Subject Numbering

At the screening visit, each patient will be sequentially allocated a study identification number by the CRF (i.e., the registration code of the patient in the CRF). The study identification should be as follows: YYYY, where YYYY is the chronological enrolled subject number (e.g., 0001, 0002, etc.). For example: 002 (patient number 002). The next enrolled patient is registered as 003.

The subjects will be identified by this study identification number for the remainder of the study. Once a patient number has been assigned, no attempt will be made to use that number again. If a patient number is allocated incorrectly, no attempt will be made to remedy the error once study treatment has been dispensed. Any replacement patients will be given the next patient number in the sequence.

## **6** STUDY PROCEDURES

#### 6.1 Flow Chart

Table 1. Trial flow chart

| | Scree | ning Period | Treatment Period<br>Study Visit | | | |
|---|---|---|---|---|---|---|
| Event | First<br>Screening | Subsequent/<br>last screening | Visit-1<br>Baseline | Visit-2 | Visit-3 | Visit-4 |
| Time | | | Week 1 | Week 4 | Week 8 | Week 12 |
| Informed consent | X | | | | | |
| Informed consent | Х | | | | | |
| biobank | ^ | | | | | |
| MDS Clinical diagnosis | X | | | | | |
| Criteria (MDS CDC) | Х | | | | | |
| Inclusion/exclusion | X | | Х | | | |
| Evaluation | X | | ^ | | | |
| Medical history <sup>1</sup> | Х | | Х | | | |
| Physical Examination <sup>2</sup> | Х | | Х | X | Х | X |

| | Screening Period | | Treatment Period Study Visit | | | |
|---|---|---|---|---|---|---|
| Event | First<br>Screening | Subsequent/<br>last screening | Visit-1<br>Baseline | Visit-2 | Visit-3 | Visit-4 |
| General neurological examination | Х | | | | | |
| Body height | | | Χ | | | |
| Vital signs <sup>3</sup> | | | Х | Х | Х | Х |
| Body weight and BMI | | | Х | Х | X | Х |
| Record of concomitant medication <sup>9</sup> | х | | Х | х | х | Х |
| Hoehn and Yahr score | Х | | Χ | Х | X | Х |
| DAT-Scan or 18F-FDOPA<br>PET <sup>4</sup> | х | | | | | |
| 31P-MRS & 1H-MRS of | | | | | ., | ., |
| the brain | | | Χ | X | X | Χ |
| FDG-PET of the brain | | | Х | Х | Х | Х |
| MDS-UPDRS (I-IV) | | | Х | Х | Х | Х |
| MDS-NMS | | | Х | Х | Х | Х |
| MoCA | | | Х | Х | X | Х |
| EQ-5L | | | Х | Х | Х | Х |
| GIDS-PD | | | Х | Х | Х | Х |
| B-SIT | | | Х | | | Х |
| Dietary registration (3 days) | | | Х | | | Х |
| Routine blood tests <sup>5</sup> | | | Х | Х | Х | Х |
| Blood collection for biobanking <sup>6</sup> | | | Х | Х | х | Х |
| Cerebrospinal fluid collection | | | X | | | X |
| Fecal sample collection | | | Χ | | | Χ |
| Urine sample collection | | | Χ | X | X | Χ |
| Treatment dispensation <sup>7</sup> | | | Χ | X | X | |
| Dopaminergic treatment stable <sup>8</sup> | х | X | | | | X |
| Adverse event | | | | Х | Х | Х |

Superscripts refer to the specifications below.

#### Specifications (details in section

- Medical history includes: family history of neurological illness (what and who), family history of PD (what and who), smoking history (period, pack-years), first PD symptoms, months since first PD symptoms, occurrence and duration of REM sleep disorder symptoms, occurrence and duration of loss of smell.
- 2. Heart and lung auscultation, abdominal palpation, any other examination dictated by patient's condition/symptoms
- 3. Blood pressure, pulse, temperature
- 4. DAT-Scan or 18F-FDOPA PET must have been performed prior to the Baseline Study Visit.
- 5. CRP, ALAT, ASAT, GT, bilirubin, ALP, creatinine, urea, RBC, Hb, WBC with differential, platelets, CK, FT4, TSH, B12, folic acid, homocysteine, methylmalonic acid, sodium, potassium, glucose. Women of childbearing potential will also have a pregnancy test performed.
- 6. EDTA blood, snap-frozen EDTA blood, platelets, serum (see lab manual for details).
- 7. To ensure correct dosages during dose escalation and if necessary to resupply.

- 8. The patient must be on a stable dopaminergic treatment regimen. When the patient is on a stable dopaminergic treatment, the screening is over, and the patient can be included in the study. The dopaminergic treatments are listed in section 5.4. There should not be more than 3 months from the last screening to the baseline visit.
- 9. Record of concomitant medication: in addition to all drugs used by the patient, the type of dopaminergic medication used and the time points in the day at which each dose is taken must be registered.

# 6.2 By Visit

# 6.2.1 Screening Visits/ Before start of Investigational Product (IP)

The first screening visit aims to determine if the patient is eligible to be included in the study. A full physical examination and anamnestic medical history is performed. If the patient fulfills the inclusion/exclusion criteria and gives informed consent, dopaminergic treatment is initiated/adjusted as described in the treatment flowchart in section 5.4.

If the patient is optimally treated with dopaminergic treatment and fulfills the inclusion/exclusion criteria, then the patient is deemed ready for enrolment and may be referred to MRI and PET. If changes are made to the dopaminergic treatment, then the subject is contacted by phone after 2-6 weeks to assess if the treatment is optimal. If the patient is optimally treated, this dopaminergic treatment is frozen for the remainder of the study and the patient is referred to MRI and PET and called in for the baseline study visit (week 0 study visit). The patient should at screening be advised to stop using any Vit B3 supplement to fulfill inclusion criteria. There should not be more than 3 months from the last screening to baseline visit.

#### Screening checklist:

- 1. Patient signs informed consent for N-DOSE
- 2. Patient signs informed consent for consent for storage and analysis of biological material ("Samtykke for lagring av biologisk material i biobank for demens og aldring")
- 3. Physical examination (general neurological examination) at first screening
- 4. MDS clinical diagnosis Criteria
- 5. Record current use of medication. Advise to stop any use of vit B3 supplements
- 6. Introduce/adjust dopaminergic treatment as described in section 5.4.
- 7. If the patient is ready for enrollment, they are referred to baseline study visit (including MRI and PET).
- 8. The patient is given the 3-day dietary registration form along with instructions on how to fill it out and deliver to the study nurse at baseline.
- 9. Register when the patient takes their dopaminergic medication (dose and time of the day).
- 10. Patient is asked to note the time of dopaminergic therapy intake on the morning of each visit
- 11. Visits should be planned so that the patient is at the Department at a time permitting the MDS-UPDRS to be conducted within <u>no less than 15min and no more than 2 hours</u> after the last intake of dopaminergic medication.
- 12. MDS-UPDRS must be conducted at the same interval from the last dopaminergic therapy dose on every visit (+/- 30min)

#### 6.2.2 Baseline/Week 0

1. Investigator verifies the informed consent for the study.

- 2. Investigator verifies anamnestic information gathered at screening, current use of medication and medical history.
- 3. Investigator verifies fulfillment of inclusion and exclusion criteria.
- 4. The study identification number is assigned (see section 5.9).
- 5. Study medication is dispensed to the subject by the study nurse and the patient is reminded to take the study medication every day including the morning of each visit.
- 6. Register the time the patient took dopaminergic medication on the morning of the visit as well as the type and dose of the medication.
- 7. The following clinical examination are performed by the study nurse or investigator (see flowchart in section 6.1):
  - Vital signs
  - o Body weight and BMI
  - o MDS CDC
  - o MDS-UPDRS: section 1&2 by study nurse/investigator, section 3&4 by investigator
  - o MDS-NMS
  - o MoCA
  - o EQ-5L
  - o GIDS-PD
- 8. Routine blood tests are done (see flowchart in section 6.1)
- 9. Samples for biobanking are taken (see flowchart in section 6.1):
  - o EDTA whole blood
  - Snap-frozen whole blood
  - o PAXgene blood for RNA
  - o Serum
  - o Fecal sample
  - o Urine sample
  - Cerebrospinal fluid
- 10. Imaging is conducted
  - o 31P-MRS & 1H-MRS
  - o FDG-PET
- 11. All data gathered during study visits is either written into the electronic journal or filled out in paper format with appropriate date and signatures. Each patient will have their own folder with gathered clinical data. The clinical tests (MDS-UPDRS, MDS-NMS, MoCA, MDS CDC, EQ-5L, GIDS-PD) are recorded in paper format.
- 12. The patient is given the 3-day dietary registration form along with instructions on how to fill it out and deliver it to the study nurse at the next visit.
- 13. Patient is reminded to note the time of dopaminergic therapy intake on the morning of the next visit
- 14. Next visit should be planned so that the patient is at the Department at a time permitting the MDS-UPDRS to be conducted within **no less than 15min and no more than 2 hours** after the last intake of dopaminergic medication.
- 15. MDS-UPDRS must be conducted at the same interval from the last dopaminergic therapy dose on every visit (+/- 30min)
- 16. B-SIT is performed by either the study nurse or investigator (see flowchart in section 6.1).

#### 6.2.3 **During treatment (visits 2-4)**

- Should the patient need replenishing of study medication, it will be logistically handled by the study nurse.
- On visit 2 points 5-11 and 13-15 from section 6.2.2 are repeated.

•

• On visit 3, points 5-15 from section 6.2.2 are repeated.

#### 6.2.4 End of study (Visit 4)

- The patient brings with them the remaining study medication which is gathered by the study nurse for a pill count. Clinical examinations are performed as listed in section 6.1.
- Points 6-11 from section 6.2.2 are repeated.
- B-SIT is performed by either the study nurse or investigator (see flowchart in section 6.1).
- At the end of the study visit, consider changes in the dopaminergic treatment.

#### 6.3 Criteria for Patient Discontinuation

Patients may be discontinued from study treatment and assessments at any time. Discontinuation and the reason for discontinuation (withdrawn from the study) will be registered. Specific reasons for discontinuing a patient for this study are:

- Voluntary discontinuation by the patient who is at any time free to discontinue his/her participation in the study, without prejudice to further treatment.
- Safety reasons as judged by the Principal Investigator.
- Incorrect enrolment, i.e., the patient does not meet the required inclusion/exclusion criteria for the study.
- Deterioration in the patient's condition which in the opinion of the Principal Investigator warrants study medication discontinuation (to be records as an AE or under Investigator Discretion).

#### 6.4 Procedures for Discontinuation

#### 6.4.1 Patient Discontinuation

Patients who are withdrawn from the study before the start of treatment will be replaced. Withdrawn patients are not followed up.

#### 6.4.2 Trial Discontinuation

The whole trial may be discontinued at the discretion of the PI or the sponsor in the event of any of the following:

- Occurrence of AEs unknown to date in respect of their nature, severity and duration.
- Medical or ethical reasons affecting the continued performance of the trial.
- Difficulties in the recruitment of patients.

The sponsor and principal investigator will inform all investigators and the Ethics Committees of the termination of the trial along with the reasons for such action. If the study is terminated early on grounds of safety and Ethics Committees will be informed within 15 days.
## 7 ASSESSMENTS

The schedule of assessments is indicated in Section 6 (see section 6.1, Flow Chart).

## 7.1 Safety and Tolerability Assessments

Safety will be monitored by AE registration at every visit. Significant findings that are present prior to the signing of informed consent must be included in the relevant medical history/ current medical condition page of the e-CRF. For details on AE collection and reporting, refer to Section 8.

#### 7.2 Clinical Assessments

#### 1. Medical history:

Performed by: investigator

- a. Family history of neurological illness:
  - i. Who
  - ii. Which illness.
- b. Family history of PD:
  - i. Who
  - ii. Was the diagnosis certain, probable or possible
- c. Smoking history:
  - i. Active smoker, previous smoker, or never smoker?
  - ii. Cigarettes smoked daily (on average)
  - iii. Duration of smoking (years)
  - iv. Pack-years (pack-years = cigarettes smoked daily / 20 x years of smoking)
- d. First PD symptoms:
  - i. Which symptoms: tremor, bradykinesia, gait abnormality, rigidity, loss of smell, other (if other = free text comment).
  - ii. History of REM sleep behavior disorder (RBD)
    - 1. RBD: yes/no
    - 2. If yes duration (i.e., for how long has the subject had it)
- e. Presence and duration of olfactory changes:
  - i. Complete loss of smell: yes/no?
  - ii. Decreased sense of smell?
  - iii. If yes duration (i.e., for how long has the subject had it)

#### 2. Vital signs:

Performed by: study nurse

- a. Blood pressure.
- b. Pulse.
- c. Temperature.

## 3. Body metrics:

Performed by: study nurse

- a. Body weight.
- b. Height.
- c. BMI.

#### 4. Physical examination:

#### Performed by: investigator

- a. Heart and lung auscultation.
  - i. Heart: normal / findings (free field)
  - ii. Lungs: normal / findings (free field)
- b. Abdominal palpation: normal / findings (free field)
- c. Any other examination dictated by patient's condition/symptoms: free field.

#### 5. General neurological examination

Performed by: investigator

a. Register any findings not related to the subject's parkinsonism: free field.

#### 6. Clinical scales & registrations:

Performed by: see individual tests below

a. MDS CDC:

Performed by: investigator

- b. MDS-UPDRS I-IV
  - i. NB! The exact time MDS-UPDRS is assessed must be registered in the eCRF. Performed by: section 1&2 by study nurse/investigator, section 3&4 by investigator
- c. MDS-NMS:

Performed by: Investigator or study nurse

d. MoCA:

Performed by: study nurse

e. EQ-5L:

Performed by: study nurse

f. GIDS-PD:

Performed by: study nurse

g. 3-day dietary record:

Performed by: self-filled by the patient

## 7.3 Routine Laboratory Tests

These will include: CRP, ALAT, ASAT, GT, bilirubin, ALP, creatinine, urea, RBC, Hb, WBC with differential, platelets, CK, FT4, TSH, B12, folic acid, homocysteine, methylmalonic acid, sodium, potassium, glucose. Women of childbearing potential will also have a pregnancy test performed.

Laboratory tests and biosampling are listed and described in detail in Appendix A.

## 7.4 Imaging studies

- **1. DAT-scan**, performed according to standard clinical routine, will confirm the presence of nigrostriatal degeneration.
- 2. 31P-MRS (CSI, multinuclear coil 15 min) will be conducted on a 3T Biograph mMR MR-PET scanner (Siemens Healthcare, Germany) to assess the intracerebral concentration of NAD, as we have done before (Fig 1A-C).
- **3. FDG-PET** imaging will be performed on the same MR-PET scanner and in the same session, to assess the metabolic response to NR treatment, as we have previously shown (Fig 1D-E). Following standard preprocessing protocols and spatial normalization, the NRRP will be assessed using ordinal trends/canonical variates analysis (OrT/CVA), a supervised form of principal component analysis (PCA)33. This multivariate approach is designed to detect and quantify regional covariance patterns

(i.e., metabolic networks) for which expression values (i.e., subject scores) increase or decrease with treatment in all or most of the subjects 34–38.

The MRI protocol is also summarized in Appendix B.

## 7.5 Molecular analyses

- 1) Metabolomics analyses will be performed in snap-frozen blood, PBMC, and CSF, using liquid chromatography-mass spectrometry (LC-MS) as described<sup>44</sup>. Absolute metabolite concentrations will be determined using in house standards. We will assess the entire NAD-metabolome, and key-metabolites involved in the Krebs' cycle, fatty acid beta-oxidation, and methylation reactions (e.g., SAM, homocysteine, folate).
- **2) Gene and protein expression.** The transcriptome will be mapped in PBMC and/or PAXgene samples by RNA-sequencing, using ribosomal depletion and sequencing at 125 bp paired-end and 100 million read pairs per sample, as we have previously described<sup>45</sup>. Quantitative proteomics will be performed in PBMC, muscle and CSF, using TMT (Tandem Mass Tags) labeling and mass spectrometry (LC-MS/MS Q-Exactive HF).
- **3) Histone acetylation profiling**. As in our previous work<sup>12</sup>, we will first assess quantitative changes in global histone acetylation status in PBMC and muscle, by immunoblotting with a pan-acetyl-lysin antibody. Next, acetylation levels of specific lysine residues (e.g., H3K27 and H4K16) will be assessed with targeted immunoblotting. Finally, genome-wide changes in the acetylation status of histone lysine residues found to be quantitatively altered by the treatment, will be assessed by chromatin-immunoprecipitation sequencing (ChIP-Seq)<sup>12</sup>.
- 4) Inflammatory cytokine concentration will be determined in CSF using ELISA as in the NADPARK trial<sup>18</sup>.
- **5) DNA methylation** will be mapped in PBMC and/or snap-frozen blood using the Illumina Infinium Epic Chip.
- 6) Neurotransmitter levels. Monoamine levels will be determined in the CSF using HPLC-MS.
- **7) Gut microbiome.** Using fecal samples, we will assess the microbiota profile (i.e., estimates of composition and abundance) by metagenomics, and function by microbial metabolomics. Metagenomics analyses will comprise 16S-rRNA sequencing-based count of operational taxonomic units (OTUs), Illumina NovaSeq short-read sequencing, and long-read sequencing by MinION technology. For microbial metabolomics, feces will be analyzed for short-chained fatty acids (SCFA) and, if feasible, NAD-related metabolites.

## 8 SAFETY MONITORING AND REPORTING

The investigator is responsible for the detection and documentation of events meeting the criteria and definition of an adverse event (AE) or serious adverse event (SAE). Each patient will be instructed to contact the investigator immediately should they manifest any signs or symptoms they perceive as serious. The methods for collection of safety data are described below.

## 8.1 Definitions

#### 8.1.1 Adverse Event (AE)

An AE is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not related to the investigational product.

The term AE is used to include both serious and non-serious AEs.

If an abnormal laboratory value/vital sign is associated with clinical signs and symptoms, the sign/symptom should be reported as an AE and the associated laboratory result/vital sign should be considered as additional information that must be collected on the relevant CRF.

Only intensity 2 and 3 is registered as AE in eCRF, see section 8.3. An AE has to interfere with everyday life to be of intensity 2 or 3.

#### 8.1.2 Serious Adverse Event (SAE)

Any untoward medical occurrence that at any dose:

- Results in death
- Is immediately life-threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability or incapacity
- Is a congenital abnormality or birth defect
- Is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.

Medical and scientific judgment is to be exercised in deciding on the seriousness of a case. Important medical events may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the subject or may require intervention to prevent one of the listed outcomes in the definitions above. In such situations, or in doubtful cases, the case should be considered as serious. Hospitalization for administrative reasons (for observation or social reasons) is allowed at the investigator's discretion and will not qualify as serious unless there is an associated adverse event warranting hospitalization.

## 8.2 Time Period for Reporting AE and SAE

Recording AE and SAEs will begin after baseline (week 0) and continue to be monitored and registered throughout the duration of the study up until 7 days after last study visit.

During the course of the study all AEs and SAEs will be proactively followed up for each patient; events should be followed up to resolution, unless the event is considered by the investigator to be unlikely to resolve due to the underlying disease. Every effort should be made to obtain a resolution for all events, even if the events continue after discontinuation/study completion.

## 8.3 Recording of Adverse Events

If the patient has experienced adverse event(s), the investigator will record the following information in the e-CRF:

- The nature of the event(s) will be described by the investigator in precise standard medical terminology (i.e., not necessarily the exact words used by the patient).
- The duration of the event will be described in terms of event onset date and event ended data.

The intensity of the adverse event: Only intensity grade 2 and 3 is registered as AE in eCRF.

#### **Assessment of Intensity**

The investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to 1 of the following categories:

- **1. Mild**: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities, and or requires clinical or diagnostic observations.
- **2. Moderate**: An event that causes sufficient discomfort to interfere with normal everyday activities, and or requires medical intervention.
- **3. Severe**: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both AEs and SAEs can be assessed as severe.

The Causal relationship of the event to the study medication will be assessed as one of the following:

- Unrelated: There is not a temporal relationship to investigational product administration (too early, or late, or investigational product not taken), or there is a reasonable causal relationship between non-investigational product, concurrent disease, or circumstance and the AE.
- Unlikely: There is a temporal relationship to investigational product administration, but there
  is not a reasonable causal relationship between the investigational product and the AE.
- Possible: There is reasonable causal relationship between the investigational product and the AE. Dechallenge information is lacking or unclear.
- o **Probable:** There is a reasonable causal relationship between the investigational product and the AE. The event responds to dechallenge. Rechallenge is not required.
- **Definite:** There is a reasonable causal relationship between the investigational product and the AE.
- It will be recorded in the eCRF the outcome of the adverse event, the action taken and whether the event is resolved or still ongoing.
- It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria in Section 8.1. An AE of severe intensity need not necessarily be considered serious. For example, nausea that persists for several hours may be considered severe nausea, but is not an SAE. On the other hand, a stroke that results in only a limited degree of disability may be considered a mild stroke, but would be an SAE.

## 8.4 Reporting Procedure

## 8.4.1 AEs and SAEs

All adverse events and serious adverse events that should be reported as defined in section 8.1.1 will be recorded in the patient's CRF.

SAEs must be reported by the investigator to the sponsor, (coordinating investigator: Haakon Berven or PI Charalampos Tzoulis, see contact information) within 24 hours after the site has gained knowledge of the SAE. Every SAE must be documented by the investigator on the SAE pages to be found in e-CRF. The initial report shall promptly be followed by detailed, written reports if necessary. The initial and follow-up reports shall identify the trial subjects by unique code numbers assigned to the latter.

The sponsor keeps detailed records of all SAEs reported by the investigators and performs an evaluation with respect to seriousness, causality and expectedness.

## 8.5 Clinical Study Report

The adverse events and serious adverse events occurring during the study will be discussed in both the main results and the safety evaluation part of the Clinical Study Report.

#### 9 DATA MANAGEMENT AND MONITORING

## 9.1 Electronic - Case Report Forms (e-CRFs)

The study nurse/investigator will enter the data required by the protocol into the electronic Case report forms (e-CRF) online. The electronical CRF that will be used is Viedoc. The Investigator is responsible for assuring that data entered into the e-CRF for his/her patient is complete, accurate, and that entry is performed in a timely manner. The signature of the investigator will attest to the accuracy of the data on each CRF. If any assessments are omitted, the reason for such omissions will be noted on the e-CRFs.

At study visit the following source date should be registered either on paper or hospital records. See section 6.1 and 6.2 for when the relevant information is gathered. This data will then be transferred to eCRF by the study nurse/investigator.

- That the patient is participating in the study, e.g., by including the enrollment number and the study code or other such study identification
- Date when Informed Consent was obtained from the patient and statement that patient received a copy of the signed and dated Informed Consent
- Results of all assessments confirming a patient's eligibility for the study
- Diseases (relevant past and current with date; both the disease studied and others, as relevant)
- Medical history
- Laboratory data
- Results of clinical assessments performed during the study
- Treatment given
- Non-Serious Adverse Events and Serious Adverse Events (if any) including causality assessments
- Date of, and reason for, discontinuation from study treatment
- Date of, and reason for, withdrawal from study

## 9.2 Study Monitoring

The investigator will be visited on a regular basis by the Clinical Study Monitor, who will check the following:

- Informed consent process
- Reporting of adverse events and all other safety data

- Adherence to protocol
- Maintenance of required regulatory documents
- Study Supply accountability log
- Data completion on the e-CRFs including source data verification (SDV).

The monitor will review the relevant e-CRFs for accuracy and completeness and will ask the site staff to adjust any discrepancies as required.

When the responsible study monitor has checked and verified the e-CRFs, the data will be entered into a computer database at the Haukeland University hospital scientific server for further handling and statistical evaluation.

Sponsor's representatives (e.g., monitors, auditors) and/or competent authorities will be allowed access to source data for source data verification in which case a review of those parts of the hospital records relevant to the study may be required.

## 9.3 Confidentiality

The investigator shall arrange for the secure retention of the patient identification and the code list. Patient files shall be kept for the maximum period of time permitted by the hospital. The study documentation (e-CRFs, Site File etc) shall be retained and stored during the study and for 5 years after study closure. All information concerning the study will be stored in a safe place inaccessible to unauthorized personnel.

#### 9.4 Database management

- Access to study after the study completion is granted by Charalampos Tzoulis.
- Data for each patient will be recorded on the eCRF. Data collection must be completed for each patient who signs an informed consent form and receives at least one dose of study treatment.
- eCRFs will be designed and produced by the Investigator and should be completed in accordance with instructions. The Investigator is responsible for maintaining adequate and accurate medical records from which accurate information will be transcribed directly into the eCRFs using a secure internet connection. The eCRFs should be filled out completely by the Investigator or designee as stated on the delegation of responsibilities form.
- The eCRFs must be reviewed, signed and dated by the Investigator.
- Data entered into the eCRF will be validated as defined in the data validation plan. Validation includes, but is not limited to, validity checks (e.g., range checks), consistency checks and customized checks (logical checks between variables to ensure that study data are accurately reported) for eCRF data and external data (e.g., laboratory data). A majority of edit checks will be triggered during data entry and will therefore facilitate efficient 'point of entry' data cleaning.
- Data management personnel will perform both manual eCRF review and review of additional
  electronic edit checks to ensure that the data are complete, consistent and reasonable. The
  electronic edit checks will run continually throughout the course of the study and the issues will
  be reviewed manually online to determine what action needs to be taken.
- Manual queries may be added to the system by clinical data management or study monitor.
   Clinical data managers and study monitors are able to remotely and proactively monitor the patient eCRFs to improve data quality.
- Pharmacokinetic data will be transferred electronically into the study database. Discrepancies

will be queried to the site and/or the laboratory until the electronic data and the database are reconciled.

- All updates to queried data will be made by authorized study center personnel only and all
  modifications to the database will be recorded in an audit trail. Once all the queries have been
  resolved, eCRFs will be locked by password protection. Any changes to locked eCRFs will be
  approved by the Investigator.
- Once the full set of eCRFs have been completed and locked, the Sponsor will authorize database lock and all electronic data will be sent to the designated statistician for analysis. Subsequent changes to the database will then be made only by written agreement.
- Adverse events and medical history will be coded from the verbatim description (Investigator term). Prior and concomitant medications and therapies will be coded according to the World Health Organization drug code.

#### 10 STATISTICAL METHODS AND DATA ANALYSIS

## 10.1 Determination of Sample Size

Our primary null hypothesis ( $H_0$ ) is that the NR-induced increases in cerebral NAD levels (measured by 31P-MRS) are not dose-responsive. The alternative hypothesis ( $H_A$ ) is that this measure is dose responsive. In the NADPARK study, all three measures showed a highly significant increase in the group receiving 1000 mg NR (n=15) compared to the placebo group (n=15). In the NADPARK study<sup>46</sup>, treatment with 1000mg of NR led to an increase in cerebral NAD-levels by a factor of 1.27 from baseline in the treatment group, whereas the change in the placebo group was negligible at -0.43%. Under the  $H_A$ , we assume that cerebral NAD levels will increase in a linear fashion in the 2000 mg NR and 3000 mg NR groups, respectively. Based on these assumptions and given a type I error rate of 5% ( $\alpha$  = 0.05) and a type II error rate of 10% ( $\beta$  = 0.1, power = 90%), we estimated that a sample size of 30 individuals will be required in the dose escalation group. Accounting for drop-out and statistical safety margin, we estimate that the study requires 40 subjects in this group.

For the secondary and exploratory outcomes, we assume that the metabolomic, transcriptomic and inflammatory cytokine analyses will have sufficient power, since they produced very large effect sizes and highly significant results in the NADPARK study with 15 individuals per group. Since no pilot data exists for the proteomic and epigenomic analyses, these will be exploratory in nature. However, in our previous experience, a sample size of 20 per group should be sufficient to detect treatment-induced differences of biological relevance.

#### 10.2 Randomization

Randomization is done by e-CRF upon enrollment to the study. Participants will be randomized into one of three groups (Placebo, NR 1000 mg for the duration of the study, NR dose escalation group).

## 10.3 Population for Analysis

Intention to treat (ITT)/Full analysis set (FAS) population: All participants, regardless of protocol adherence.

The Safety Analysis Set (SAS) will include all patients having received at least one study treatment infusion after randomisation.

The Per Protocol Analysis Set (PPS) will include all randomized patients meeting the study eligibility criteria and with no major protocol deviations affecting the treatment efficacy.

The following are pre-defined major protocol deviations regarded to affect the efficacy of the intervention:

- Entering the trial when the eligibility criteria should have prevented trial entry.
- Discontinuation of intervention prior to 84 ± 7 days.
- Major change in concomitant anti-Parkinson medication.
- Received or used other intervention than allocated.
- Adherence to allocated treatment below 85%.
- Visit date interval larger than 28 ± 7 days between individual visits (i.e.: V1 and V2, V2 and V3 and V3 and V4)\*.
- Visit date interval larger than 84 ± 7 days from V1 to V4\*.
- Not fasting before neuroimaging.

\*Due to updated findings from a pharmacokinetic study (ClinicalTrials.gov, NCT: NCT05698771, in revision) that NAD levels increase and reach a plateau within 1-2 weeks of NR treatment both in healthy individuals and persons with Parkinson's disease. A 3 week period should therefore be sufficient to assess the effects of increasing NR dosage.

## 10.4 Planned analyses

All statistical analyses will take place after the completion of the study. All randomized patients will be included in the primary analyses and sensitivity analyses will be carried out comparing results from the ITT, SAS and PPS data sets. In the case of missing assessments, the subject will be included if possible.

The *primary analysis* of the primary endpoint will be performed using analysis of covariance (ANCOVA) between the dose stable (DS-group) and dose escalation group (DS-group), i.e. the regression of NAD levels measured by <sup>31</sup>P-MRS at week 12 depending on randomization group and adjusted for <sup>31</sup>P-MRS at baseline. No additional adjustments/covariates will be used. As this is the single primary outcome, alpha will be set at 0.05. No correction for multiple testing will be performed.

The *secondary analysis* of the primary endpoint will be the comparison of change over time from baseline to week 4, week 8 and week 12, between the DE-group and the DS-group. This will be assessed using a linear mixed model (LME), i.e. NAD (<sup>31</sup>P-MRS) at weeks 4,8 and 12 depending on randomization group, time and their interaction adjusted for random individual intercept.

The *primary analysis* of the secondary endpoint will be performed using ANCOVA between the dose stable (DS-group) and dose escalation group (DS-group), i.e. the regression of NAD or NAD metabolite levels measured by HPLC-MS at week 12 depending on randomization group and adjusted for NAD or NAD metabolite at baseline. No additional adjustments/covariates will be used.

The analysis of exploratory endpoints will be performed in a similar manner as for the primary and secondary endpoints. ANCOVA will be used to compare endpoints at week 12, and LME will be used to compare change from baseline to week 4, week 8 and week 12.

In addition, for PET analyses, changes in network scores with treatment will be evaluated for each group separately using permutation tests. Relationships between network values, brain NAD levels and MDS-UPDRS motor ratings or between treatment-related changes in these variables will be evaluated using Pearson's product-moment correlations, whereas Spearman rank-order correlation coefficients will be computed for non-normally distributed variables.

Omics data will undergo rigorous quality control and filtering according to established best practice procedures, as we have previously described 12,45,47,48. The between visit change in this data will be assessed by a pairwise comparison between each NR group and the placebo group, using linear models with appropriate covariates as we have previously described 12,45,47,48. Comparison of adverse events and abnormal laboratory test results between the treatment and placebo groups will be analyzed descriptively.

Further details for the analysis are outlined in the statistical analysis plan (SAP) for the trial, and we refer the reader to this document.

## **10.5** Statistical Analysis

#### Dependent variable

Primary analysis:

Cerebral NAD levels (measured by <sup>31</sup>P-MRS)

Secondary, exploratory and safety analyses:

- Adverse events, categorized as either moderate or severe.
- Levels of CSF NAD and NAD-metabolites (measured by LC-MS).
- Levels of NRRP expression (measured by FDG-PET)
- Levels of PDRP expression (measured by FDG-PET)
- Routine blood tests
- Total MDS-UPDRS
- MDS-UPDRS Part I
- MDS-UPDRS Part II
- MDS-UPDRS Part III
- MDS-UPDRS Part IV
- MDS-NMS
- MoCA
- GIDS-PD
- EQ-5D-5L
- Levels of NAD-related and other metabolites in PBMC, frozen blood, urine and CSF
- Expression of RNA and protein of genes and pathways involved in proteasomal and lysosomal biogenesis and function.
- Histone panacetylation levels
- Levels of specific lysine residues H3K27 and H4K16 acetylation

- Genome-wide distribution of histone lysine residues found to be quantitatively altered by the treatment (measured by ChIP-Seq).
- Level of inflammatory cytokines in patient serum and CSF.
- Gene and protein expression levels in PAXgene blood.
- Levels of one carbon metabolism metabolites, measured by HPLC-MS metabolomics in PBMC and CSF.
- Levels of monoamine neurotransmitters in CSF.
- Levels and genomic distribution of DNA methylation.
- Gut microbiome composition.
- Fecal metabolomics, including fatty acid levels.
- Sense of smell, measured by B-SIT.

#### Statistical hypothesis

#### Primary analysis:

- Our primary null hypothesis (H<sub>0</sub>) is that the NR-induced increases in cerebral NAD levels (measured by <sup>31</sup>P-MRS) is not dose-responsive. The alternative hypothesis (H<sub>A</sub>) is that this increase is dose responsive.

#### Secondary analysis:

- Mean change between the NR dose escalation arm and NR 1000 mg arm for the dependent variables mentioned above.
- Mean change between and within the NR dose escalation arm, NR 1000 mg arm and placebo arm for the dependent variables mentioned above.

## 11 STUDY MANAGEMENT

#### 11.1 Investigator Delegation Procedure

The principal investigator is responsible for making and updating a "delegation of tasks" listing all the involved co-workers and their role in the project. He will ensure that appropriate training relevant to the study is given to all of these staff, and that any new information of relevance to the performance of this study is forwarded to the staff involved.

#### 11.2 Protocol Adherence

Investigators ascertain they will apply due diligence to avoid protocol deviations.

All significant protocol deviations will be recorded and reported in the Case Report Form (CRF).

#### 11.3 Study Amendments

If it is necessary for the study protocol to be amended, the amendment and/or a new version of the study protocol (Amended Protocol) must be notified to and the Ethics Committee according to EU and national regulations.

#### 11.4 Audit and Inspections

Authorized representatives of the Ethics Committee may visit the center to perform inspections, including source data verification. Likewise, the representatives from the sponsor may visit the center to perform an audit. The purpose of an audit or inspection is to systematically and independently examine all study-

related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, Good Clinical Practice (ICH GCP), and any applicable regulatory requirements. The principal investigator will ensure that the inspectors and auditors will be provided with access to source data/documents.

## 12 ETHICAL AND REGULATORY REQUIREMENTS

The study will be conducted in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/Good Clinical Practice and applicable regulatory requirements. Registration of patient data will be carried out in accordance with national personal data laws.

#### 12.1 Ethics Committee Approval

Application to REK has been submitted. The investigator is responsible for informing the ethics committee of any serious and unexpected adverse events and/or major amendments to the protocol as per national requirements.

#### 12.2 Other Regulatory Approvals

Statens legemiddelverket (SLV)/Direktoratet for medisinske produkter (DMP) has deemed that the project is not a clinical trial due to the fact that NR is not classified as a drug, but as a nutritional supplement.

#### 12.3 Informed Consent Procedure

All subjects will be presented verbally and with written informed consent to be signed prior to enrollment to the study. The informed consent will be presented at the first screening. Informed consent will be handled according to GCP principles. A copy of the informed consent will be given to the subject.

#### 12.4 Subject Identification

Upon entry in screening, each subject is given a patient study number, this study number is used for the remainder of the study. The Patient study number is in the format XXYYY where XX is the study site number and YYY is the patient ID number.

The investigator is responsible for keeping a list of all patients (who have received study treatment or undergone any study specific procedure) including patient's date of birth and personal number, full names and last known addresses.

The patients will be identified in the CRFs by the patient study number and initials.

## 13 TRIAL SPONSORSHIP AND FINANCING

Research Council of Norway (RCN), Neuro-SysMed, (ES633272) 2020-2028

#### 14 TRIAL INSURANCE

The Patients are insured by the government through the "Norsk Pasientskade Erstatning" (NPE).

## 15 PUBLICATION POLICY

Upon study completion and finalization of the study report the results of this study will either be submitted for publication and/or posted in a publicly accessible database of clinical study results.

The results of this study will also be submitted to the Ethics Committee according to EU and national regulations.

All personnel who have contributed significantly with the planning and performance of the study (Vancouver convention 1988) may be included in the list of authors.

## 16 REFERENCES

- 1. de Rijk MC, Launer LJ, Berger K, et al. Prevalence of Parkinson's disease in Europe: A collaborative study of population-based cohorts. Neurologic Diseases in the Elderly Research Group. Neurology 2000;54(11 Suppl 5):S21-3.
- 2. Gooch CL, Pracht E, Borenstein AR. The burden of neurological disease in the United States: A summary report and call to action. Ann Neurol 2017;81(4):479–484.
- 3. Gustavsson A, Svensson M, Jacobi F, et al. Cost of disorders of the brain in Europe 2010. Eur Neuropsychopharmacol 2011;21(10):718–79.
- 4. Lautrup S, Sinclair DA, Mattson MP, Fang EF. NAD+ in Brain Aging and Neurodegenerative Disorders. Cell Metabolism 2019;30(4):630–655.
- 5. Katsyuba E, Romani M, Hofer D, Auwerx J. NAD+ homeostasis in health and disease. Nat Metab 2020;2(1):9–31.
- 6. Johnson S, Imai S. NAD + biosynthesis, aging, and disease [Internet]. F1000Res 2018;7[cited 2021 May 9 ] Available from: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5795269/
- 7. Braidy N, Liu Y. NAD+ therapy in age-related degenerative disorders: A benefit/risk analysis. Exp. Gerontol. 2020;132:110831.
- 8. Schapira AH, Cooper JM, Dexter D, et al. Mitochondrial complex I deficiency in Parkinson's disease. Lancet 1989;1(8649):1269.
- 9. Hattori N, Tanaka M, Ozawa T, Mizuno Y. Immunohistochemical studies on complexes I, II, III, and IV of mitochondria in Parkinson's disease. Ann. Neurol. 1991;30(4):563–571.
- 10. Flønes IH, Fernandez-Vizarra E, Lykouri M, et al. Neuronal complex I deficiency occurs throughout the Parkinson's disease brain, but is not associated with neurodegeneration or mitochondrial DNA damage. Acta Neuropathol 2018;135(3):409–425.
- 11. Hirsch EC, Hunot S. Neuroinflammation in Parkinson's disease: a target for neuroprotection? Lancet Neurol 2009;8(4):382–397.
- 12. Toker L, Tran GT, Sundaresan J, et al. Genome-wide histone acetylation analysis reveals altered transcriptional regulation in the Parkinson's disease brain. Molecular Neurodegeneration 2021;16(1):31.

- 13. Park G, Tan J, Garcia G, et al. Regulation of Histone Acetylation by Autophagy in Parkinson Disease. The Journal of biological chemistry 2016;291(7):3531–40.
- 14. Gonzalez-Hunt CP, Sanders LH. DNA damage and repair in Parkinson's disease: Recent advances and new opportunities. J Neurosci Res 2021;99(1):180–189.
- 15. Bieganowski P, Brenner C. Discoveries of nicotinamide riboside as a nutrient and conserved NRK genes establish a Preiss-Handler independent route to NAD+ in fungi and humans. Cell 2004;117(4):495–502.
- 16. Conze DB, Crespo-Barreto J, Kruger CL. Safety assessment of nicotinamide riboside, a form of vitamin B3. Hum Exp Toxicol 2016;35(11):1149–1160.
- 17. Dollerup OL, Christensen B, Svart M, et al. A randomized placebo-controlled clinical trial of nicotinamide riboside in obese men: safety, insulin-sensitivity, and lipid-mobilizing effects. Am. J. Clin. Nutr. 2018;108(2):343–353.
- 18. Brakedal B, Dölle C, Riemer F, et al. The NADPARK study: A randomized phase I trial of nicotinamide riboside supplementation in Parkinson's disease. Cell Metabolism 2022;34(3):396-407.e6.
- 19. Conze D, Brenner C, Kruger CL. Safety and Metabolism of Long-term Administration of NIAGEN (Nicotinamide Riboside Chloride) in a Randomized, Double-Blind, Placebo-controlled Clinical Trial of Healthy Overweight Adults. Sci Rep 2019;9(1):9772.
- 20. EFSA Panel on Nutrition. European Food Safety Authority Safety of nicotinamide riboside chloride [Internet]. 2019.Available from: http://www.efsa.europa.eu/en/efsajournal/pub/5775
- Haukeland University Hospital. NR-SAFE: a Safety Study Investigating Treatment With High-dose Nicotinamide Riboside (NR) in Parkinson's Disease [Internet]. clinicaltrials.gov; 2022.[cited 2022 Jul 28] Available from: https://clinicaltrials.gov/ct2/show/NCT05344404
- 22. Trammell SA, Schmidt MS, Weidemann BJ, et al. Nicotinamide riboside is uniquely and orally bioavailable in mice and humans. Nat Commun 2016;7:12948.
- 23. Martens CR, Denman BA, Mazzo MR, et al. Chronic nicotinamide riboside supplementation is well-tolerated and elevates NAD+ in healthy middle-aged and older adults. Nat Commun 2018;9(1):1286.
- 24. Elhassan YS, Kluckova K, Fletcher RS, et al. Nicotinamide Riboside Augments the Aged Human Skeletal Muscle NAD+ Metabolome and Induces Transcriptomic and Anti-inflammatory Signatures. Cell Rep 2019;28(7):1717-1728.e6.
- 25. Okur MN, Mao B, Kimura R, et al. Short-term NAD+ supplementation prevents hearing loss in mouse models of Cockayne syndrome. NPJ Aging Mech Dis 2020;6:1.
- 26. Brown KD, Maqsood S, Huang JY, et al. Activation of SIRT3 by the NAD(+) precursor nicotinamide riboside protects from noise-induced hearing loss. Cell Metab 2014;20(6):1059–68.
- 27. Han S, Du Z, Liu K, Gong S. Nicotinamide riboside protects noise-induced hearing loss by recovering the hair cell ribbon synapses. Neurosci. Lett. 2020;725:134910.
- 28. Harlan BA, Killoy KM, Pehar M, et al. Evaluation of the NAD+ biosynthetic pathway in ALS patients and effect of modulating NAD+ levels in hSOD1-linked ALS mouse models. Exp. Neurol. 2020;327:113219.

- 29. Sorrentino V, Romani M, Mouchiroud L, et al. Enhancing mitochondrial proteostasis reduces amyloid-β proteotoxicity. Nature 2017;552(7684):187–193.
- 30. Xie X, Gao Y, Zeng M, et al. Nicotinamide ribose ameliorates cognitive impairment of aged and Alzheimer's disease model mice. Metab Brain Dis 2019;34(1):353–366.
- 31. Schöndorf DC, Ivanyuk D, Baden P, et al. The NAD+ Precursor Nicotinamide Riboside Rescues Mitochondrial Defects and Neuronal Loss in iPSC and Fly Models of Parkinson's Disease. Cell Rep 2018;23(10):2976–2988.
- 32. Haukeland University Hospital. NAD-PARK: A Double-blinded Randomized Pilot Trial of NAD-supplementation in Drug naïve Parkinson's Disease [Internet]. clinicaltrials.gov; 2020.[cited 2021 Mar 18] Available from: https://clinicaltrials.gov/ct2/show/NCT03816020
- 33. Hirano S, Eckert T, Flanagan T, Eidelberg D. Metabolic Networks for Assessment of Therapy and Diagnosis in Parkinson's Disease. Mov Disord 2009;24(0 2):S725–S731.
- 34. Bloem BR, Okun MS, Klein C. Parkinson's disease [Internet]. The Lancet 2021;0(0)[cited 2021 Apr 17 ] Available from: https://www.thelancet.com/journals/lancet/article/PIIS0140-6736(21)00218-X/abstract
- 35. Jadavji NM, Wieske F, Dirnagl U, Winter C. Methylenetetrahydrofolate reductase deficiency alters levels of glutamate and γ-aminobutyric acid in brain tissue. Mol Genet Metab Rep 2015;3:1–4.
- 36. Romano S, Savva GM, Bedarf JR, et al. Meta-analysis of the Parkinson's disease gut microbiome suggests alterations linked to intestinal inflammation. npj Parkinsons Dis. 2021;7(1):1–13.
- 37. Payne T, Appleby M, Buckley E, et al. A Double-Blind, Randomized, Placebo-Controlled Trial of Ursodeoxycholic Acid (UDCA) in Parkinson's Disease. Movement Disorders 2023;38(8):1493–1502.
- 38. Chaudhuri KR, Schrag A, Weintraub D, et al. The Movement Disorder Society Nonmotor Rating Scale: Initial Validation Study. Mov Disord 2020;35(1):116–133.
- 39. Goetz CG, Tilley BC, Shaftman SR, et al. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Scale presentation and clinimetric testing results: MDS-UPDRS: Clinimetric Assessment. Mov. Disord. 2008;23(15):2129–2170.
- 40. Camacho M, Greenland JC, Williams-Gray CH. The Gastrointestinal Dysfunction Scale for Parkinson's Disease. Mov Disord 2021;36(10):2358–2366.
- 41. Nasreddine ZS, Phillips NA, Bédirian V, et al. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc 2005;53(4):695–699.
- 42. Janssen MF, Bonsel GJ, Luo N. Is EQ-5D-5L Better Than EQ-5D-3L? A Head-to-Head Comparison of Descriptive Systems and Value Sets from Seven Countries. Pharmacoeconomics 2018;36(6):675–697.
- 43. Postuma RB, Berg D, Stern M, et al. MDS clinical diagnostic criteria for Parkinson's disease. Movement disorders: official journal of the Movement Disorder Society 2015;30(12):1591–601.
- 44. Trammell SA, Brenner C. Targeted, LCMS-based Metabolomics for Quantitative Measurement of NAD(+) Metabolites. Computational and structural biotechnology journal 2013;4:e201301012.

- 45. Nido GS, Dick F, Toker L, et al. Common gene expression signatures in Parkinson's disease are driven by changes in cell composition. Acta Neuropathol Commun 2020;8(1):55.
- 46. Brakedal B, Dölle C, Riemer F, et al. The NADPARK study: A randomized phase I trial of nicotinamide riboside supplementation in Parkinson's disease. Cell Metab 2022;34(3):396-407.e6.
- 47. Dick F, Nido GS, Alves GW, et al. Differential transcript usage in the Parkinson's disease brain [Internet]. PLoS Genet 2020;16(11)[cited 2020 Nov 29 ] Available from: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7660910/
- 48. Dick F, Tysnes O-B, Alves GW, et al. Altered transcriptome-proteome coupling indicates aberrant proteostasis in Parkinson's disease. medRxiv 2021;2021.03.18.21253875.
- 49. Ladefoged CN, Hansen AE, Henriksen OM, et al. Al-driven attenuation correction for brain PET/MRI: Clinical evaluation of a dementia cohort and importance of the training group size. Neuroimage 2020;222:117221.

## 17 LIST OF APPENDICES

- A. Lab Manual
- B. Imaging Manual
- C. Clinical Rating Scales

## **APPENDIX A**

## LABORATORY MANUAL FOR N-DOSE

Helse Bergen, Haukeland University Hospital

| <b>Protocol:</b><br>N-DOSE | | | | | | | |
|---|---|---|---|---|---|---|---|
| REK Numb | er: | | | | | | |
| | | randomized,<br>ide in Parkinso | • | dose | optimization | trial | of |

STANDARD OPERATING PROCEDURE (SOP) FOR SAMPLING AND PREPARATION OF BIOLOGICAL MATERIAL (LAB MANUAL)

Project Management Committee for the study

**Charalampos Tzoulis** 

Haakon Berven

## 1 GENERAL INFORMATION

The purpose of this document is to give an overview of the biological material collected for biobanking in the N-DOSE clinical trial. At different time points during the clinical trial the following biological samples are collected, processed and stored based on standard operating procedures: whole blood, serum, plasma, PBMCs, blood cells. The samples are stored at Biobank Haukeland and at the Neuro-SysMed Center.

In the following chapters you will find a detailed description of how to collect, prepare, and store samples at HUS. It is critically important that the samples are prepared correctly and standardized, and that all deviations from the protocol are documented. This information will be registered in LabVantage when the Biobank Information system is in operation and at the Neuro-SysMed Center.

# 2 HEMATOLOGY, BIOCHEMISTRY, HORMONE, SEROLOGY AND SAFETY LABORATORY PARAMETERS

This chapter describes the biological material that should be collected for hematology, biochemistry, hormone and serology analyses and for serum hCG pregnancy test. The collection should be done as specified in the Flow Chart. The local study site laboratory will be used for the analyses of these components, as indicated in the Study Protocol. Protocols for collection of biological material for research and biobanking are described in Chapter 3 and 4.

| Flow chart | | | | | TUBES |
|---|---|---|---|---|---|
| Visits | V1 /<br>Baseline | V2 | V3 | V4 | |
| Week | 0 | 4 | 8 | 12 | |
| Routine: | | | | | |
| hCG <sup>1</sup> | Х | | | | |
| CRP | Х | Х | Х | Х | |
| ALAT | Х | Х | Х | Х | |
| ASAT | Х | х | Х | Х | |
| GT | Х | х | Х | Х | |
| Bilirubin | Х | х | Х | Х | |
| ALP | Х | х | Х | Х | |
| Creatinine | Х | Х | Х | Х | |
| Urea | Х | х | Х | Х | |
| RBC | Х | х | Х | Х | |
| Hb | Х | х | Х | Х | |
| WBC with differential | х | х | Х | Х | |
| Platelets | х | х | Х | Х | |
| CK | Х | х | Х | Х | |
| FT4 | Х | Х | Х | Х | |
| TSH | Х | Х | Х | Х | |
| B12 | Х | Х | Х | Х | |
| Folic acid | Х | Х | Х | Х | |
| homocysteine | Х | Х | Х | Х | |
| Methylmalonic acid | х | х | Х | Х | |
| Sodium | Х | Х | Х | Х | |
| Potassium | Х | Х | Х | Х | |
| Glucose | Х | Х | Х | Х | |
| Biobank: | | | | | |
| EDTA whole blood | х | | | | FluidX, 0,7ml, 8 aliquotes |
| Snap-frozen whole blood | х | Х | Х | Х | |
| PAXgene blood for RNA | х | Х | Х | Х | PAXgene tubes |
| Platelets | х | Х | Х | Х | |
| Serum | х | Х | Х | Х | FluidX, 0,7ml, 8 aliquotes |
| Fecal sample | х | | | Х | |
| Urine sample | х | Х | Х | Х | |
| Cerebrospinal fluid | Х | | | Х | |

#### 2.1.1 Safety laboratory (blood)

All safety laboratory parameters will be collected at the timepoints as indicated in the Flow Chart (page 47), and include hematology, liver enzymes/parameters, clinical chemistry, thyroid status. The samples will be analyzed at the local laboratory at the study site. The respective reference ranges must be provided to the central study administration for uploading into the eCRF.

#### 3 SAMPLING FOR BIOBANK AND RESEARCH

## 3.1 Mandatory research and biobank samples

Chapter 3.1 gives an overview of all mandatory samples collected for research and biobanking. The sample processing protocols are in Chapter 4.

#### 3.1.1 Whole blood EDTA

EDTA blood will be collected at HUS

#### 3.1.2 Whole blood EDTA – snap-frozen

Snap-frozen EDTA blood will be collected at HUS

#### 3.1.3 RNA PAXgene tubes

Blood in PAXgene tubes for RNA extraction will be collected at HUS

#### 3.1.4 Whole blood for Serum

Serum will be collected at HUS

#### 3.1.5 Platelets

Platelets will be collected at HUS

#### 3.1.6 Cerebrospinal fluid (CSF)

CSF will be collected at HUS

#### 3.1.7 Feces

Feces will be collected at HUS

## 3.1.8 Urine

Urine will be collected at HUS

#### 4 SAMPLE PROCESSING AND STORAGE

## 4.1 Whole blood (EDTA): standard

Performed at: HUS

#### Material and instrumentation:

| Item | How many | Supplier | Cat no | Comment |
|---|---|---|---|---|
| VACUETTE® TUBE 2 ml K2E K2EDTA | 2 | Greiner Bio-One<br>International | 454024 | |
| 0.7 ml FluidX tubes | 8 | Pedro Consulting | 68-0702-<br>11N | |
| Pipettes & tips | | | | |
| Barcode reader | | | | |
| -80°C freezer | | Study center | | |

#### Collection, preparation and storage:

- 1. Collect whole blood into Vacuette tubes for EDTA blood
- 2. Aliquot 500  $\mu$ L blood into 8 x 0.7 ml FluidX tubes.
- 3. Freeze the aliquots at -80°C within 60 min after sample collection.
- 4. Use the barcode reader for registration of the sample and log all deviations on the same registration form.
- 5. Sample aliquots are stored at -80C and shipped on dry ice in the original FluidX boxes (x 48 tubes).
- Samples must <u>never</u> be allowed to warm or thaw except from when to be used in analyses.
   Any deviation from this must be <u>registered</u>. The number and date of thawing an aliquot for analyses must be registered.

Contact person for biosampling and laboratory preparation: Siri Hinteregger, MBF

Contact person for Biobank:

Hilde Kristin Garberg



FluidX tubes box (x48)



FluidX tubes

## 4.2 Whole blood (EDTA): snap-frozen

#### Performed at: HUS

Snap-frozen whole blood will be used for the analysis of NAD+. NAD degrades very rapidly after sample collection and the concern is that measurements in any sample that requires extensive processing may not prove reliable.

#### Material and instrumentation:

| Item | How many | Supplier | Cat no | Comment |
|---|---|---|---|---|
| VACUETTE® TUBE 2 ml K2E K2EDTA | 1 | Greiner Bio-One | 454024 | |
| | | International | | |
| Screw cap micro tubes, 0.5 ml, | 8 | Sarstedt | 72.730.006 | |
| sterile | | | | |
| Multi dispenser pipette & tips | | | | |
| Liquid nitrogen in a thermos | | | | |
| -80°C freezer | | Study center | | |
| Timer | | | | |

## NB! The time from blood drawing (i.e. moment the blood starts flowing into the tube) and freezing MUST be 2 min!

#### Collection, preparation and storage:

- 1. Print labels. For one patient: 8x
- 2. Mark 8 x 0.5 ml micro tubes with labels
- 3. Laboratory technician must be next to the patient at the blood drawing with all equipment ready.
- 4. Laboratory technicians must wear gloves and a lab coat.
- 5. Collect whole blood into the Vacuette tube.
- 6. **START THE TIMER** when blood starts flowing into the tube.
- 7. Gently invert the EDTA tube at least 10 times. **DO NOT SHAKE**
- 8. Aliquot 8 x 200  $\mu$ l of blood from the 2 ml EDTA tube into 8 x 0.5 ml micro tubes (easiest using a multi dispenser pipette).
- 9. Close micro tubes
- 10. When the timer shows 2min: immerse all the micro tubes simultaneously in liquid nitrogen.
- 11. Transfer the frozen EDTA-aliquots -80°C freezer for storage.
- 12. Sample aliquots are stored at -80C in freezer-compatible cardboard or plastic storage boxes.
- 13. Samples are shipped on dry ice.
- 14. Samples must <u>never</u> be allowed to warm or thaw except from when to be used in analyses. Any deviation from this must be <u>registered</u>. The number and date of thawing an aliquot for analyses must be registered.

If the 2 min interval is not respected - still collect the samples but register the time interval.

Responsible: Hanne Linda Nakkestad

## 4.3 RNA PAXgene tubes

#### Performed at: HUS

#### Rationale:

The Paxgene Blood RNA collection system is intended for the purification of intracellular RNA from whole blood and is optimized for the stabilization of 4.8  $\times$ 10e6 – 1.1  $\times$  10e7 leukocytes/ml. This protocol describes the collection of whole blood in Paxgene RNA tubes from Qiagen for long-term storage at -80° C.

Important: Paxgene collection tubes **must** be at room temperature prior to collection. Follow standard procedure for venipuncture for tubes with stabilizing agents e.g., butterfly collection

#### Material and instrumentation:

- PAXgene blood RNA tubes (PreAnalytix, Cat. No. 762165)
- BD Vacutainer SafetyLok Blood collection set (BD, Cat. No. 367281) or similar
   Butterfly and safety lock or similar
- Sample labels capable of storage at -80 °C
- Phlebotomy materials: Tourniquet, alcohol swabs, gauze
- Barcode reader
- -80°C freezer

#### Collection, preparation, storage and shipment:

Before starting, ensure PAXgene tubes are at ambient temperature and labeled appropriately with temperature resistant labels. Draw PAXgene tubes last, after other blood tubes. If the PAXgene tubes are the only tubes, draw a small amount of blood into a discard tube.

- 1. Using the Blood Collection set, collect blood into the PAXgene tube using standard venipuncture techniques. Ensure that the donor's arm is in a downward position, and that the PAXgene tube is <a href="held vertically">held vertically</a> below the donor's arm.
- 2. Collect 2.5 ml of blood into each PAXgene tube. so that the tube gets filled with **exactly** 2.5 ml blood. This is essential so that the final concentration of the reagents will be correct. If PAXgene is the first sample to be taken, collect some blood in another tube first, to get rid of the air in the collection system, so that the PAXgene tube gets exactly 2.5 ml blood.
- 3. Allow at least 10 s for the blood draw to occur and ensure that blood has stopped flowing into the tube before removing the needle from the tube.
- 4. Immediately after blood collection mix the tube by gentle inversion (180°) 10 times
- 5. Temporarily store the PAXgene upright at RT for between **2-24 hrs**.
- 6. Temporarily store the PAXGene tube for at least 24 hrs at -20°C
- 7. After at least 24 hrs at -20°C, move the PAXgene tube for long-term storage at -80 °C
- 8. Sample aliquots are stored at -80C in freezer-compatible cardboard or plastic storage boxes.
- 9. Samples are shipped on dry ice.
- 10. Samples must <u>never</u> be allowed to warm or thaw except from when to be used in analyses. Any deviation from this must be <u>registered</u>.

#### Responsible:



Contact person for biosampling and laboratory preparation: Siri Hinteregger, MBF Contact person for Biobank: Hilde Kristin Garberg

## 4.4 Serum for biobanking

#### Performed at: HUS

It is important to let the blood coagulate in an upright position at RT for 60 minutes. Centrifuge the sample and immediately aliquot and freeze the aliquots within 90 minutes after sample collection. Register the samples according to the local protocol and log all deviations on the same registration form.

#### Material and instrumentation:

- 3 x 5 ml BD VACUTAINER serum glass tube with no additive (367614)
- 8 x 0.7 ml FluidX (68-0702-11)
- Centrifuge for vacutainer tubes
- Barcode reader
- -80°C freezer

#### Collection, preparation and storage:

- 7. Collect whole blood into BD VACUTAINER glass tubes containing no additive.
- 8. Incubate in an upright position at room temperature for 60 min (no longer than 60 min) to allow clotting.
- 9. Centrifuge for 12 min at 1400 x g at room temperature.
- 10. Inspect serum for turbidity. Turbid samples should be centrifuged again to remove remaining insoluble matter. A new centrifugation must be indicated as a deviation.
- 11. Aliquot 500  $\mu$ L serum into 8 x 0.7 ml FluidX tubes.
- 12. Freeze the aliquots at -80°C within 90 min after sample collection.
- 13. Use the barcode reader for registration of the sample. Register the samples according to the local protocol and log all deviation on the same registration form.
- 14. Sample aliquots are stored at -80C and shipped on dry ice in the original FluidX boxes (x 48 tubes).
- 15. Samples must <u>never</u> be allowed to warm or thaw except from when to be used in analyses. Any deviation from this must be <u>registered</u>. Number and date of thawing an aliquot for analyses must be registered.



#### Responsible:

Contact person for biosampling and laboratory preparation: Siri Hinteregger, MBF

Contact person for Biobank: Hilde Kristin Garberg

## 4.5 Platelet isolation and cryopreservation for mitochondrial research

Performed at: Bergen

#### Material and instrumentation

| Item | How many | Supplier | Cat no | Comment |
|---|---|---|---|---|
| VACUETTE® TUBE 9 ml ACD-A | 1 | Greiner Bio-One | 456055 | |
| 10 ml Falcon centrifugation tubes | | | | |
| DMSO | | | | |
| Pipettes & tips | | | | |
| -80°C freezer | | Study center | | |

#### Collection, preparation and storage:

- 1. Collect whole blood in vacutainer ACD tubes (yellow cap) 9ml?
- 2. Mix gently by slowly inverting the tube
- 3. Spin at room temperature at 200g for 20min, no brake
- 4. After the spin, three distinct layers can be observed:
  - a. the top: straw-colored layer contains platelets
- 5. Transfer about two thirds of the **top layer** into a new 10ml Falcon tube
- 6. Freeze the cells in their own plasma adding DMSO at a final concentration of 5-6%
- 7. Store at -80°C



#### Responsible:

Contact person for biosampling and laboratory preparation: Siri Hinteregger, MBF

Contact person for Biobank: Hilde Kristin Garberg

## 4.6 Collection, of cerebrospinal fluid

#### Material and instrumentation:

| Item | How many | Supplier | Cat no | Comment |
|---|---|---|---|---|
| Standard lumbar puncture equipment | | | | |
| Standard CSF cell count tubes | 2 | | | |
| 5 ml PolyPropylene (PP) cryo-s tube with red PP cap | 2 | Greiner Bio-One via<br>VWR | 479-4154 | 2 uker |
| 0.7 ml FluidX tubes (PP) | 15 | Pedro Consulting | 68-0702-11N | |
| 5 ml PP tube for dementia biomarkers | 1 | Sarstedt | 63-504-027 | |
| Barcode reader | | | | |
| Centrifuge for centrifugation tubes | | Study center | | |

| PP PIPETTE TIPS (ART 1000µL REACH) | VWR | 732-2215<br>(2079-HR) | Alternative tip will be used |
|---|---|---|---|
| Pipettes | Study center | | |
| -80°C freezer | Study center | | |

## 4.6.1 Collection of cerebrospinal fluid

#### **Absolute contraindications for the procedure:**

- Thrombocytes less than 40 x 10<sup>9</sup>/L
- Use of anticoagulation (except ASA)
- INR >1.7 (warfarin users)
- Local infection at the biopsy site
- Any other center-specific clinical routines and/or guidelines MUST be followed

#### During lumbar punction the following procedures should take place:

- 1. If noticeably bloody tap, discard the first 1-2 ml until CSF is clear
- 2. 10 drops spinal fluid collected in standard tube for cell count (erythrocytes and leucocytes)
- 3. 5 ml x 2 is collected in 5 ml sterile PolyPropylene tubes (479-4154) for biobanking (see materials and preparation below)
- 4. 2 ml is collected in 5 ml PP tube for dementia biomarkers (63-504-027) for clinical analysis of abeta42, t-tau and p-tau181.
- 5. 10 drops spinal fluid collected in standard tube for cell count (erythrocytes and leucocytes)

#### NB! Do not use pressure measurements tubing – collect CSF DIRECTLY into the tubes

NB! Only polypropylene (PP) pipette tips should be used to collect and handle the CSF!

#### 4.6.2 Processing and storage of cerebrospinal fluid

- 1. The collected 5ml x 2 CSF in "5 ml PolyPropylene (PP) cryo-s tube with red PP cap"
  - a. NB! The sample has to be centrifuged within 30 min from collection!
  - b. Centrifuge within 30 min at 2,000 g, at 4 °C, for 10 min
  - c. Transfer the supernatant to 2 x new "5 ml PolyPropylene (PP) cryo-s tube with red PP cap" use PP pipette tips
  - d. Mix carefully by inverting the tube x 7-10 times (or mild vortexing)
  - e. Aliquot 500 μl CSF per tube into 0.7 ml FluidX tubes use PP pipette tips
  - f. Freeze the aliquots at -80°C.
  - g. Sample aliquots are stored at -80C and shipped on dry ice in the original FluidX boxes (x 48 tubes).
  - h. Samples must <u>never</u> be allowed to warm or thaw except from when to be used in analyses. Any deviation from this must be <u>registered</u>. Number and date of thawing an aliquot for analyses must be registered.

## 2. The collected 2 ml CSF in 5 ml PP tube for dementia biomarkers will be used for analysis of abeta42, t-tau and p-tau181:

- a. Transfer to -80C immediately after collection.
- b. Samples are stored at -80C in freezer-compatible cardboard or plastic storage boxes.
- c. Samples are shipped on dry ice.
- d. Further handling:

- i. Bergen will send batches of 20 samples to Akershus University Hospital for dementia marker analysis
- ii. Trondheim will send batches of 20 samples to Akershus University Hospital for dementia marker analysis
- iii. London will send this along with the rest of the CSF sample to Bergen (see below).
- **3.** Samples must <u>never</u> be allowed to warm or thaw except from when to be used in analyses. Any deviation from this must be <u>registered</u>. The number and date of thawing an aliquot for analyses must be registered.

#### Responsible:

Contact person for biosampling and laboratory preparation: Siri Hinteregger, MBF Contact person for Biobank: Hilde Kristin Garberg

## 4.7 Fecal sample for biobanking

## **Performed at: HUS**

Fecal samples from the last 24h will be collected according to standard clinical routines and stored at -80C. The patient must bring a 3-day diet registration from together with the fecal sample om the morning of each visit. For details on fecal sample collection and storage, see document: "SOP for fecal sample collection" (Prosedyre for avføringsprøvetaking hjemme).

## Responsible:

Bergen: Birgitte Betrentsen

## 4.8 Urine for biobanking

Performed at: HUS

Morning urine will be collected according to standard clinical routines, aliquoted and stored at -80C.

Responsible:

Bergen: Hanne Linda Nakkestad

## **5** CONTACT PERSONS

The following chapter summarizes the contact persons and responsible investigators for the substudies:

## 5.1 Helse Bergen

#### 5.1.1 Biobank Haukeland

Contact persons regarding biobanking, sample shipment, sample registration

Ann Cathrine Kroksveen 55971970 / 92031413, ann.cathrine.kroksveen@helse-

bergen.no

Hilde Garberg 55975854 / 55973149, hilde.kristin.garberg@helse-bergen.no

## 5.1.2 Laboratory Clinic

Contact person regarding safety laboratory, serology and hormone analyses

Siri Hinteregger 55973124, <a href="mailto:siri.hinteregger@helse-bergen.no">siri.hinteregger@helse-bergen.no</a>

## 5.1.3 Department of Neurology

Contact person for cells, CSF collection

Kibret Mazinga 90236164, kibret.yimer.mazengia@helse-bergen.no

Brage Brakedal 55975045 / 99777962, <u>bragebrakedal@gmail.com</u>

Kristoffer Haugarvoll <u>55975045 / 98266741, haugarvoll@gmail.com</u>

Geir Olve Skeie <u>55975045 / 48103361, Geir.Skeie@uib.no</u>

Gry Hilde NIlsen 95274886, Gry.Nilsen@uib.no

Hanne Linda Nakkestad 97571149, <a href="mailto:hanne.linda.nakkestad@helse-bergen.no">hanne.linda.nakkestad@helse-bergen.no</a>

## APPENDIX B - MRI AND FDG-PET - PROTOCOL, N-DOSE

#### Revised May 2025

#### Contact persons:

- Frank Riemer (frank.riemer@helse-bergen.no)
- Njål Brekke (njal.brekke@helse-bergen.no)
- Vivian Skjeie (vivian.skjeie@helse-bergen.no)
- Cecilie Brekke Rygh (cecilie.brekke.rygh@helse-bergen.no)

#### Bergen:

#### **Equipment:**

Scanner: Siemens Biograph mMR 3T (PET/MR)

Software: E11P

Coils: RAPID Biomedical 31P – H\_Head Coil 3T Human head V-XQ-HQ-030-01921 V01 for

SIEMENS Biograph mMR 3T

To PACS: Clinical protocol

To fPACS: All sequences (entire examination)

#### **Protocol:**

#### Participant preparation:

The participant should fast a minimum of 6 hours before injection of 18F-FDG. A peripheral venous catheter (PVC) is then placed in the medial cubital vein. Blood glucose is measured. The required blood glucose level is below 8 mmol/L. 30 minutes before the scan 250 MBq of 18F-FDG is injected into the PVC. The participant is required to lie in a quiet, dark environment during the interval after injection and before scanning to minimize brain activity. The participants should not use mobile phones or headphones during this period. Eyes must be closed for fMRI sequences. Imaging is to be taken up to 72 hours before or after physical examination of participants.

Positioning: Localizer. Auto align if possible.

Scan parameters: Scan labelled by study ID.

## MRI sequences:

- Localizer for planning of MR and PET 1.0 min.
- 3D T1 (sagittal, 1x1x1 mm, 3D-BRAVO or MPRAGE) 5.5 min.
- Attenuation correction map, generated using DeepMRAC<sup>1</sup> 2.0 min.
- 31P-MRS calibration: FID, multinuclear coil, generated using xnuccalc2 from NMproc-Dockers – 2 min.
- 31P-MRS sequence: CSI, multinuclear coil 15 min.

Total imaging time: 25.5 min imaging time - 35 min including changing the coil for CSI.

#### Specific procedures for 31P-MRS image analysis:

69

Spectra from the occipital region will be aligned using an adaption of the Spectral Registration implementation from Gannet 3.022<sup>2,3</sup>, subject to thresholding on SNR (>=3) to eliminate the majority of out-of-brain voxels.

Voxels will then be averaged before being processed in Matlab 9.5 (the MathWorks, Natick, MA) using the OXSA toolbox<sup>4</sup> utilizing first order phase correction and fitting with AMARES.

Custom prior information was created based on literature values for membrane phospholipids (MP), glycerophosphocholine (GPC), glycerophosphoethanolamine (GPE), inorganic phosphate (Pi), phosphocoline (PC), phosphoethanolamine (PE) as well as alpha-, beta- and gamma resonances of adenosine triphosphate (ATP- $\alpha$ , - $\beta$ , and - $\gamma$ , respectively) in reference to the phosphocreatine (PCr) peak<sup>5-7</sup>.

Additional information for the properties of nicotinamide adenine dinucleotide (NAD) was added based on the framework developed by Lu and colleagues<sup>8</sup> by calculating field-strength dependent chemical shift differences, relative amplitudes and frequency separations for oxidized and reduced NAD (NAD<sup>+</sup> and NADH, respectively).

Linewidths will be fixed to be equal for NAD $^+$ , NADH and ATP- $\alpha$ . At 3T, and to comply with normal-mode specific absorption rate (SAR) restrictions, peak separation for NAD $^+$  and NADH is likely to be limited and therefore only combined values of total NAD (NAD $^+$  and NADH together) will most likely be reported.

Fitted peak amplitudes and areas are used to calculate total NAD in proportion to a normalisation constant such as ATP- $\alpha$  or PCr. This normalised NAD-value will be used for the planned statistical analysis defined in the trial SAP.

#### Specific procedures for NRRP and PDRP image analysis of FDG-PET images

FDG-PET scans will be transferred electronically to the Center for Neurosciences at The Feinstein Institutes for Medical Research (Manhasset, NY, USA) and analyzed using automated computing pipelines implemented in MATLAB R2023b (MathWorks, Natick, MA). Images will first be preprocessed using Statistical Parametric Mapping (SPM12) software (<a href="http://fil.ion.ucl.ac.uk/spm">http://fil.ion.ucl.ac.uk/spm</a>; Wellcome Centre for Human Neuroimaging, London, UK). FDG-PET scans acquired at visits V1, V 2, V3 and V4 will be aligned to produce a mean image, which will be spatially normalized in standard Montreal Neurological Institute (MNI) anatomic space along with the individual scans from each time point. The normalized images will then be smoothed with a 10-mm Gaussian filter in three dimensions to enhance the signal to noise ratio.

In the previous NADPARK phase-I study<sup>9</sup>, we identified a specific NR-related metabolic pattern (NRRP) from paired metabolic scan data from participants in the NR 1000 mg group analyzed using ordinal trends/canonical variates analysis (OrT/CVA)—a supervised form of principal component analysis (PCA)<sup>10</sup>. This multivariate approach was designed to detect and quantify regional covariance patterns (i.e., metabolic networks) for which expression values (i.e., subject scores) increase or decrease with treatment in all or most of the subjects<sup>11–15</sup>. The significance of the resulting OrT/CVA topographies, i.e., the NRRP<sup>9</sup>, was assessed using nonparametric tests, i.e., permutation testing of the subject scores to show that the observed ordinal trend does not occur by chance. Likewise, the reliability of the voxel loadings (i.e., region weights) on the resulting NRRP network topography was assessed using bootstrap resampling procedures<sup>12,16</sup>.

For this study protocol, pre-processed FDG-PET scans of individual subjects will be used to compute the expression values (subject scores) of NRRP at baseline and the follow-up timepoints, using the GCVA PCA software (available at <a href="https://www.nitrc.org/projects/gcva">https://www.nitrc.org/projects/gcva</a> pca) for Ordinal Trend

(OrT/CVA) Analysis<sup>10</sup>. NRRP subject scores will be standardized (z-scored) to computed expression values for this pattern in an age-matched group of healthy volunteers scanned at the Feinstein Institutes.

FDG-PET scans will also be used to compute the expression values of the PD-related metabolic pattern (termed PDRP)<sup>17</sup> which was identified and validated previously in several independent patient populations. Subject scores for PDRP and ADRP of individual subjects will be computed automatically on a single-scan basis at each study visit and in a blinded fashion, using in-house Scan Analysis and Visualization (ScAnVP) software (available at <a href="http://feinsteinneuroscience.org">http://feinsteinneuroscience.org</a>). The subject scores of each pattern will be standardized (z-scored) in reference to corresponding scores of age-matched healthy controls.

Outcome measures of the NRRP and PDRP z-scores for individual subjects at each study visit will be reported in tabular format and transferred electronically to the Norway group for the planned statistical analysis defined in the trial SAP.

#### References

- 1. Ladefoged C.N., Hansen A.E., Henriksen O.M., et al. Al-driven attenuation correction for brain PET/MRI: Clinical evaluation of a dementia cohort and importance of the training group size. *Neuroimage* **222**, 117221 (2020).
- 2. Edden, R. A., Puts, N. A., Harris, A. D., Barker, P. B. & Evans, C. J. Gannet: A batch-processing tool for the quantitative analysis of gamma-aminobutyric acid—edited MR spectroscopy spectra. *Journal of Magnetic Resonance Imaging* **40**, 1445–1452 (2014).
- 3. Near, J. *et al.* Frequency and phase drift correction of magnetic resonance spectroscopy data by spectral registration in the time domain. *Magnetic Resonance in Medicine* **73**, 44–50 (2015).
- 4. Purvis, L. A. *et al.* OXSA: An open-source magnetic resonance spectroscopy analysis toolbox in MATLAB. *PloS one* **12**, e0185356 (2017).
- 5. Deelchand, D. K., Nguyen, T.-M., Zhu, X.-H., Mochel, F. & Henry, P.-G. Quantification of in vivo 31P NMR brain spectra using LCModel. *NMR in Biomedicine* **28**, 633–641 (2015).
- 6. Peeters, T. H., van Uden, M. J., Rijpma, A., Scheenen, T. W. & Heerschap, A. 3D 31P MR spectroscopic imaging of the human brain at 3 T with a 31P receive array: An assessment of 1H decoupling, T1 relaxation times, 1H-31P nuclear Overhauser effects and NAD+. *NMR in Biomedicine* e4169 (2019).
- 7. Ren, J., Shang, T., Sherry, A. D. & Malloy, C. R. Unveiling a hidden 31P signal coresonating with extracellular inorganic phosphate by outer-volume-suppression and localized 31P MRS in the human brain at 7T. *Magnetic resonance in medicine* **80**, 1289–1297 (2018).
- 8. Lu, M., Zhu, X.-H., Zhang, Y. & Chen, W. Intracellular redox state revealed by in vivo 31P MRS measurement of NAD+ and NADH contents in brains. *Magnetic resonance in medicine* **71**, 1959–1972 (2014).
- 9. Brakedal, B. *et al.* The NADPARK study: A randomized phase I trial of nicotinamide riboside supplementation in Parkinson's disease. *Cell Metabolism* **34**, 396-407.e6 (2022).
- 10. Habeck, C. *et al.* A new approach to spatial covariance modeling of functional brain imaging data: ordinal trend analysis. *Neural computation* **17**, 1602–1645 (2005).

- 11. Ko, J. H. *et al.* Network modulation following sham surgery in Parkinson's disease. *The Journal of clinical investigation* **124**, 3656–3666 (2014).
- 12. Mure, H. *et al.* Parkinson's disease tremor-related metabolic network: characterization, progression, and treatment effects. *Neuroimage* **54**, 1244–1253 (2011).
- 13. Mure, H. *et al.* Improved sequence learning with subthalamic nucleus deep brain stimulation: evidence for treatment-specific network modulation. *Journal of Neuroscience* **32**, 2804–2813 (2012).
- 14. Niethammer, M. *et al.* Gene therapy reduces Parkinson's disease symptoms by reorganizing functional brain connectivity. *Science translational medicine* **10**, (2018).
- 15. Tang, C. C. et al. Metabolic network as a progression biomarker of premanifest Huntington's disease. *The Journal of clinical investigation* **123**, 4076–4088 (2013).
- 16. Habeck, C. & Stern, Y. Multivariate data analysis for neuroimaging data: overview and application to Alzheimer's disease. *Cell biochemistry and biophysics* **58**, 53–67 (2010).
- 17. Schindlbeck, K. A. & Eidelberg, D. Network imaging biomarkers: insights and clinical applications in Parkinson's disease. *The Lancet Neurology* **17**, 629–640 (2018).
### **APPENDIX C - CLINICAL RATING SCALES**

### 1 GENERAL INFORMATION

The following appendix lists the clinical rating scales used in the N-DOSE study. Where clinical rating scales were used in specific sequences, this has been specified.

#### 2 **MRS-UPDRS**

#### The MDS-Sponsored Revision of the Unified Parkinson's Disease Rating Scale

For Part 1, part 3 and part 4, the English version was used. For part 2, the Norwegian version of the questionnaire was used.

MRS-UPDRS - Page 1



# **MDS-UPDRS**

The MDS-sponsored Revision of the Unified Parkinson's Disease Rating Scale

Authored by: Christopher G. Goetz Stanley Fahn Pablo Martinez-Martin Werner Poewe Cristina Sampaio Glenn T. Stebbins Matthew B. Stern Barbara C. Tilley Richard Dodel Bruno Dubois Robert Holloway Joseph Jankovic

Jaime Kulisevsky Anthony E. Lang Andrew Lees Sue Leurgans Peter A LeWitt David Nyenhuis Warren Olanow Olivier Rascol Anette Schrag Jeanne A. Teresi Jacobus J. van Hilten Nancy LaPelle

Tel +1 (414) 276-2145 Fax +1 (414) 276-3349 555 E. Wells Street, Suite 1100 Milwaukee, WI 53202-3823

www.movementdisorders.org info@movementdisorders.org

Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved.

#### **MDS Permissions**

The MDS-sponsored revision of the UPDRS (MDS-UPDRS) is owned and licensed by the International Parkinson and Movement Disorder Society (MDS). Permission is required to use the scale and can be obtained by submitting a Permissions Request Form on the MDS website. For licensing inquiries, please e-mail <a href="mailto:info@movementdisorders.org">info@movementdisorders.org</a>.

Unauthorized reproduction, distribution, translation, or sale of any portion of the MDS-UPDRS is strictly prohibited. Changes, modifications and derivative works of the scale are not permitted without the express authorization of MDS. Including but not limited to the following, the MDS-UPDRS may not be incorporated into clinical trials, training materials, certification programs, software programs, electronic platforms, electronic medical records, databases, or devices except by permission of MDS.

Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved.

#### MDS-UPDRS

The Movement Disorder Society (MDS)-sponsored new version of the UPDRS is founded on the critique that was formulated by the Task Force for Rating Scales in Parkinson's Disease (Mov Disord 2003;18:738-750). Thereafter, the MDS recruited a Chairperson to organize a program to provide the Movement Disorder community with a new version of the UPDRS that would maintain the overall format of the original UPDRS, but address issues identified in the critique as weaknesses and ambiguities. The Chairperson identified subcommittees with chairs and members. Each part was written by the appropriate subcommittee members and then reviewed and ratified by the entire group. These members are listed below.

The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). Part I has two components: IA concerns a number of behaviors that are assessed by the investigator with all pertinent information from patients and caregivers, and IB is completed by the patient with or without the aid of the caregiver, but independently of the investigator. These sections can, however, be reviewed by the rater to ensure that all questions are answered clearly and the rater can help explain any perceived ambiguities. Part II is designed to be a self-administered questionnaire like Part IB, but can be reviewed by the investigator to ensure completeness and clarity. Of note, the official versions of Part IA, Part IB and Part II of the MDS-UPDRS do not have separate "ON" or "OFF" ratings. However, for individual programs or protocols the same questions can be used separately for "ON" and "OFF". Part III has instructions for the rater to give or demonstrate to the patient; it is completed by the rater. Part IV has instructions for the rater and also instructions to be read to the patient. This part integrates patient-derived information with the rater's clinical observations and judgments and is completed by the rater.

The authors of this new version are:

Chairperson: Christopher G. Goetz

Part I: Werner Poewe (chair), Bruno Dubois, Anette Schrag Part II: Matthew B. Stern (chair), Anthony E. Lang, Peter A. LeWitt Part III: Stanley Fahn (chair), Joseph Jankovic, C. Warren Olanow
Part IV: Pablo Martinez-Martin (chair), Andrew Lees, Olivier Rascol, Bob van Hilten

Development Standards: Glenn T. Stebbins (chair), Robert Holloway, David Nyenhuis

Appendices: Cristina Sampaio (chair), Richard Dodel, Jaime Kulisevsky Statistical Testing: Barbara Tilley (chair), Sue Leurgans, Jean Teresi Consultant: Stephanie Shaftman, Nancy LaPelle

International Parkinson and Movement Disorder Society 555 East Wells Street, Suite 1100 Milwaukee, WI USA 53202

Telephone: 414-276-2145

Email: info@movementdisorders.org

July 1, 2008

Last updated August 13, 2019 | Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 1
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

#### Part I: Non-Motor Aspects of Experiences of Daily Living (nM-EDL)

Overview: This portion of the scale assesses the non-motor impact of Parkinson's disease (PD) on patients' experiences of daily living. There are 13 questions. Part IA is administered by the rater (six questions) and focuses on complex behaviors. Part IB is a component of the self-administered Patient Questionnaire that covers seven questions on non-motor experiences of daily living.

#### Part IA

In administering Part IA, the examiner should use the following guidelines:

- Mark at the top of the form the primary data source as patient, caregiver, or patient and caregiver in equal proportion.
- The response to each item should refer to a period encompassing the prior week including the day on which the information is collected.
- All items must have an integer rating (no half points, no missing scores). In the event that an item does not apply
  or cannot be rated (e.g., amputee who cannot walk), the item is marked "UR" for Unable to Rate.
- 4. The answers should reflect the usual level of function and words such as "usually," "generally," "most of the time" can be used with patients.
- 5. Each question has a text for you to read (Instructions to patients/caregiver). After that statement, you can elaborate and probe based on the target symptoms outlined in the Instructions to examiner. You should NOT READ the RATING OPTIONS to the patient/caregiver, because these are written in medical terminology. From the interview and probing, you will use your medical judgment to arrive at the best response.
- Patients may have co-morbidities and other medical conditions that can affect their function. You and the patient must rate the problem as it exists and do not attempt to separate elements due to Parkinson's disease from other conditions.

#### EXAMPLE OF NAVIGATING THROUGH THE RESPONSE OPTIONS FOR PART IA

Suggested strategies for obtaining the most accurate answer:

After reading the instructions to the patient, you will need to probe the entire domain under discussion to determine normal vs. problematic: If your questions do not identify any problem in this domain, record 0 and move on to the next question.

If your questions identify a problem in this domain, you should work next with a reference anchor at the mid-range (option 2 or Mild) to find out if the patient functions at this level, better or worse. You will not be reading the choices of responses to the patient as the responses use clinical terminology. You will be asking enough probing questions to determine the response that should be coded.

Work up and down the options with the patient to identify the most accurate response, giving a final check by excluding the options above and below the selected response.



Last updated August 13, 2019 | Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 2
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| Patient Name | or Subject ID | Site ID | (mm-dd-yyyy)<br>Assessment Date | Investiga | tor's Initials |
|---|---|---|---|---|---|
| Pa | ırt I: Non-Motor / | MDS UPI<br>Aspects of Experie | DRS<br>nces of Daily Living (n | M-EDL) | |
| Part IA: Complex I | behaviors: [complet | ted by rater] | | | |
| Primary source of ir | nformation: | | | | |
| ☐ Patient | ☐ Caregiver | ☐ Patient an | d Caregiver in Equal Proporti | on | |
| WEEK. If you are no | | blem, you can simply res | have felt MOST OF THE TIN | | |
| slowing, impaired re<br>activities of daily livi<br>Instructions to patie<br>following conversati | niner: Consider all type<br>easoning, memory losing as perceived by the<br>ent [and caregiver]: Officials, paying attention | ss, deficits in attention a<br>the patient and/or caregi<br>over the past week have<br>n, thinking clearly, or find | you had problems remember<br>ding your way around the hou | act on ing things, | SCORE |
| Instructions to exan<br>slowing, impaired re<br>activities of daily livi<br>Instructions to patie<br>following conversati<br>town? [If yes, exam | niner: Consider all type<br>easoning, memory los<br>ing as perceived by t<br>ent [and caregiver]: O<br>ions, paying attention<br>iner asks patient or c | ss, deficits in attention a<br>the patient and/or caregi-<br>over the past week have<br>n, thinking clearly, or find<br>caregiver to elaborate ar | nd orientation. Rate their imp<br>ver.<br>you had problems remember | act on ing things, | SCORE |
| Instructions to exam<br>slowing, impaired re<br>activities of daily livi<br>Instructions to patie<br>following conversati | niner: Consider all type<br>easoning, memory losing as perceived by the entire (and caregiver): Officers, paying attention iner asks patient or consider the constitution of the constitution | ss, deficits in attention a<br>the patient and/or caregin<br>over the past week have<br>n, thinking clearly, or find<br>caregiver to elaborate ar<br>ment. | nd orientation. Rate their imp<br>ver.<br>you had problems rememben<br>ding your way around the hou | act on<br>ing things,<br>se or in | SCORE |
| Instructions to exan<br>slowing, impaired re<br>activities of daily livi<br>Instructions to patie<br>following conversati<br>town? [If yes, exam<br>0: Normal: | niner: Consider all type<br>easoning, memory losing as perceived by the sent [and caregiver]: Officers, paying attention iner asks patient or constitute impaired the patient's ability Clinically evident consider a sent appreciation of the patient's ability clinically evident consider a sent appreciation of the patient's ability clinically evident consider a sent appreciation of the patient's ability clinically evident consideration. | ss, deficits in attention a<br>the patient and/or caregi-<br>over the past week have<br>in, thinking clearly, or find<br>caregiver to elaborate ar<br>ment.<br>isted by patient or caregiver to carry out normal action | nd orientation. Rate their imporer. you had problems remember the hound probes for information.] | act on ing things, se or in | SCORE |
| Instructions to exan slowing, impaired re activities of daily livinstructions to patie following conversatiown? [If yes, exam 0: Normal: 1: Slight: | niner: Consider all typessoning, memory losing as perceived by the net [and caregiver]: Officers, paying attention iner asks patient or construction of the patient's ability. Clinically evident or the patient's ability. Cognitive deficits in | ss, deficits in attention a<br>the patient and/or careginal<br>over the past week have<br>n, thinking clearly, or find<br>caregiver to elaborate are<br>ment. iated by patient or caregory out normal active<br>or to carry out normal active to carry out normal active | nd orientation. Rate their imporer. you had problems remember thing your way around the hound probes for information.] giver with no concrete interferenties and social interactions. I only minimal interference will wities and social interactions. preclude the patient's ability to | act on ing things, se or in ence with | SCORE |

| 1.2 HALLUCINATI | ONS AND PSYCHOSIS | SCORE |
|---|---|---|
| Instructions to exar<br>(spontaneous false<br>and gustatory). Det<br>impressions) as we | <u>miner</u> : Consider both illusions (misinterpretations of real stimuli) and hallucinations sensations). Consider all major sensory domains (visual, auditory, tactile, olfactory, ermine presence of unformed (for example sense of presence or fleeting false as formed (fully developed and detailed) sensations. Rate the patient's insight into identify delusions and psychotic thinking. | |
| | ent [and caregiver]: Over the past week have you seen, heard, smelled, or felt things there? [If yes, examiner asks patient or caregiver to elaborate and probes for | |
| 0: Normal: | No hallucinations or psychotic behavior. | |
| 1: Slight: | Illusions or non-formed hallucinations, but patient recognizes them without loss of insight. $ \\$ | |
| 2: Mild: | Formed hallucinations independent of environmental stimuli. No loss of insight. | |
| 3: Moderate: | Formed hallucinations with loss of insight. | |
| 4: Severe: | Patient has delusions or paranola. | |
| 1.3 DEPRESSED | | |
| Instructions to exar<br>enjoyment. Determi | MOOD miner: Consider low mood, sadness, hopelessness, feelings of emptiness, or loss of ine their presence and duration over the past week and rate their interference with to carry out daily routines and engage in social interactions. | |
| Instructions to examenjoyment. Determithe patient's ability Instructions to patient of the patie | miner: Consider low mood, sadness, hopelessness, feelings of emptiness, or loss of ine their presence and duration over the past week and rate their interference with to carry out daily routines and engage in social interactions. Sent [and caregiver]: Over the past week have you felt low, sad, hopeless, or unable to it, was this feeling for longer than one day at a time? Did it make it difficult for you all activities or to be with people? [If yes, examiner asks patient or caregiver to | |
| Instructions to examenjoyment. Determithe patient's ability Instructions to patient of the patie | miner: Consider low mood, sadness, hopelessness, feelings of emptiness, or loss of ine their presence and duration over the past week and rate their interference with to carry out daily routines and engage in social interactions. Sent [and caregiver]: Over the past week have you felt low, sad, hopeless, or unable to it, was this feeling for longer than one day at a time? Did it make it difficult for you all activities or to be with people? [If yes, examiner asks patient or caregiver to | |
| Instructions to examenjoyment. Determithe patient's ability Instructions to patient of the patient's ability Instructions to patient of the patient's ability Instructions to patient of the patient o | miner: Consider low mood, sadness, hopelessness, feelings of emptiness, or loss of ine their presence and duration over the past week and rate their interference with to carry out daily routines and engage in social interactions. Lent [and caregiver]: Over the past week have you felt low, sad, hopeless, or unable to be to some the same of | |
| Instructions to exarenjoyment. Determithe patient's ability Instructions to patie enjoy things? If yes carry out your usua elaborate and probe 0: Normal: | miner: Consider low mood, sadness, hopelessness, feelings of emptiness, or loss of ine their presence and duration over the past week and rate their interference with to carry out daily routines and engage in social interactions. **ent [and caregiver]: Over the past week have you felt low, sad, hopeless, or unable to it, was this feeling for longer than one day at a time? Did it make it difficult for you all activities or to be with people? [If yes, examiner asks patient or caregiver to es for information.] No depressed mood. Episodes of depressed mood that are not sustained for more than one day at a time. No interference with patient's ability to carry out normal activities and social | |
| Instructions to exarenjoyment. Determithe patient's ability Instructions to patie enjoy things? If yes carry out your usua elaborate and probe 0: Normal: 1: Slight: | miner: Consider low mood, sadness, hopelessness, feelings of emptiness, or loss of ine their presence and duration over the past week and rate their interference with to carry out daily routines and engage in social interactions. **Ent [and caregiver]: Over the past week have you felt low, sad, hopeless, or unable to it, was this feeling for longer than one day at a time? Did it make it difficult for you all activities or to be with people? [If yes, examiner asks patient or caregiver to es for information.] No depressed mood. Episodes of depressed mood that are not sustained for more than one day at a time. No interference with patient's ability to carry out normal activities and social interactions. Depressed mood that is sustained over days, but without interference with | |
| Instructions to examenjoyment. Determithe patient's ability Instructions to patien enjoy things? If yes carry out your usual elaborate and probe 0: Normal: 1: Slight: 2: Mild: | <ul> <li>miner: Consider low mood, sadness, hopelessness, feelings of emptiness, or loss of ine their presence and duration over the past week and rate their interference with to carry out daily routines and engage in social interactions.</li> <li>ent [and caregiver]: Over the past week have you felt low, sad, hopeless, or unable to it, was this feeling for longer than one day at a time? Did it make it difficult for you all activities or to be with people? [If yes, examiner asks patient or caregiver to es for information.]</li> <li>No depressed mood.</li> <li>Episodes of depressed mood that are not sustained for more than one day at a time. No interference with patient's ability to carry out normal activities and social interactions.</li> <li>Depressed mood that is sustained over days, but without interference with normal activities and social interactions.</li> <li>Depressed mood that interferes with, but does not preclude the patient's ability</li> </ul> | |

| 1.4 AN | XIOUS MO | DOD | SCORE |
|---|---|---|---|
| over the | e past week | <u>miner:</u> Determine nervous, tense, worried, or anxious feelings (including panic attacks) cand rate their duration and interference with the patient's ability to carry out daily ge in social interactions. | |
| yes, wa<br>activitie | s this feelir | ient [and caregiver]: Over the past week have you felt nervous, worried, or tense? If<br>ng for longer than one day at a time? Did it make it difficult for you to follow your usual<br>with other people? [If yes, examiner asks patient or caregiver to elaborate and probes | |
| 0: | Normal: | No anxious feelings. | |
| 1: | Slight: | Anxious feelings present but not sustained for more than one day at a time. No interference with patient's ability to carry out normal activities and social interactions. | |
| 2: | Mild: | Anxious feelings are sustained over more than one day at a time, but without interference with patient's ability to carry out normal activities and social interactions. | |
| 3: | Moderate: | Anxious feelings interfere with, but do not preclude, the patient's ability to carry out normal activities and social interactions. | |
| 4: | Severe: | Anxious feelings preclude patient's ability to carry out normal activities and social interactions. | |
| 1.5 AP | | miner: Consider level of spontaneous activity, assertiveness, motivation, and initiative | |
| Instruct<br>and rate | ions to exa<br>e the impac<br>er should a | <u>miner</u> : Consider level of spontaneous activity, assertiveness, motivation, and initiative of of reduced levels on performance of daily routines and social interactions. Here the attempt to distinguish between apathy and similar symptoms that are best explained by | |
| Instruct<br>and rate<br>examine<br>depress | ions to exa<br>e the impac<br>er should a<br>sion. | ct of reduced levels on performance of daily routines and social interactions. Here the | |
| Instruct<br>and rate<br>examine<br>depress<br>Instruct<br>or being | ions to exa<br>e the impac<br>er should a<br>sion. | ct of reduced levels on performance of daily routines and social interactions. Here the attempt to distinguish between apathy and similar symptoms that are best explained by item [and caregiver]: Over the past week, have you felt indifferent to doing activities | |
| Instruct<br>and rate<br>examine<br>depress<br>Instruct<br>or being<br>0: | ions to exa<br>e the impacer should a<br>sion.<br>tions to pati<br>g with people | ct of reduced levels on performance of daily routines and social interactions. Here the ittempt to distinguish between apathy and similar symptoms that are best explained by sient [and caregiver]: Over the past week, have you felt indifferent to doing activities le? [If yes, examiner asks patient or caregiver to elaborate and probes for information.] | |
| Instruct and rate examine depress Instruct or being 0: | ions to exa<br>e the impacer should a<br>sion.<br>tions to pati<br>g with peop.<br>Normal: | to freduced levels on performance of daily routines and social interactions. Here the ittempt to distinguish between apathy and similar symptoms that are best explained by lent [and caregiver]: Over the past week, have you felt indifferent to doing activities le? [If yes, examiner asks patient or caregiver to elaborate and probes for information.] No apathy. Apathy appreciated by patient and/or caregiver, but no interference with daily | |
| Instruct and rate examine depress Instruct or being 0: 1: | ions to exa<br>e the impacer should a<br>sion.<br>tions to pati<br>g with people<br>Normal:<br>Slight: | ct of reduced levels on performance of daily routines and social interactions. Here the ittempt to distinguish between apathy and similar symptoms that are best explained by sient [and caregiver]: Over the past week, have you felt indifferent to doing activities le? [If yes, examiner asks patient or caregiver to elaborate and probes for information.] No apathy. Apathy appreciated by patient and/or caregiver, but no interference with daily activities and social interactions. Apathy interferes with isolated activities and social interactions. | |
| Instruct and rate examine depress Instruct or being 0: 1: 2: 3: | ions to exa e the impace er should a sion. tions to pati g with peop Normal: Slight: | ct of reduced levels on performance of daily routines and social interactions. Here the ittempt to distinguish between apathy and similar symptoms that are best explained by sient [and caregiver]: Over the past week, have you felt indifferent to doing activities le? [If yes, examiner asks patient or caregiver to elaborate and probes for information.] No apathy. Apathy appreciated by patient and/or caregiver, but no interference with daily activities and social interactions. Apathy interferes with isolated activities and social interactions. | |

80

| | | SCORE |
|---|---|---|
| 1.6 FEATURES OF | F DOPAMINE DYSREGULATION SYNDROME | |
| excessive gambling<br>interests (e.g., unus<br>other repetitive acti<br>extra non-prescribed<br>impact of such abnorand social relations | niner: Consider involvement in a variety of activities including atypical or (e.g. casinos or lottery tickets), atypical or excessive sexual drive or sual interest in pornography, masturbation, sexual demands on partner), wities (e.g. hobbies, dismantling objects, sorting or organizing), or taking d medication for non-physical reasons (i.e., addictive behavior). Rate the ormal activities/behaviors on the patient's personal life and on his/her family (including need to borrow money or other financial difficulties like cards, major family conflicts, lost time from work, or missed meals or sleep wity). | |
| urges that are hard<br>hard to stop? [Give | ent [and caregiver]: Over the past week, have you had unusually strong<br>to control? Do you feel driven to do or think about something and find it<br>patient examples such as gambling, cleaning, using the computer, taking<br>essing about food or sex, all depending on the patient.] | |
| 0: Normal: | No problems present. | |
| 1: Slight: | Problems are present but usually do not cause any difficulties for the patient or family/caregiver. | |
| 2: Mild: | Problems are present and usually cause a few difficulties in the patient's personal and family life. | |
| 3: Moderate: | Problems are present and usually cause a lot of difficulties in the patient's personal and family life. | |
| 4: Severe: | Problems are present and preclude the patient's ability to carry out normal activities or social interactions or to maintain previous standards in personal and family life. | |
| Other Sensation, | questions in Part I (Non-motor Experiences of Daily Living) [Sleep, Daytime Sleepiness,<br>Urinary Problems, Constipation Problems, Lightheadedness on Standing, and Fatigue<br>nt Questionnaire along with all questions in Part II [Motor Experiences of Daily Living]. | |

| | Spørreskjema for pasienter |
|---|---|
| Instruksjoner: | |
| Det er 20 spørsmål. V<br>er kanskje ikke aktuel<br>problemer, bare svar ( | tar for seg erfaringer i dagliglivet.<br>i prøver å være grundige, og noen av disse spørsmålene<br>le for deg nå eller noen gang. Hvis du ikke har<br>of for NEI.<br>ørsmål nøye og les alle svarene før du velger det som |
| den siste uken inklude<br>dagen enn på andre tid | gjennomsnittlige eller vanlige funksjonsnivå i løpet av<br>ert i dag. Noen pasienter kan gjøre ting bedre på en tid av<br>der. Men bare ett svar er tillatt for hvert spørsmål, så<br>svaret som best beskriver hva du kan gjøre <u>mesteparten</u> |
| | sykdommer i tillegg til Parkinsons sykdom. Ikke prøv å<br>undre sykdommer. Bare svar på spørsmålet så godt du |
| Bruk bare 0, 1, 2, 3, 4 | i svarene, ikke noe annet. Ikke la noen svar stå åpne. |
| | ren kan gå igjennom spørsmålene med deg, men det er<br>skal fylle ut spørreskjemaet, enten alene eller sammen<br>n. |
| Hvem fyller ut dette s | pørreskjemaet? (svar det som passer best) |
| Pasient | |
| Omsorgsperson | |
| Pasient og omsorgspe | rson i like stor grad |

| | otoriske aspekter ved erfaringer i dagliglivet (iM-EDL) |
|---|---|
| 1.7 SØVNVAN | SKER |
| | uken, har du hatt problemer med å sovne om kvelden eller forblittt våken<br>Tenk over hvor uthvilt du følte deg etter å ha våknet om morgenen. |
| 0: Normal: | Ingen problemer. |
| 1: Meget lett: | Søvnvansker er tilstede, men gir vanligvis ikke<br>problemer med å få en full natts søvn. |
| 2: Mild: | Søvnvansker gir noen problemer med å få en full natts<br>søvn. |
| 3: Moderat: | Søvnvansker gir mye problemer med å få en full natts<br>søvn, men jeg sover vanligvis mer enn halve natten. |
| 4: Alvorlig: | Vanligvis sover jeg ikke mesteparten av natten. |
| 1.8 SØVNIGH | ET PÅ DAGTID |
| | ET PÅ DAGTID<br>te uken, har du hatt problemer med å holde deg våken på dagtid? |
| I løpet av den sist | te uken, har du hatt problemer med å holde deg våken på dagtid? |
| I løpet av den sist<br>0: Normal: | te uken, har du hatt problemer med å holde deg våken på dagtid? Ingen søvnighet på dagtid. Søvnighet på dagtid forekommer, men jeg kan stå imot |
| I løpet av den sist<br>0: Normal:<br>1: Meget lett: | Ingen søvnighet på dagtid. Søvnighet på dagtid forekommer, men jeg kan stå imot og holder meg våken. Noen ganger sovner jeg når jeg er alene og slapper av, |
| I løpet av den sist<br>0: Normal:<br>1: Meget lett:<br>2: Mild: | Ingen søvnighet på dagtid. Søvnighet på dagtid forekommer, men jeg kan stå imot og holder meg våken. Noen ganger sovner jeg når jeg er alene og slapper av, for eksempel når jeg leser eller ser TV. Av og til sovner jeg når jeg ikke burde, for eksempel når |
| I løpet av den sist 0: Normal: 1: Meget lett: 2: Mild: 3: Moderat: | Ingen søvnighet på dagtid. Søvnighet på dagtid forekommer, men jeg kan stå imot og holder meg våken. Noen ganger sovner jeg når jeg er alene og slapper av, for eksempel når jeg leser eller ser TV. Av og til sovner jeg når jeg ikke burde, for eksempel når jeg spiser eller snakker med andre mennesker. Jeg sovner ofte når jeg ikke burde, for eksempel når jeg |
| I løpet av den sist 0: Normal: 1: Meget lett: 2: Mild: 3: Moderat: | Ingen søvnighet på dagtid. Søvnighet på dagtid forekommer, men jeg kan stå imot og holder meg våken. Noen ganger sovner jeg når jeg er alene og slapper av, for eksempel når jeg leser eller ser TV. Av og til sovner jeg når jeg ikke burde, for eksempel når jeg spiser eller snakker med andre mennesker. Jeg sovner ofte når jeg ikke burde, for eksempel når jeg |

| I løpet av den siste uken, har du hatt ubehagelige følelser i kroppen som smerter, verking, prikkinger eller kramper? O: Normal: Ingen ubehagelige følelser. 1: Meget lett: Jeg har slike følelser, men jeg kan gjøre ting og være sammen med andre mennesker uten vanskeligheter. 2: Mild: Disse følelsene gir meg noen problemer når jeg gjør ting eller er sammen med andre mennesker. 3: Moderat: Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? O: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen og bruker truseinnlegg eller har blærekateter. | prikkinger eller kramper? 0: Normal: Ingen ubehagelige følelser. 1: Meget lett: Jeg har slike følelser, men jeg kan gjøre ting og være sammen med andre mennesker uten vanskeligheter. 2: Mild: Disse følelsene gir meg noen problemer når jeg gjør ting eller er sammen med andre mennesker. 3: Moderat: Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker. 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | | OG ANDRE SANSEOPPLEVELSER |
|---|---|---|---|
| 1: Meget lett: Jeg har slike følelser, men jeg kan gjøre ting og være sammen med andre mennesker uten vanskeligheter. 2: Mild: Disse følelsene gir meg noen problemer når jeg gjør ting eller er sammen med andre mennesker. 3: Moderat: Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 1: Meget lett: Jeg har slike følelser, men jeg kan gjøre ting og være sammen med andre mennesker uten vanskeligheter. 2: Mild: Disse følelsene gir meg noen problemer når jeg gjør ting eller er sammen med andre mennesker. 3: Moderat: Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | | |
| sammen med andre mennesker uten vanskeligheter. 2: Mild: Disse følelsene gir meg noen problemer når jeg gjør ting eller er sammen med andre mennesker. 3: Moderat: Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. | sammen med andre mennesker uten vanskeligheter. 2: Mild: Disse følelsene gir meg noen problemer når jeg gjør ting eller er sammen med andre mennesker. 3: Moderat: Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. | 0: Normal: | Ingen ubehagelige følelser. |
| eller er sammen med andre mennesker. 3: Moderat: Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | eller er sammen med andre mennesker. Disse følelsene gir meg mye problemer, men de hindrer meg ikke fra å gjøre ting eller være sammen med andre mennesker. Lio Vannlatingsproblemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? Ingen problemer med kontrollen over vannlatingen. Ingen problemer med kontrollen over vannlatingen. Ingen problemer med kontrollen over vannlatingen. Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. Jeg kan ikke kontrollere vannlatingen og bruker | 1: Meget lett: | |
| meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. | meg ikke fra å gjøre ting eller være sammen med andre mennesker. 4. Alvorlig: Disse følelsene hindrer meg i å gjøre ting eller være sammen med andre mennesker 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 2: Mild: | |
| 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 1.10 VANNLATINGSPROBLEMER I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 3: Moderat: | meg ikke fra å gjøre ting eller være sammen med andre |
| I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | I løpet av den siste uken, har du hatt problemer med kontroll over vannlatingen? For ekser et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 4. Alvorlig: | |
| et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | et plutselig behov for å late vannet, en trang til å late vannet for hyppig, eller uhell med vannlatingen? 0: Normal: Ingen problemer med kontrollen over vannlatingen. 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 1.10 VANNLA | TINGSPROBLEMER |
| 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 1: Meget lett: Jeg må late vannet ofte eller med en gang jeg kjenner trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | et plutselig behov | |
| trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | trang. Men disse problemene gir meg ingen vanskeligheter i mine daglige aktiviteter. 2: Mild: Vannlatingsproblemer gir meg noe problemer i daglige aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 0: Normal: | Ingen problemer med kontrollen over vannlatingen. |
| aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | aktiviteter, men jeg har ikke hatt uhell med vannlatingen. 3: Moderat: Vannlatingsproblemer gir meg mye problemer i daglige aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | 1: Meget lett: | trang. Men disse problemene gir meg ingen |
| aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | aktiviteter, inkludert uhell med vannlatingen. 4: Alvorlig: Jeg kan ikke kontrollere vannlatingen og bruker | | aktiviteter, men jeg har ikke hatt uhell med |
| | | 2: Mild: | |
| | | 3: Moderat: | aktiviteter, inkludert uhell med vannlatingen. Jeg kan ikke kontrollere vannlatingen og bruker |

| Har du i løpet av den siste uken hatt problemer md forstoppelse som medfører at du har vanskeligheter med å få avføring? 0: Normal: Ingen forstoppelse. 1: Meget lett: Jeg har hatt forstoppelse, jeg bruker ekstra krefter på å ha avføring. Dette forstyrrer imidlertid ikke mine daglige aktiviteter eller velvære. 2: Mild: Forstoppelse medfører problemer i aktiviteter eller velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller besvimer. | vanskeligheter med å få avføring? 0: Normal: Ingen forstoppelse. 1: Meget lett: Jeg har hatt forstoppelse, jeg bruker ekstra krefter på å ha avføring. Dette forstyrrer imidlertid ikke mine daglige aktiviteter eller velvære. 2: Mild: Forstoppelse medfører problemer i aktiviteter eller velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | | MER MED FORSTOPPELSE |
|---|---|---|---|
| 1: Meget lett: Jeg har hatt forstoppelse, jeg bruker ekstra krefter på å ha avføring. Dette forstyrrer imidlertid ikke mine daglige aktiviteter eller velvære. 2: Mild: Forstoppelse medfører problemer i aktiviteter eller velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 1: Meget lett: Jeg har hatt forstoppelse, jeg bruker ekstra krefter på å ha avføring. Dette forstyrrer imidlertid ikke mine daglige aktiviteter eller velvære. 2: Mild: Forstoppelse medfører problemer i aktiviteter eller velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | | |
| ha avføring. Dette forstyrrer imidlertid ikke mine daglige aktiviteter eller velvære. 2: Mild: Forstoppelse medfører problemer i aktiviteter eller velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | ha avføring. Dette forstyrrer imidlertid ikke mine daglige aktiviteter eller velvære. 2: Mild: Forstoppelse medfører problemer i aktiviteter eller velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 0: Normal: | Ingen forstoppelse. |
| velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | velvære. 3: Moderat: Forstoppelse medfører mye problemer i aktiviteter eller velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 1: Meget lett: | ha avføring. Dette forstyrrer imidlertid ikke mine |
| velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | velvære. Det hindrer meg imidlertid ikke i aktiviteter. 4: Alvorlig: Jeg trenger vanligvis fysisk hjelp av noen for å tømme tarmen. 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 2: Mild: | |
| 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 1.12 SVIMMELHET I STÅENDE STILLING Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 3: Moderat: | |
| Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | Har du i løpet av den siste uken følt deg svimmel, tåkete eller at du vil besvime når du rei deg opp fra sittende eller liggende stiling? 0: Normal: Ingen svimmelhet eller tåkefølelse. 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 4: Alvorlig: | |
| 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | TT 1 11 / | dan sista ultan falt dan szimmal, táltata allan at du zil haszima nån du nai |
| 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | 1: Meget lett: Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | | |
| 2: Mild: Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. 3: Moderat: Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | deg opp fra sitten | de eller liggende stiling? |
| meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | meg eller legge meg ned for å unngå å besvime eller falle. 4: Alvorlig: Svimmelhet eller tåkefølelse fører til at jeg faller eller | deg opp fra sitten<br>0: Normal: | de eller liggende stiling? Ingen svimmelhet eller tåkefølelse. Svimmelhet eller tåkefølelse forekommer. Det hindrer |
| | | deg opp fra sitten<br>0: Normal:<br>1: Meget lett: | de eller liggende stiling? Ingen svimmelhet eller tåkefølelse. Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge |
| | | deg opp fra sitten<br>0: Normal:<br>1: Meget lett:<br>2: Mild: | Ingen svimmelhet eller tåkefølelse. Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller |
| | | deg opp fra sitten 0: Normal: 1: Meget lett: 2: Mild: 3: Moderat: | Ingen svimmelhet eller tåkefølelse. Svimmelhet eller tåkefølelse forekommer. Det hindrer meg imidlertid ikke i å gjøre noe. Svimmelhet eller tåkefølelse medfører at jeg må holde meg fast, men jeg trenger ikke å sette meg eller legge meg ned. Svimmelheteller tåkefølelse medfører at jeg må sette meg eller legge meg ned for å unngå å besvime eller falle. Svimmelhet eller tåkefølelse fører til at jeg faller eller |

| 1.13 UTMATT | тетнет |
|---|---|
| Har du stort sett f<br>eller trist. | følt deg utmattet den siste uken? Denne følelsen er <u>ikke</u> ledd i å være tre |
| 0: Normal: | Ingen utmattethet. |
| 1: Meget lett: | Utmattethet forekommer. Det medfører imidlertid ikke problemer med å gjøre ting eller være sammen med mennesker. |
| 2: Mild: | Utmattethet medfører noen problemer med å gjøre ting<br>eller være sammen med mennesker. |
| 3: Moderat: | Utmattethet medfører mye problemer med å gjøre ting<br>eller være sammen med mennesker. Det stopper meg<br>imidlertid ikke fra å gjøre noe. |
| | minderate have he algore nee. |
| | Utmattethet hindrer meg i å gjøre ting eller være sammen med mennesker. |
| Del II: Motori | Utmattethet hindrer meg i å gjøre ting eller være sammen med mennesker. |
| Del II: Motori<br>2.1 TALE<br>I løpet av den sist | Utmattethet hindrer meg i å gjøre ting eller være sammen med mennesker. iske aspekter ved erfaringer i dagliglivet (M-EDL) te uken, har du hatt problemer med talen? |
| Del II: Motori | Utmattethet hindrer meg i å gjøre ting eller være sammen med mennesker. |
| Del II: Motori<br>2.1 TALE<br>I løpet av den sist<br>0: Normal: | Utmattethet hindrer meg i å gjøre ting eller være sammen med mennesker. iske aspekter ved erfaringer i dagliglivet (M-EDL) te uken, har du hatt problemer med talen? Ikke i det hele tatt (Ingen problemer). Talen min er svak, skurret og ujevn, men det medfører |
| Del II: Motori<br>2.1 TALE<br>I løpet av den sist<br>0: Normal:<br>1: Meget lett: | Utmattethet hindrer meg i å gjøre ting eller være sammen med mennesker. iske aspekter ved erfaringer i dagliglivet (M-EDL) te uken, har du hatt problemer med talen? Ikke i det hele tatt (Ingen problemer). Talen min er svak, skurret og ujevn, men det medfører ikke at andre ber meg gjenta meg. Talen min medfører at andre av og til ber meg gjenta, |

| I løpet av den siste uken, har du vanligvis hatt for mye spytt mens du er våken eller mens sover? 1: Meget lett: Jeg har for mye spytt, men sikler ikke. 2: Mild: Jeg sikler noe mens jeg sover, men ikke når jeg er våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger emæringssonde på grunn av problemer med tygging og svelging. | 1: Meget lett: Jeg har for mye spytt, men sikler ikke. 2: Mild: Jeg sikler noe mens jeg sover, men ikke når jeg er våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ermæringssonde på grunn av problemer med | I longt av den sist | a ukan har du vanliggis hatt for mya saytt mans du ar våkan allar mans d |
|---|---|---|---|
| 1: Meget lett: Jeg har for mye spytt, men sikler ikke. 2: Mild: Jeg sikler noe mens jeg sover, men ikke når jeg er våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger emæringssonde på grunn av problemer med | 1: Meget lett: Jeg har for mye spytt, men sikler ikke. 2: Mild: Jeg sikler noe mens jeg sover, men ikke når jeg er våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ermæringssonde på grunn av problemer med | _ | e uken, når du vanngvis nad for mye spyd mens du er vaken ener mens d |
| 2: Mild: Jeg sikler noe mens jeg sover, men ikke når jeg er våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 2: Mild: Jeg sikler noe mens jeg sover, men ikke når jeg er våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 0: Normal: | Ikke i det hele tatt (ingen problemer). |
| våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | våken. 3: Moderat: Jeg sikler noe når jeg er våken, men jeg trenger vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 1: Meget lett: | Jeg har for mye spytt, men sikler ikke. |
| vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | vanligvis ikke tørkepapir eller lommetørkle. 4: Alvorlig: Jeg sikler så mye at jeg regelmessig trenger tørkepapir eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal umngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 2: Mild: | |
| eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal umgå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | eller lommetørkle for å beskytte klærne mine. 2.3 TYGGING OG SVELGING I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 3: Moderat: | |
| I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 4: Alvorlig: | |
| I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | I løpet av den siste uken, har du vanligvis problemer med å svelge tabletter eller spise måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | | |
| måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for at skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | måltider? Må tablettene være delt eller knust eller maten bløt, kuttet opp eller most for skal unngå å svelge vrangt? 0: Normal: Ingen problemer. 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 2.3 TYGGING | G OG SVELGING |
| 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 1: Meget lett: Jeg vet jeg tygger sakte og bruker ekstra krefter på å svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger emæringssonde på grunn av problemer med | måltider? Må tabl | ettene være delt eller knust eller maten bløt, kuttet opp eller most for at |
| svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | svelge, men jeg svelger ikke vrangt eller behøver maten min spesielt tilberedt. 2: Mild: Jeg må ha tablettene delt eller maten spesielt tilberedt på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 0: Normal: | Ingen problemer. |
| på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | på grunn av problemer med tygging eller svelging, men jeg har ikke svelget vrangt i løpet av den siste uken. 3: Moderat: Jeg har svelget vrangt minst en gang i løpet av den siste uken. 4: Alvorlig: Jeg trenger emæringssonde på grunn av problemer med | 1: Meget lett: | svelge, men jeg svelger ikke vrangt eller behøver maten |
| uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | uken. 4: Alvorlig: Jeg trenger ernæringssonde på grunn av problemer med | 2: Mild: | på grunn av problemer med tygging eller svelging, men |
| | | 3: Moderat: | |
| | | 4: Alvorlig: | |

| 2.4 SPISING | uken, har du vanligvis hatt problemer md å håndtere mat og bruke |
|---|---|
| | du for eksempel problemer med å håndtere fingermat eller bruke gafler, |
| 0: Normal: | Ingen problemer |
| 1: Meget lett: | Jeg er langsom, men trenger ikke hjelp og søler ikke<br>mens jeg spiser. |
| 2: Mild: | Jeg er langsom når jeg spiser og søler mat av og til. Jeg<br>kan trenge hjelp med noen oppgaver slik som å skjære<br>opp kjøtt. |
| 3: Moderat: | Jeg trenger hjelp med mange spiseoppgaver men kan klare noen alene. |
| 4: Alvorlig: | Jeg trenger hjelp til de fleste eller alle spiseoppgaver. |
| 2.5 PÅKLEDNI | ing. |
| | uken, har du hatt problemer med å kle på deg? Er du for eksempel<br>ger hjelp med å kneppe knapper, bruke glidelåser, ta på eller av klær eller |
| 0: Normal: | Ikke i det hele tatt (ingen problemer). |
| 1: Meget lett: | Jeg er langsom, men trenger ikke hjelp. |
| 2: Mild: | Jeg er langsom og trenger hjelp til noen få oppgaver<br>(knapper, armbånd) |
| 3. Moderat: | Jeg trenger hjelp til mange påkledningsoppgaver. |
| 4: Alvorlig: | Jeg trenger hjelp til de fleste eller alle<br>påkledningsoppgaver. |

| 0: Normal: Ikke i det hele tatt (ingen problemer). 1: Meget lett; Jeg er langsom, men jeg trenger ikke hjelp. 2: Mild: Jeg trenger noen til å hjelpe meg med enkelte hygieneoppgaver. 3. Moderat: Jeg trenger hjelp til mange hygieneoppgaver. 4: Alvorlig: Jeg trenger hjelp til de fleste eller alle hygieneoppgaver. 2.7 HÅNDSKRIFT I løpet av den siste uken, har andre vanligvis hatt problemer med å lese håndskriften og: Normal: Ikke i det hele tatt (ingen problemer). 1: Meget lett: Jeg skriver langsomt, klønete eller ujevnt, men alle ord er tydelige. 2: Mild: Noen ord er utydelige og vanskelige å lese. 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller ar du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). 1: Meget lett: Jeg er litt langsom, men utfører disse aktivitetene lett. | |
|---|---|
| 2: Mild: Jeg trenger noen til å hjelpe meg med enkelte hygieneoppgaver. 3. Moderat: Jeg trenger hjelp til mange hygieneoppgaver. 4: Alvorlig: Jeg trenger hjelp til de fleste eller alle hygieneoppgaver. 2.7 HÅNDSKRIFT I løpet av den siste uken, har andre vanligvis hatt problemer med å lese håndskriften og Normal: Ikke i det hele tatt (ingen problemer). 1: Meget lett: Jeg skriver langsomt, klønete eller ujevnt, men alle ord er tydelige. 2: Mild: Noen ord er utydelige og vanskelige å lese. 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| hygieneoppgaver. 3. Moderat: Jeg trenger hjelp til mange hygieneoppgaver. 4: Alvorlig: Jeg trenger hjelp til de fleste eller alle hygieneoppgaver. 2.7 HÅNDSKRIFT I løpet av den siste uken, har andre vanligvis hatt problemer med å lese håndskriften og og vanskelige i lese håndskriften og og vanskelige. 1: Meget lett: Jeg skriver langsomt, klønete eller ujevnt, men alle ord er tydelige. 2: Mild: Noen ord er utydelige og vanskelige å lese. 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| 4: Alvorlig: Jeg trenger hjelp til de fleste eller alle hygieneoppgaver. 2.7 HÅNDSKRIFT I løpet av den siste uken, har andre vanligvis hatt problemer med å lese håndskriften og 0: Normal: Ikke i det hele tatt (ingen problemer). 1: Meget lett: Jeg skriver langsomt, klønete eller ujevnt, men alle ord er tydelige. 2: Mild: Noen ord er utydelige og vanskelige å lese. 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| 2.7 HÅNDSKRIFT I løpet av den siste uken, har andre vanligvis hatt problemer med å lese håndskriften d 0: Normal: Ikke i det hele tatt (ingen problemer). 1: Meget lett: Jeg skriver langsomt, klønete eller ujevnt, men alle ord er tydelige. 2: Mild: Noen ord er utydelige og vanskelige å lese. 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| I løpet av den siste uken, har andre vanligvis hatt problemer med å lese håndskriften den og in state uken, har andre vanligvis hatt problemer med å lese håndskriften den og in state uken. Ikke i det hele tatt (ingen problemer). Ikke i det hele tatt (ingen problemer). Ikke i det hele tatt (ingen problemer). Ikke i det hele tatt (ingen problemer med å lese håndskriften den og ingen problemer). Ikke i det hele tatt (ingen problemer med å utøve hobbyer eller at du liker å gjøre? Ikke i det hele tatt (ingen problemer). | |
| 1: Meget lett: Jeg skriver langsomt, klønete eller ujevnt, men alle ord er tydelige. 2: Mild: Noen ord er utydelige og vanskelige å lese. 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | din? |
| er tydelige. 2: Mild: Noen ord er utydelige og vanskelige å lese. 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| 3: Moderat: Mange ord er utydelige og vanskelige å lese. 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| 4: Alvorlig: De fleste eller alle ordene er uleselige. 2.8 HOBBYER OG ANDRE AKTIVITETER I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| <ul> <li>2.8 HOBBYER OG ANDRE AKTIVITETER</li> <li>I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller at du liker å gjøre?</li> <li>0: Normal: Ikke i det hele tatt (ingen problemer).</li> </ul> | |
| I løpet av den siste uken, har du vanligvis hatt problemer med å utøve hobbyer eller a<br>du liker å gjøre? 0: Normal: Ikke i det hele tatt (ingen problemer). | |
| | ndre ti |
| Meget lett: Jeg er litt langsom, men utfører disse aktivitetene lett. | |
| 2: Mild: Jeg har noen vanskeligheter med å utføre disse aktivitetene. | |
| 3: Moderat: Jeg har store problemer med å utføre disse aktivitetene, men gjør likevel de fleste. | |
| 4: Alvorlig: Jeg er ikke i stand til å utføre de fleste eller alle disse aktivitetene | |

| 2.9 SNU SEG I<br>I løpet av den sis | SENGEN<br>te uken, har du vanligvis hatt problemer med å snu deg i sengen? |
|---|---|
| 0: Normal: | Ikke i det hele tatt (Ingen problemer) |
| 1: Meget lett: | Jeg har noen problemer med å snu meg, men jeg trenger<br>ikke hjelp. |
| 2: Mild: | Jeg har mye problemer med å snu meg, og trenger av og til hjelp fra noen andre. |
| 3: Moderat: | Jeg trenger ofte hjelp fra noen andre for å snu meg. |
| 4: Alvorlig: | Jeg kan ikke snu meg uten hjelp fra andre. |
| 2.10 SKJELV<br>I løpet av den sis | TNG<br>te uken, har du hatt regelmessig skjelving eller risting? |
| 0: Normal: | Ikke i det hele tatt, jeg har ikke skjelvinger eller ristinger. |
| 1: Meget lett: | Ristinger eller skjelvinger forekommer, men forårsaker ikke problemer i noen aktiviteter. |
| 2: Mild: | Ristinger og skjelvinger forårsaker problemer bare i<br>noen få aktiviteter. |
| 3: Moderat: | Ristinger og skjelvinger forårsaker problemer i mange av mine daglige aktiviteter. |
| 4: Alvorlig: | Ristinger eller skjelvinger forårsaker problemer i de fleste eller alle aktiviteter. |
| | E SEG UT AV SENGEN, EN BIL ELLER EN DYP STOL<br>te uken, har du vanligvis hatt problemer med å komme deg ut av sengen,<br>yp stol? |
| 0: Normal: | Ikke i det hele tatt (ingen problemer). |
| 1: Meget lett: | Jeg er langsom eller klossete, men klarer det vanligvis<br>på første forsøk. |
| 2: Mild: | Jeg trenger mer enn ett forsøk eller trenger hjelp av og til. |
| 3: Moderat: | Jeg trenger noen ganger hjelp for å komme opp, men<br>for det meste klarer jeg det fortsatt selv. |
| | Jeg trenger hjelp mesteparten eller hele tiden. |

| 2.12 GANGE ( | OG BALANSE |
|---|---|
| | e uken, har du vanligvis hatt problemer med balanse og gange? |
| 0: Normal: | Ikke i det hele tatt (ingen problemer) |
| 1. Meget lett: | Jeg er litt langsom eller kan dra på et ben. Jeg bruker<br>aldri ganghjelpemidler. |
| 2: Mild: | Jeg bruker av og til et ganghjelpemiddel, men jeg<br>trenger ikke hjelp fra en annen person. |
| 3: Moderat: | Jeg bruker vanligvis et ganghjelpemiddel (stokk, rullator) for å gå trygt uten å falle. Men jeg trenger vanligvis ikke støtte fra en annen person. |
| 4: Alvorlig: | Jeg bruker vanligvis støtte av en annen person for å gå<br>trygt uten å falle. |
| - | NING<br>e uken, på en vanlig dag mens du går, stopper du plutselig eller stivner<br>ne henger fast i gulvet? |
| 0: Normal: | Ikke i det hele tatt (Ingen problemer). |
| 1: Meget lett: | Jeg stivner til kortvarig, men kan lett starte å gå igjen.<br>Jeg trenger ikke hjelp fra andre eller et<br>ganghjelpemiddel (stokk eller rullator) på grunn av<br>tilstivning. |
| 2: Mild: | Jeg stivner til og har problemer med å begynne å gå igjen, men jeg trenger ikke hjelp fra andre eller et ganghjelpemiddel (stokk eller rullator) på grunn av tilstivning. |
| 3: Moderat: | Når jeg stivner til har jeg store problemer med å begynne å gå igjen, og på grunn av tilstivning trenger jeg av og til å bruke et ganghjelpemiddel eller hjelp fra andre. |
| 4: Alvorlig: | På grunn av tilstivning trenger jeg et ganghjelpemiddel eller hjelp av noen mesteparten eller hele tiden. |
| problemer du<br>Ikke alle pasie<br>er det viktig å | n på spørreskjemaet. Det kan hende vi har spurt om<br>ikke har, og kanskje har vi nevnt problemer du aldri vil f<br>nter får alle disse problemene, men fordi de kan forekom<br>stille alle disse spørsmålene til alle pasienter. Tusen takk<br>d og oppmerksomhet på å fullføre dette spørreskjemaet. |

| | Part III: Motor Examination |
|---|---|
| | view: This portion of the scale assesses the motor signs of PD. In administering Part III of the MDS-UPDRS examiner should comply with the following guidelines: |
| | ne top of the form, mark whether the patient is on medication for treating the symptoms of Parkinson's disease if on levodopa, the time since the last dose. |
| | , if the patient is receiving medication for treating the symptoms of Parkinson's disease, mark the patient's cal state using the following definitions: ON is the typical functional state when patients are receiving medication and have a good response. OFF is the typical functional state when patients have a poor response in spite of taking medications. |
| rth<br>Idi<br>Ieg | investigator should "rate what you see." Admittedly, concurrent medical problems such as stroke, paralysis, itis, contracture, and orthopedic problems such as hip or knee replacement and scoliosis may interfere with idual items in the motor examination. In situations where it is absolutely impossible to test (e.g., amputations, ia, limb in a cast), use the notation "UR" for Unable to Rate. Otherwise, rate the performance of each task as the ent performs in the context of co-morbidities. |
| dl i | ems must have an integer rating (no half points, no missing ratings). |
| or<br>ur | cific instructions are provided for the testing of each item. These should be followed in all instances. The stigator demonstrates while describing tasks the patient is to perform and rates function immediately thereafter. Global Spontaneous Movement and Rest Tremor items (3.14 and 3.17), these items have been placed osefully at the end of the scale because clinical information pertinent to the score will be obtained throughout the examination. |
| a | Is the patient on medication for treating the symptoms of Parkinson's disease? |
| b | If the patient is receiving medication for treating the symptoms of Parkinson's disease, mark the patient's clinical state using the following definitions: |
| | $\square$ ON: On is the typical functional state when patients are receiving medication and have a good response. |
| | $\square$ OFF: Off is the typical functional state when patients have a poor response in spite of taking medications. |
| С | Is the patient on levodopa ? |
| | 3.C1 If yes, minutes since last levodopa dose: |

| 3.1 SPEECH | | SCORE |
|---|---|---|
| Instructions to exam<br>necessary. Sugges<br>doctor's office. Eva | miner: Listen to the patient's free-flowing speech and engage in conversation if ted topics: ask about the patient's work, hobbies, exercise, or how he got to the luate volume, modulation (prosody) and clarity, including slurring, palilalia (repetition achyphemia (rapid speech, running syllables together). | |
| 0: Normal: | No speech problems. | |
| 1: Slight: | Loss of modulation, diction, or volume, but still all words easy to understand. | |
| 2: Mild: | Loss of modulation, diction, or volume, with a few words unclear, but the overall sentences easy to follow. | |
| 3: Moderate: | Speech is difficult to understand to the point that some, but not most, sentences are poorly understood. | |
| 4: Severe: | Most speech is difficult to understand or unintelligible. | |
| | miner. Observe the patient sitting at rest for 10 seconds, without talking and also | |
| Instructions to exam | <u>miner</u> : Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous | |
| Instructions to examination while talking. Observed | <u>miner</u> : Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous | |
| Instructions to examiling talking. Observing smiling, and parting | <u>miner</u> : Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous g of lips. | |
| Instructions to exar<br>while talking. Obso<br>smiling, and parting<br>0: Normal: | miner: Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous g of lips. Normal facial expression. | |
| Instructions to example talking. Obsessmiling, and parting 0: Normal: 1: Slight: 2: Mild: | miner: Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous g of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, masked facies present in the lower face as well, namely fewer movements around the mouth, such as less | |
| Instructions to example talking. Obsessmiling, and parting 0: Normal: 1: Slight: 2: Mild: | miner: Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous g of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, masked facies present in the lower face as well, namely fewer movements around the mouth, such as less spontaneous smiling, but lips not parted. | |
| Instructions to examination of the second of | miner: Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous g of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, masked facies present in the lower face as well, namely fewer movements around the mouth, such as less spontaneous smiling, but lips not parted. Masked facies with lips parted some of the time when the mouth is at rest. | |
| Instructions to examination of the second of | miner: Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous g of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, masked facies present in the lower face as well, namely fewer movements around the mouth, such as less spontaneous smiling, but lips not parted. Masked facies with lips parted some of the time when the mouth is at rest. | |
| Instructions to examination of the second of | miner: Observe the patient sitting at rest for 10 seconds, without talking and also erve eye-blink frequency, masked facies or loss of facial expression, spontaneous g of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, masked facies present in the lower face as well, namely fewer movements around the mouth, such as less spontaneous smiling, but lips not parted. Masked facies with lips parted some of the time when the mouth is at rest. | |

| 3.3 RIGIDITY | | SCORE |
|---|---|---|
| a relaxed posit | examiner: Rigidity is judged on slow passive movement of major joints with the patient in ion and the examiner manipulating the limbs and neck. First, test without an activation st and rate neck and each limb separately. For arms, test the wrist and elbow joints | |
| simultaneously<br>activation man | For legs, test the hip and knee joints simultaneously. If no rigidity is detected, use an euver such as tapping fingers, fist opening/closing, or heel tapping in a limb not being to the patient to go as limp as possible as you test for rigidity. | Neck |
| 0: Norma | l: No rigidity. | |
| 1: Slight: | Rigidity only detected with activation maneuver. | |
| 2: Mild: | Rigidity detected without the activation maneuver, but full range of motion is easily achieved. | RUE |
| 3: Moder | ate: Rigidity detected without the activation maneuver; full range of motion is achieved with effort. | |
| 4: Severe | Rigidity detected without the activation maneuver and full range of motion not achieved. | LUE |
| | | RLE |
| | | LLE |
| 3.4 FINGER 1 | **APPINO | |
| Instructions to perform the tas thumb 10 time | examiner: Each hand is tested separately. Demonstrate the task, but do not continue to sk while the patient is being tested. Instruct the patient to tap the index finger on the s as quickly AND as big as possible. Rate each side separately, evaluating speed, itations, halts, and decrementing amplitude. | |
| 0: Norma | I: No problems. | |
| 1: Slight: | Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the tapping movement; b) slight slowing; c) the amplitude decrements near the end of the 10 taps. | R |
| 2: Mild: | Any of the following: a) 3 to 5 interruptions during tapping; b) mild slowing; c) the amplitude decrements midway in the 10-tap sequence. | |
| 3: Moder | ate: Any of the following: a) more than 5 interruptions during tapping or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) the amplitude decrements starting after the 1st tap. | L |
| | : Cannot or can only barely perform the task because of slowing, interruptions, or | |

| 3.5 HA | ND MOVE | MENTS | SCORE |
|---|---|---|---|
| perform<br>bent at<br>AND as<br>her to d | the task w<br>the elbow s<br>quickly as | miner. Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to make a tight fist with the arm so that the palm faces the examiner. Have the patient open the hand 10 times as fully possible. If the patient fails to make a tight fist or to open the hand fully, remind him/each side separately, evaluating speed, amplitude, hesitations, halts, and litude. | |
| 0: | Normal: | No problems. | |
| 1: | Slight: | Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) the amplitude decrements near the end of the task. | R |
| 2: | Mild: | Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowing; c) the amplitude decrements midway in the task. | |
| 3: | Moderate: | Any of the following: a) more than 5 interruptions during the movement or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) the amplitude decrements starting after the 1st open-and-close sequence. | L |
| 4: | Severe: | Cannot or can only barely perform the task because of slowing, interruptions, or decrements. | |
| Instruct<br>perform<br>his/her | ions to exal<br>the task w<br>body with tl | SUPINATION MOVEMENTS OF HANDS miner: Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to extend the arm out in front of the palms down, and then to turn the palm up and down alternately 10 times as fast | |
| Instruct<br>perform<br>his/her<br>and as | ions to exal<br>the task w<br>body with tl | <u>miner</u> : Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to extend the arm out in front of he palms down, and then to turn the palm up and down alternately 10 times as fast sible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and | |
| Instruct<br>perform<br>his/her<br>and as<br>decrem | ions to exal<br>the task w<br>body with the<br>fully as pos | <u>miner</u> : Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to extend the arm out in front of he palms down, and then to turn the palm up and down alternately 10 times as fast sible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and | |
| Instruct<br>perform<br>his/her<br>and as<br>decrem<br>0: | ions to exal<br>the task w<br>body with the<br>fully as pos<br>enting amp | miner: Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to extend the arm out in front of he palms down, and then to turn the palm up and down alternately 10 times as fast sible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and litude. | |
| Instruct<br>perform<br>his/her<br>and as<br>decrem<br>0: | ions to exal<br>the task w<br>body with the<br>fully as posenting amp<br>Normal: | miner: Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to extend the arm out in front of he palms down, and then to turn the palm up and down alternately 10 times as fast sible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and slitude. No problems. Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) the amplitude decrements near | R |
| Instruct<br>perform<br>his/her<br>and as<br>decrem<br>0:<br>1: | the task w<br>body with the fully as posenting amp<br>Normal:<br>Slight: | miner: Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to extend the arm out in front of he palms down, and then to turn the palm up and down alternately 10 times as fast sible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and litude. No problems. Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) the amplitude decrements near the end of the sequence. Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowing; | R |
| Instruct perform his/her and as decrem 0: 1: 2: | the task w<br>body with the fully as posenting amp<br>Normal:<br>Slight: | miner: Test each hand separately. Demonstrate the task, but do not continue to hile the patient is being tested. Instruct the patient to extend the arm out in front of he palms down, and then to turn the palm up and down alternately 10 times as fast sible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and slitude. No problems. Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) the amplitude decrements near the end of the sequence. Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowing; c) the amplitude decrements midway in the sequence. Any of the following: a) more than 5 interruptions during the movement or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) the | R |

| foot separabeing teste he toes 10, hesitation Normal: light: loderate: evere: | iner: Have the patient sit in a straight-backed chair with arms, both feet on the floor. rately. Demonstrate the task, but do not continue to perform the task while the ed. Instruct the patient to place the heel on the ground in a comfortable position and times as big and as fast as possible. Rate each side separately, evaluating speed, as, halts, and decrementing amplitude. No problems. Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the tapping movement; b) slight slowing; c) amplitude decrements near the end of the ten taps. Any of the following: a) 3 to 5 interruptions during the tapping movements; b) mild slowing; c) amplitude decrements midway in the task. Any of the following: a) more than 5 interruptions during the tapping movements or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) amplitude decrements after the 1st tap. Cannot or can only barely perform the task because of slowing, interruptions or decrements. | R |
|---|---|---|
| light: lidd: loderate: evere: AGILITY as to examifeet comfo | Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the tapping movement; b) slight slowing; c) amplitude decrements near the end of the ten taps. Any of the following: a) 3 to 5 interruptions during the tapping movements; b) mild slowing; c) amplitude decrements midway in the task. Any of the following: a) more than 5 interruptions during the tapping movements or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) amplitude decrements after the 1st tap. Cannot or can only barely perform the task because of slowing, interruptions or decrements. | |
| lild: loderate: evere: AGILITY as to exami feet comfo | or hesitations of the tapping movement; b) slight slowing; c) amplitude decrements near the end of the ten taps. Any of the following: a) 3 to 5 interruptions during the tapping movements; b) mild slowing; c) amplitude decrements midway in the task. Any of the following: a) more than 5 interruptions during the tapping movements or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) amplitude decrements after the 1st tap. Cannot or can only barely perform the task because of slowing, interruptions or decrements. | |
| evere: AGILITY as to exami feet comfo | slowing; c) amplitude decrements midway in the task. Any of the following: a) more than 5 interruptions during the tapping movements or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) amplitude decrements after the 1st tap. Cannot or can only barely perform the task because of slowing, interruptions or decrements. | |
| evere: AGILITY as to exami feet comfo | or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) amplitude decrements after the 1st tap. Cannot or can only barely perform the task because of slowing, interruptions or decrements. | L |
| AGILITY us to exami | decrements. iner. Have the patient sit in a straight-backed chair with arms. The patient should | |
| ns to exami<br>feet comfo | <u>iner</u> . Have the patient sit in a straight-backed chair with arms. The patient should | |
| possible. F | | |
| light: | Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) amplitude decrements near the end of the task. | R |
| lild: | Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowness; c) amplitude decrements midway in the task. | |
| loderate: | Any of the following: a) more than 5 interruptions during the movement or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing in speed; c) amplitude decrements after the 1st tap. | |
| evere: | Cannot or can only barely perform the task because of slowing, interruptions, or decrements. | |
| tii<br>Oi<br>Iii | ng amplit<br>mal:<br>ght:<br>d:<br>oderate: | ng amplitude. mal: No problems. ght: Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) amplitude decrements near the end of the task. d: Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowness; c) amplitude decrements midway in the task. deferate: Any of the following: a) more than 5 interruptions during the movement or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing in speed; c) amplitude decrements after the 1st tap. vere: Cannot or can only barely perform the task because of slowing, interruptions, |

This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the Internation and Movement Disorder Society.

| 3.9 ARISING FROM | 1 CHAIR | SCORE |
|---|---|---|
| floor and sitting back<br>across the chest and<br>maximum of two mon<br>with arms folded acro<br>patient to push off us | iner: Have the patient sit in a straight-backed chair with arms, with both feet on the in the chair (if the patient is not too short). Ask the patient to cross his/her arms I then to stand up. If the patient is not successful, repeat this attempt up to a re times. If still unsuccessful, allow the patient to move forward in the chair to arise oss the chest. Allow only one attempt in this situation. If unsuccessful, allow the sing his/her hands on the arms of the chair. Allow a maximum of three trials of it successful, assist the patient to arise. After the patient stands up, observe the | |
| 0: Normal: | No problems. Able to arise quickly without hesitation. | |
| 1: Slight: | Arising is slower than normal; or may need more than one attempt; or may need to move forward in the chair to arise. No need to use the arms of the chair. | |
| 2: Mild: | Pushes self up from the arms of the chair without difficulty. | |
| 3: Moderate: | Needs to push off, but tends to fall back; or may have to try more than one time using the arms of the chair, but can get up without help. | |
| 4: Severe: | Unable to arise without help. | |
| | <u>niner</u> . Testing gait is best performed by having the patient walking away from and<br>er so that both right and left sides of the body can be easily obse <b>rv</b> ed | |
| Instructions to exam<br>towards the examine<br>simultaneously. The<br>the examiner. This if<br>heel strike during wa | | |
| Instructions to exam<br>towards the examine<br>simultaneously. The<br>the examiner. This if<br>heel strike during wa | er so that both right and left sides of the body can be easily observed<br>e patient should walk at least 10 meters (30 feet), then turn around and return to<br>tem measures multiple behaviors: stride amplitude, stride speed, height of foot lift,<br>alking, turning, and arm swing, but not freezing. Assess also for "freezing of gait" | |
| Instructions to exam<br>towards the examine<br>simultaneously. The<br>the examiner. This if<br>heel strike during wa<br>(next item 3.11) whil | er so that both right and left sides of the body can be easily observed expatient should walk at least 10 meters (30 feet), then turn around and return to tem measures multiple behaviors: stride amplitude, stride speed, height of foot lift, alking, turning, and arm swing, but not freezing. Assess also for "freezing of gait" le patient is walking. Observe posture for item 3.13. | |
| Instructions to exam<br>towards the examine<br>simultaneously. The<br>the examiner. This is<br>heel strike during wa<br>(next item 3.11) while<br>0: Normal: | er so that both right and left sides of the body can be easily observed expatient should walk at least 10 meters (30 feet), then turn around and return to tem measures multiple behaviors: stride amplitude, stride speed, height of foot lift, alking, turning, and arm swing, but not freezing. Assess also for "freezing of gait" lee patient is walking. Observe posture for item 3.13. No problems. | |
| Instructions to exam<br>towards the examine<br>simultaneously. The<br>the examiner. This if<br>heel strike during wa<br>(next item 3.11) while<br>0: Normal:<br>1: Slight: | er so that both right and left sides of the body can be easily observed expatient should walk at least 10 meters (30 feet), then turn around and return to tem measures multiple behaviors: stride amplitude, stride speed, height of foot lift, alking, turning, and arm swing, but not freezing. Assess also for "freezing of gait" le patient is walking. Observe posture for item 3.13. No problems. Independent walking with minor gait impairment. | |
| Instructions to exam towards the examines the examiner. This is heel strike during wa (next item 3.11) while 0: Normal: 1: Slight: 2: Mild: | er so that both right and left sides of the body can be easily observed expatient should walk at least 10 meters (30 feet), then turn around and return to term measures multiple behaviors: stride amplitude, stride speed, height of foot lift, alking, turning, and arm swing, but not freezing. Assess also for "freezing of gait" leepatient is walking. Observe posture for item 3.13. No problems. Independent walking with minor gait impairment. Independent walking but with substantial gait impairment. Requires an assistance device for safe walking (walking stick, walker) but not a | |

| episodes. Observe | F GAIT iner: While assessing gait, also assess for the presence of any gait freezing for start hesitation and stuttering movements especially when turning and reaching To the extent that safety permits, patients may NOT use sensory tricks during the | SCORE |
|---|---|---|
| 0: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: | No freezing. Freezes on starting, turning, or walking through doorway with a single halt during any of these events, but then continues smoothly without freezing during straight walking. Freezes on starting, turning, or walking through doorway with more than one halt during any of these activities, but continues smoothly without freezing during straight walking. Freezes once during straight walking. Freezes multiple times during straight walking. | |
| quick, forceful pull of comfortably apart at the patient on what falling. There should observation of the repurposely milder and the examiner with e backwards. The exto allow enough roopatient to flex the both can be backwards or falling ratings begin with the test so that the ratin | iner: The test examines the response to sudden body displacement produced by a not the shoulders while the patient is standing erect with eyes open and feet and parallel to each other. Test retropulsion. Stand behind the patient and instruct is about to happen. Explain that s/he is allowed to take a step backwards to avoid a be a solid wall behind the examiner, at least 1-2 meters away to allow for the umber of retropulsive steps. The first pull is an instructional demonstration and is donot rated. The second time the shoulders are pulled briskly and forcefully towards are nough force to displace the center of gravity so that patient MUST take a step aminer needs to be ready to catch the patient, but must stand sufficiently back so as more for the patient to take several steps to recover independently. Do not allow the oldy abnormally forward in anticipation of the pull. Observe for the number of steps. Up to and including two steps for recovery is considered normal, so abnormal ree steps. If the patient fails to understand the test, the examiner can repeat the g is based on an assessment that the examiner feels reflects the patient's limitations restanding or lack of preparedness. Observe standing posture for item 3.13. No problems. Recovers with one or two steps. 3-5 steps, but subject recovers unaided. More than 5 steps, but with absence of postural response; falls if not caught by examiner. Very unstable, tends to lose balance spontaneously or with just a gentle pull on the shoulders. | |

| 3.13 POSTURE | | |
|---|---|---|
| during walking, and stand up straight and | niner. Posture is assessed with the patient standing erect after arising from a chair, while being tested for postural reflexes. If you notice poor posture, tell the patient to d see if the posture improves (see option 2 below). Rate the worst posture seen in ion points. Observe for flexion and side-to-side leaning. | |
| 0: Normal: | No problems. | |
| 1: Slight: | Not quite erect, but posture could be normal for older person. | |
| 2: Mild: | Definite flexion, scoliosis or leaning to one side, but patient can correct posture to normal posture when asked to do so. | |
| 3: Moderate: | Stooped posture, scoliosis or leaning to one side that cannot be corrected volitionally to a normal posture by the patient. | |
| 4: Severe: | Flexion, scoliosis or leaning with extreme abnormality of posture. | |
| small amplitude and | iner: This global rating combines all observations on slowness, hesitancy, and poverty of movement in general, including a reduction of gesturing and of crossing sment is based on the examiner's global impression after observing for | |
| | es while sitting, and the nature of arising and walking. | |
| spontaneous gesture | es while sitting, and the nature of arising and walking. | |
| spontaneous gesture 0: Normal: | es while sitting, and the nature of arising and walking. No problems. | |
| spontaneous gesture 0: Normal: 1: Slight: | No problems. Slight global slowness and poverty of spontaneous movements. | |
| spontaneous gesture 0: Normal: 1: Slight: 2: Mild: | No problems. Slight global slowness and poverty of spontaneous movements. Mild global slowness and poverty of spontaneous movements. | |
| o: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: 3.15 POSTURAL To Instructions to exame to be included in this patient to stretch the | No problems. Slight global slowness and poverty of spontaneous movements. Mild global slowness and poverty of spontaneous movements. Moderate global slowness and poverty of spontaneous movements. | |
| o: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: 3.15 POSTURAL To be included in this patient to stretch the the fingers comfortat seconds. | No problems. Slight global slowness and poverty of spontaneous movements. Mild global slowness and poverty of spontaneous movements. Moderate global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. REMOR OF THE HANDS iner: All tremor, including re-emergent rest tremor, that is present in this posture is rating. Rate each hand separately. Rate the highest amplitude seen. Instruct the arms out in front of the body with palms down. The wrist should be straight and only separated so that they do not touch each other. Observe this posture for 10 | |
| o: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: 3.15 POSTURAL To Instructions to exame to be included in this patient to stretch the fingers comfortate seconds. 0: Normal: | No problems. Slight global slowness and poverty of spontaneous movements. Mild global slowness and poverty of spontaneous movements. Moderate global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. REMOR OF THE HANDS iner: All tremor, including re-emergent rest tremor, that is present in this posture is rating. Rate each hand separately. Rate the highest amplitude seen. Instruct the arms out in front of the body with palms down. The wrist should be straight and only separated so that they do not touch each other. Observe this posture for 10 No tremor. | R |
| o: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: 3.15 POSTURAL To be included in this patient to stretch the fingers comfortat seconds. | No problems. Slight global slowness and poverty of spontaneous movements. Mild global slowness and poverty of spontaneous movements. Moderate global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. REMOR OF THE HANDS iner: All tremor, including re-emergent rest tremor, that is present in this posture is rating. Rate each hand separately. Rate the highest amplitude seen. Instruct the arms out in front of the body with palms down. The wrist should be straight and only separated so that they do not touch each other. Observe this posture for 10 | R |
| o: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: 3.15 POSTURAL To Instructions to exam to be included in this patient to stretch the the fingers comfortat seconds. 0: Normal: | No problems. Slight global slowness and poverty of spontaneous movements. Mild global slowness and poverty of spontaneous movements. Moderate global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. REMOR OF THE HANDS iner: All tremor, including re-emergent rest tremor, that is present in this posture is rating. Rate each hand separately. Rate the highest amplitude seen. Instruct the arms out in front of the body with palms down. The wrist should be straight and only separated so that they do not touch each other. Observe this posture for 10 No tremor. | R |
| spontaneous gesture 0: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: 3.15 POSTURAL To the included in this patient to stretch the the fingers comfortal seconds. 0: Normal: 1: Slight: | No problems. Slight global slowness and poverty of spontaneous movements. Mild global slowness and poverty of spontaneous movements. Moderate global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. Severe global slowness and poverty of spontaneous movements. REMOR OF THE HANDS iner: All tremor, including re-emergent rest tremor, that is present in this posture is a rating. Rate each hand separately. Rate the highest amplitude seen. Instruct the larms out in front of the body with palms down. The wrist should be straight and only separated so that they do not touch each other. Observe this posture for 10 No tremor. Tremor is present but less than 1 cm in amplitude. | R |

| 3.16 KINETIC TRE | EMOR OF THE HANDS | SCORE |
|---|---|---|
| outstretched position<br>reaching as far as performed slowly e<br>with the other hand | niner: This is tested by the finger-to-nose maneuver. With the arm starting from the on, have the patient perform at least three finger-to-nose maneuvers with each hand possible to touch the examiner's finger. The finger-to-nose maneuver should be nough not to hide any tremor that could occur with very fast arm movements. Repeat , rating each hand separately. The tremor can be present throughout the movement aches either target (nose or finger). Rate the highest amplitude seen. | |
| 0: Normal: | No tremor. | |
| 1: Slight: | Tremor is present but less than 1 cm in amplitude. | R |
| 2: Mild: | Tremor is at least 1 but less than 3 cm in amplitude. | |
| 3: Moderate: | Tremor is at least 3 but less than 10 cm in amplitude. | |
| 4: Severe: | Tremor is at least 10 cm in amplitude. | L |
| | OR AMPLITUDE niner: This and the next item have been placed purposefully at the end of the w the rater to gather observations on rest tremor that may appear at any time during | |
| | , , , | |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. It tude and not the persistence or the intermittency of the tremor. It is patient should sit quietly in a chair with the hands placed on the arms of the part of the comfortably supported on the floor for 10 seconds with no other arms is assessed separately for all four limbs and also for the lip/jaw. Rate only the tent tall seen at any time as the final rating. | RUE |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the o) and the feet comfortably supported on the floor for 10 seconds with no other error is assessed separately for all four limbs and also for the lip/jaw. Rate only the e that is seen at any time as the final rating. | RUE |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplituding the example of the exampl | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the o) and the feet comfortably supported on the floor for 10 seconds with no other error is assessed separately for all four limbs and also for the lip/jaw. Rate only the e that is seen at any time as the final rating. | RUE |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplitude Extremity rating materials and the extremity rating maximum amplitudes. | when quietly sitting, during walking, and during activities when some body parts are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the ) and the feet comfortably supported on the floor for 10 seconds with no other error is assessed separately for all four limbs and also for the lip/jaw. Rate only the e that is seen at any time as the final rating. | |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tremaximum amplitude Extremity rating: 0: Normal: | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the and the feet comfortably supported on the floor for 10 seconds with no other armor is assessed separately for all four limbs and also for the lip/jaw. Rate only the that is seen at any time as the final rating. | |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplitude Extremity rating. O: Normal: 1: Slight: | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the o) and the feet comfortably supported on the floor for 10 seconds with no other ernor is assessed separately for all four limbs and also for the lip/jaw. Rate only the e that is seen at any time as the final rating. No tremor. < 1 cm in maximal amplitude. | LUE |
| the exam, including moving but others a Rate only the ampli As part of this ratin chair (not in the lap directives. Rest tre maximum amplitudi Extremity ratin 0: Normal: 1: Slight: 2: Mild: | when quietly sitting, during walking, and during activities when some body parts are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the of any and the feet comfortably supported on the floor for 10 seconds with no other emor is assessed separately for all four limbs and also for the lip/jaw. Rate only the entity is seen at any time as the final rating. No tremor. < 1 cm in maximal amplitude. ≥ 1 cm but < 3 cm in maximal amplitude. | |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplitude Extremity rating. O: Normal: 1: Slight: 2: Mild: 3: Moderate: | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the and the feet comfortably supported on the floor for 10 seconds with no other arms is assessed separately for all four limbs and also for the lip/jaw. Rate only the that is seen at any time as the final rating. No tremor. < 1 cm in maximal amplitude. ≥ 1 cm but < 3 cm in maximal amplitude. ≥ 3 cm but < 10 cm in maximal amplitude. ≥ 10 cm in maximal amplitude. | LUE |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplitude Extremity ratin 0: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the and the feet comfortably supported on the floor for 10 seconds with no other arms is assessed separately for all four limbs and also for the lip/jaw. Rate only the that is seen at any time as the final rating. No tremor. < 1 cm in maximal amplitude. ≥ 1 cm but < 3 cm in maximal amplitude. ≥ 3 cm but < 10 cm in maximal amplitude. ≥ 10 cm in maximal amplitude. | LUE |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplituding Extremity rating 0: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: Lip/Jaw rating | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the and the feet comfortably supported on the floor for 10 seconds with no other emor is assessed separately for all four limbs and also for the lip/jaw. Rate only the entat is seen at any time as the final rating. No tremor. < 1 cm in maximal amplitude. ≥ 1 cm but < 3 cm in maximal amplitude. ≥ 3 cm but < 10 cm in maximal amplitude. ≥ 10 cm in maximal amplitude. | LUE |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplituding Extremity rating 0: Normal: 1: Slight: 2: Mild: 3: Moderate: 4: Severe: Lip/Jaw rating 0: Normal: | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the o) and the feet comfortably supported on the floor for 10 seconds with no other emor is assessed separately for all four limbs and also for the lip/jaw. Rate only the e that is seen at any time as the final rating. In the patient should sit quietly in a chair with the hands placed on the arms of the o) and the feet comfortably supported on the floor for 10 seconds with no other emor is assessed separately for all four limbs and also for the lip/jaw. Rate only the e that is seen at any time as the final rating. So No tremor. In the final rating are the final rating are the final rating are the final rating and the final rating are the final r | LUE |
| the exam, including moving but others a Rate only the ampli As part of this rating chair (not in the lap directives. Rest tre maximum amplitude Extremity rating. 1: Slight: 2: Mild: 3: Moderate: 4: Severe: Lip/Jaw rating. 0: Normal: 1: Slight: | when quietly sitting, during walking, and during activities when some body parts are are at rest. Score the maximum amplitude that is seen at any time as the final score. tude and not the persistence or the intermittency of the tremor. g, the patient should sit quietly in a chair with the hands placed on the arms of the and the feet comfortably supported on the floor for 10 seconds with no other armor is assessed separately for all four limbs and also for the lip/jaw. Rate only the that is seen at any time as the final rating. No tremor. < 1 cm in maximal amplitude. ≥ 1 cm but < 3 cm in maximal amplitude. ≥ 10 cm in maximal amplitude. S No tremor. < 1 cm in maximal amplitude. | LUE |

This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| ns to examinemor during to all the end. Normal: Normal: Normal: Noderate: Severe: Severe: | Ton Part III ratings Ton Part III ratings esias (chorea or dystonia) present during examination? Ton Part III ratings esias (chorea or dystonia) present during examination? To No Dart III ratings esias (chorea or dystonia) present durings? Ton Part III ratings Ton Part III ratings Ton Part III ratings | |
|---|---|---|
| Slight: Mild: Moderate: Severe: ESIA IMPAC Were dyskine | Tremor at rest is present ≤ 25% of the entire examination period. Tremor at rest is present 26-50% of the entire examination period. Tremor at rest is present 51-75% of the entire examination period. Tremor at rest is present > 75% of the entire examination period. Ton Part III ratings esias (chorea or dystonia) present during examination? □ No □ Yes | |
| Mild: Moderate: Severe: ESIA IMPAC Were dyskine | Tremor at rest is present 26-50% of the entire examination period. Tremor at rest is present 51-75% of the entire examination period. Tremor at rest is present > 75% of the entire examination period. TON PART III RATINGS esias (chorea or dystonia) present during examination? | |
| Moderate: Severe: ESIA IMPAC Were dyskine | Tremor at rest is present 51-75% of the entire examination period. Tremor at rest is present > 75% of the entire examination period. T ON PART III RATINGS esias (chorea or dystonia) present during examination? | |
| Severe: ESIA IMPAC Were dyskine | Tremor at rest is present > 75% of the entire examination period. T ON PART III RATINGS esias (chorea or dystonia) present during examination? | |
| ESIA IMPAC<br>Were dyskine | T ON PART III RATINGS esias (chorea or dystonia) present during examination? | |
| Were dyskine | esias (chorea or dystonia) present during examination? | |
| f yes, did the | ese movements interfere with your ratings? | |
| symptomatic | z. | |
| ilateral involv | mement without impairment of balance. | |
| evere disabi | lity; still able to walk or stand unassisted. | |
| /heelchair bo | ound or bedridden unless aided. | |
| | symptomation involvillateral involvillateral involvillateral involvillateral involvillateral involvessistance to evere disabilitation. | AND YAHR STAGE symptomatic. nilateral involvement only. ilateral involvement without impairment of balance. liid to moderate involvement; some postural instability but physically independent; needs sistance to recover from pull test. evere disability; still able to walk or stand unassisted. //heelchair bound or bedridden unless aided. |

#### Part IV: Motor Complications

Overview and Instructions: In this section, the rater uses historical and objective information to assess two motor complications, dyskinesias and motor fluctuations that include OFF-state dystonia. Use all information from patient, caregiver, and the examination to answer the six questions that summarize function over the past week including today. As in the other sections, rate using only integers (no half points allowed) and leave no missing ratings. If the item cannot be rated, place "UR" for Unable to Rate. You will need to choose some answers based on percentages, and therefore you will need to establish how many hours the patient is generally awake and use this figure as the denominator for "OFF" time and dyskinesias. For "OFF dystonia", the total "OFF" time will be the denominator. Operational definitions for examiner's use.

Dyskinesias: Involuntary random movements:

Words that patients often recognize for dyskinesias include "irregular jerking", "wiggling", "twitching." It is essential to stress to the patient the difference between dyskinesias and tremor, a common error when patients are assessing dyskinesias.

Dystonia: Contorted posture, often with a twisting component: Words that patients often recognize for dystonia include "spasms", "cramps", "posture."

Motor fluctuation: Variable response to medication:

Words that patients often recognize for motor fluctuation include "wearing out", "wearing off", "roller-coaster effect", "on-off", "uneven medication effects."

OFF: Typical functional state when patients have a poor response in spite of taking mediation or the typical functional response when patients are on NO treatment for parkinsonism. Words that patients often recognize include "low time", "bad time", "shaking time", "slow time", "time when my medications don't work."

ON: Typical functional state when patients are receiving medication and have a good response:

Words that patients often recognize include "good time", "walking time", "time when my medications work."

#### A. DYSKINESIAS [exclusive of OFF-state dystonia]

| 4.1 TIME SPENT WITH DYSKINESIAS | |
|---|---|
| Instructions to examiner: Determine the hours in the using dyskinesias. Calculate the percentage. If the patient has out as a reference to ensure that patients and caregivers use your own acting skills to enact the dyskinetic movem show them dyskinetic movements typical of other patient and nighttime painful dystonia. | s dyskinesias in the office, you can point them understand what they are rating. You may also lents you have seen in the patient before or ts. Exclude from this question early morning |
| Instructions to patient [and caregiver]: Over the past week, how many hours do you usually sleep on a daily basis, including nighttime sleep and daytime napping? Alright, if you sleep hrs, you are awake hrs. Out of those awake hours, how many hours in total do you have wiggling, twitching, or jerking movements? Do not count the times when you have tremor, which is a regular back and forth shaking or times when you have painful foot cramps or spasms in the early moming or at nighttime. I will ask about those later. Concentrate only on these types of wiggling, jerking, and irregular movements. Add up all the time during the waking day when these usually occur. How many hours (use this number for your calculations). | |
| 0: Normal: No dyskinesias. | |
| 1: Slight: ≤ 25% of waking day. | |
| 2: Mild: 26 - 50% of waking day. | Total Hours Awake: |
| 3: Moderate: 51 - 75% of waking day. | Total Hours with Dyskinesia: |
| 4: Severe: > 75% of waking day. | 3. % Dyskinesia = ((2/1)*100): |

Last updated August 13, 2019 | Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 2'
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| 4.2 FUNCTIONAL II | MPACT OF DYSKINESIAS | | 00055 |
|---|---|---|---|
| instructions to exam<br>function in terms of a | iner: Determine the degree to which dysk | patient's and caregiver's response to your | SCORE |
| | nen these jerking movements occurred? D | I you usually have trouble doing things or<br>old they stop you from doing things or | |
| 0: Normal: | No dyskinesias or no impact by dyskin | nesias on activities or social interactions. | |
| 1: Slight: | Dyskinesias impact on a few activities activities and participates in all social | , but the patient usually performs all interactions during dyskinetic periods. | |
| 2: Mild: | Dyskinesias impact on many activities activities and participates in all social | , but the patient usually performs all interactions during dyskinetic periods. | |
| 3: Moderate: | • | e point that the patient usually does not sually participate in some social activities | |
| 4: Severe: | Dyskinesias impact on function to the<br>perform most activities or participate i<br>dyskinetic episodes. | point that the patient usually does not in most social interactions during | |
| | B. MOTOR FLUC | CTUATIONS | |
| spent in the "OFF" st<br>can point to this state | ner: Use the number of waking hours deri<br>ate. Calculate the percentage. If the patie<br>as a reference. You may also use your k<br>Additionally you may use your own acting | ent has an OFF period in the office, you knowledge of the patient to describe a | |
| seen in the patient be<br>number of OFF hours<br>Instructions to patien<br>their medications thr<br>medications but still<br>these low periods "O<br>hrs each day. Out of | efore or show them OFF function typical of the control of the cont | kinson's disease have a good effect from at "ON" time. Other patients take their low time, or shaking time. Doctors call be before that you are generally awakeotal do you usually have this type of low | |
| seen in the patient be<br>number of OFF hours<br>Instructions to patien<br>their medications that<br>medications but still<br>these low periods "O<br>hrs each day. Out of<br>level or OFF function | is, because you will need this number for o<br>t [and caregiver]: Some patients with Parioughout their awake hours and we call that<br>have some hours of low time, bad time, si<br>FF" time. Over the past week, you told me<br>these awake hours, how many hours in to | completing 4.6. kinson's disease have a good effect from at "ON" time. Other patients take their low time, or shaking time. Doctors call be before that you are generally awakeotal do you usually have this type of low | |
| teen in the patient be<br>number of OFF hours<br>instructions to patien<br>their medications that<br>medications but still<br>these low periods "O<br>hars each day. Out of<br>evel or OFF function | is, because you will need this number for of tand caregiver]: Some patients with Parisughout their awake hours and we call the have some hours of low time, bad time, si FF" time. Over the past week, you told me these awake hours, how many hours in to? (use this number for your calculated) | completing 4.6. kinson's disease have a good effect from at "ON" time. Other patients take their low time, or shaking time. Doctors call be before that you are generally awakeotal do you usually have this type of low | |
| instructions to patient be<br>instructions to patien<br>their medications that<br>medications but still<br>these low periods "O<br>ins each day. Out of<br>evel or OFF function<br>0: Normal: | is, because you will need this number for of tand caregiver]: Some patients with Parkunghout their awake hours and we call the have some hours of low time, bad time, so FF" time. Over the past week, you told me these awake hours, how many hours in to? (use this number for your calculation. | completing 4.6. kinson's disease have a good effect from at "ON" time. Other patients take their low time, or shaking time. Doctors call be before that you are generally awakeotal do you usually have this type of low | |
| wheen in the patient becaumber of OFF hours Instructions to patient their medications but still these low periods "Ones each day. Out of evel or OFF functions 1: Slight: | is, because you will need this number for of the fand caregiver]: Some patients with Park paydout their awake hours and we call the have some hours of low time, bad time, significantly from the factor of the fac | completing 4.6. kinson's disease have a good effect from at "ON" time. Other patients take their ow time, or shaking time. Doctors call be before that you are generally awake otal do you usually have this type of low ions). | |
| teen in the patient becaumber of OFF hours Instructions to patien their medications that medications but still these low periods "O ars each day. Out of evel or OFF function 0: Normal: 1: Slight: 2: Mild: | is, because you will need this number for of tand caregiver]: Some patients with Parioughout their awake hours and we call that have some hours of low time, bad time, silf="f" time. Over the past week, you told me these awake hours, how many hours in to? (use this number for your calculated to the call time. No OFF time. ≤ 25% of waking day. | completing 4.6. kinson's disease have a good effect from at "ON" time. Other patients take their low time, or shaking time. Doctors call be before that you are generally awakeotal do you usually have this type of low | |

Last updated August 13, 2019 | Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 28
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| | NCTIONAL II | MPACT OF FLUCTUATIONS | SCORE |
|---|---|---|---|
| Instructi<br>function<br>betweer<br>patients<br>occurs. | ions to examination terms of and the ON state in the the the patie | ner: Determine the degree to which motor fluctuations impact on the patient's daily ctivities and social interactions. This question concentrates on the difference e and the OFF state. If the patient has no OFF time, the rating must be 0, but if ild fluctuations, it is still possible to be rated 0 on this item if no impact on activities nt's and caregiver's response to your question and your own observations during e at the best answer. | |
| the pas<br>the rest | t week. Do yo<br>of the day wh | t <u>[and_caregiver]</u> : Think about when those low or "OFF" periods have occurred over<br>ou usually have more problems doing things or being with people than compared to<br>len you feel your medications working? Are there some things you usually do<br>that you have trouble with or stop doing during a low period? | |
| 0: | Normal: | No fluctuations or no impact by fluctuations on performance of activities or social interactions. | |
| 1: | Slight: | Fluctuations impact on a few activities, but during OFF, the patient usually performs all activities and participates in all social interactions that typically occur during the ON state. | |
| 2: | Mild: | Fluctuations impact many activities, but during OFF, the patient still usually performs all activities and participates in all social interactions that typically occur during the ON state. | |
| 3: | Moderate: | Fluctuations impact on the performance of activities during OFF to the point that the patient usually does not perform some activities or participate in some social interactions that are performed during ON periods. | |
| 4: | Severe: | Fluctuations impact on function to the point that, during OFF, the patient usually does not perform most activities or participate in most social interactions that are performed during ON periods. | |
| 4.5 CO | MPLEXITY O | F MOTOR FLUCTUATIONS | |
| | ione to evami | | |
| of day, i<br>supplem<br>a specia<br>from mil | food intake, o<br>nent with your<br>al time, mostly<br>Id), only some | ner: Determine the usual predictability of OFF function whether due to dose, time r other factors. Use the information provided by the patients and caregivers and r own observations. You will ask if the patient can count on them always coming at a coming at a special time (in which case you will probe further to separate slight etimes coming at a special time, or are they totally unpredictable? Narrowing down llow you to find the correct answer. | |
| of day, is supplem a special from mile the percentage of the supplementage of the supplementa | food intake, on the ment with your all time, mostly id), only some centage will all ions to patient uring day or when your low to they mostly | r other factors. Use the information provided by the patients and caregivers and r own observations. You will ask if the patient can count on them always coming at y coming at a special time (in which case you will probe further to separate slight etimes coming at a special time, or are they totally unpredictable? Narrowing down | |
| of day, supplem a special from milithe perconstruction in the perconstruction of the special from the perconstruction of the special from the | food intake, or nent with your al time, mostly Id), only some centage will al tions to patient uring day or when your low or they mostly w periods total | r other factors. Use the information provided by the patients and caregivers and r own observations. You will ask if the patient can count on them always coming at y coming at a special time (in which case you will probe further to separate slight etimes coming at a special time, or are they totally unpredictable? Narrowing down llow you to find the correct answer. If and caregiver: For some patients, the low or "OFF" periods happen at certain when they do activities like eating or exercising. Over the past week, do you usually periods will occur? In other words, do your low periods always come at a certain ty come at a certain time? Do they only sometimes come at a certain time? Are | |
| of day, supplem a specia from mil the perconstruct. Instruct. times die know with time? Le your low | food intake, or nent with your al time, mostly ld), only some centage will al tions to patient uring day or when your low to periods total. Normal: | r other factors. Use the information provided by the patients and caregivers and r own observations. You will ask if the patient can count on them always coming at y coming at a special time (in which case you will probe further to separate slight etimes coming at a special time, or are they totally unpredictable? Narrowing down llow you to find the correct answer. If and caregiver: For some patients, the low or "OFF" periods happen at certain when they do activities like eating or exercising. Over the past week, do you usually periods will occur? In other words, do your low periods always come at a certain time? Do they only sometimes come at a certain time? Are lly unpredictable?" | |
| of day, supplem a specia from mil the percular times di know whitime? Le your low 0: | food intake, or nent with your al time, mostly Id), only some centage will al ions to patient uring day or when your low to they mostly v periods total. Normal: Slight: | r other factors. Use the information provided by the patients and caregivers and r own observations. You will ask if the patient can count on them always coming at y coming at a special time (in which case you will probe further to separate slight etimes coming at a special time, or are they totally unpredictable? Narrowing down llow you to find the correct answer. If and caregiver: For some patients, the low or "OFF" periods happen at certain when they do activities like eating or exercising. Over the past week, do you usually periods will occur? In other words, do your low periods always come at a certain ty come at a certain time? Do they only sometimes come at a certain time? Are lly unpredictable?" No motor fluctuations. | |
| of day, supplem a specia from mil the perconnected times disknow what time? Let your low 0: | food intake, or nent with your al time, mostly Id), only some centage will al time to patient uring day or when your low your low your low your low your low. Normal: Slight: Mild: | r other factors. Use the information provided by the patients and caregivers and r own observations. You will ask if the patient can count on them always coming at y coming at a special time (in which case you will probe further to separate slight etimes coming at a special time, or are they totally unpredictable? Narrowing down llow you to find the correct answer. It fand caregiver]: For some patients, the low or "OFF" periods happen at certain then they do activities like eating or exercising. Over the past week, do you usually periods will occur? In other words, do your low periods always come at a certain time? Do they only sometimes come at a certain time? Are lly unpredictable?" No motor fluctuations. OFF times are predictable all or almost all of the time (> 75%). | |

Last updated August 13, 2019 | Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 25
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| 4.6 PAINFUL OFF | -STATE DYSTONIA | | |
|---|---|---|---|
| OFF episodes usua<br>"OFF" time (4.3). O | ally includes painful dystonia? You h | fluctuations, determine what proportion of the<br>lave already determined the number of hours of<br>are associated with dystonia and calculate the | |
| have hours of<br>these low or "OFF" | flow or "OFF" time when your Parki<br>periods, do you usually have painfu | estions I asked earlier, you said you generally<br>nson's disease is under poor control. During<br>Il cramps or spasms? Out of the total hrs<br>hese painful cramps come, how many hours wo | |
| 0: Normal: | No dystonia OR NO OFF TIME. | | |
| 1: Slight: | ≤ 25% of time in OFF state. | | |
| 2: Mild: | 26-50% of time in OFF state. | | |
| 3: Moderate: | 51-75% of time in OFF state. | | |
| 4: Severe: | > 75% of time in OFF state. | | |
| | | 1. Total Hours OFF: | - |
| | | Total OFF Hours with Dystonia: | - |
| | | 3. % OFF Dystonia = ((2/1)*100): | - |
| | rating of your Parkinson's disease. | <u>o patient</u> : READ TO PATIENT<br>. I know the questions and tasks have taken se<br>. In doing so, I may have asked about problems | |
| even have, and I n<br>problems, but beca | nay have mentioned problems that y | you may never develop at all. Not all patients d<br>to ask all the questions to every patient. Thank | evelop all these |

| Patient Name or Subject ID | | Site ID | | | (mm-dd-yyyy)<br>Assessment Date | Inves | estigator's Initials | | |
|---|---|---|---|---|---|---|---|---|---|
| IDS | UPDRS Score Sheet | | | | | | | | |
| | | | Patier | nt | | 3.3b | Rigidity- RUE | | |
| 1.A | Source of information | | | Caregiver | | 3.3c | Rigidity- LUE | | |
| ) T | | Ш | Patier | Patient + Caregiver | | | | | |
| 2art I<br>1.1 | T | _ | | | | 3.3d<br>3.3e | Rigidity- RLE<br>Rigidity- LLE | | |
| 1.2 | Cognitive impairment Hallucinations and psychosis | | | | | 3.4a | | | |
| 1.3 | Hallucinations and psychosis Depressed mood | | | | 3.4b | Finger tapping- Right hand Finger tapping- Left hand | | | |
| 1.4 | Anxious mood | | | | | 3.5a | Hand movements – Right hand | | |
| 1.5 | Apathy | | | | | 3.5b | Hand movements - Left hand | | |
| 1.6 | Features of DDS | | | | | 3.6a | Pronation- supination movements- Right | | |
| 1.0 | r catales of DDO | - | Datio | Patient<br>Caregiver<br>Patient + Caregiver | | 3.6b | Pronation- supination movements – Right | | |
| 1.6a | Who is filling out questionnaire | | Care | | | 3.7a | Toe tapping- Right foot | and . | |
| 1.7 | Sleep problems | | | | | 3.7b | Toe tapping- Left foot | | |
| 1.8 | Daytime sleepiness | | | | | 3.8a | Leg agility-Right leg | | |
| 1.9 | Pain and other sensations | | | | | 3.8b | Leg agility-Left leg | | |
| 1.10 | Urinary problems | | | | | 3.9 | Arising from chair | | |
| 1.11 | Constipation problems | | | | | 3.10 | Gait | | |
| 1.12 | Light headedness on standing | | | | | 3.11 | Freezing of gait | | |
| 1.13 | Fatigue | | | | | 3.12 | Postural stability | | |
| Part I | | - | | | | 3.13 | Posture | | |
| 2.1 | Speech | | | | | 3.14 | Global spontaneity of movement | | |
| 2.2 | Saliva and drooling | | | | | 3.15a | Postural tremor-Right hand | | |
| 2.3 | Chewing and swallowing | | | | | 3.15b | Postural tremor-Left hand | | |
| 2.4 | Eating tasks | | | | | 3.16a | Kinetic tremor-Right hand | | |
| 2.5 | Dressing | | | | | 3.16b | Kinetic tremor-Left hand | | |
| 2.6 | Hygiene | | | | | 3.17a | Rest tremor amplitude- RUE | | |
| 2.7 | Handw riting | | | | | 3.17b | Rest tremor amplitude- LUE | | |
| 2.8 | Doing hobbies and other activities | | | | | 3.17c | Rest tremor amplitude- RLE | | |
| 2.9 | Turning in bed | | | | | 3.17d | Rest tremor amplitude- LLE | | |
| 2.10 | Tremor | | | | | 3.17e | Rest tremor amplitude- Lip/jaw | | |
| 2.11 | Getting out of bed | | | | | 3.18 | Constancy of rest tremor | | |
| 2.12 | Walking and balance | | | | | | Were dyskinesias present? | | ☐ No ☐ Yes |
| 2.13 | Freezing | | | | | | Did these movements interfere with rating | gs? | □ No □ Yes |
| 3a | Is the patient on medication? | F | No | | Yes | | Hoehn and Yahr Stage | | |
| 3b | Patient's clinical state | 늗 | Off | = | On | Part IV | 7 | | |
| 3c | Is the patient on levodopa? | F | No | _ | Yes | 4.1 | Time spent with dyskinesias | | |
| 3.C1 | If yes, minutes since last dose: | ۲ | J | <u> </u> | | 4.2 | Functional impact of dyskinesias | | |
| Part I | | | | | | 4.3 | Time spent in the OFF state | | |
| 3.1 | Speech | | | | | 4.3 | Functional impact of fluctuations | | |
| 3.1 | | | | | | 4.4 | - | | |
| 3.2<br>3.3a | Facial expression Rigidity- Neck | | | | | 4.5 | Complexity of motor fluctuations Painful OFF-state dystonia | | |

#### 3 MDS-NMS

International Parkinson and Movement Disorder Society - Non-Motor Rating Scale

MDS-NMS - Page 1



#### MDS-NMS - Page 2

#### **MDS Permissions**

The International Parkinson and Movement Disorder Society – Non-Motor Rating Scale (MDS-NMS) is owned and licensed by the International Parkinson and Movement Disorder Society (MDS). Permission is required to use the scale and can be obtained by submitting a Permissions Request Form on the MDS website. For licensing inquiries, please e-mail info@movementdisorders.org.

Unauthorized reproduction, distribution, translation, or sale of any portion of the MDS-NMS is strictly prohibited. Changes, modifications, and derivative works of the scale are not permitted without the express authorization of MDS. Including but not limited to the following, the MDS-NMS may not be incorporated into clinical trials, training materials, certification programs, software programs, electronic platforms, electronic medical records, databases, or devices except by permission of MDS.

Copyright © 2019 International Parkinson and Movement Disorder Society. All rights reserved.
| Patier | | Non-Motor Rating Scale (MDS-NMS) |
|---|---|---|
| Patier | | RATER-ADMINISTERED VERSION |
| Patier | | Rate symptoms over past 4 weeks |
| | nt Name or Iden | tifier: |
| Date: | | |
| Respo | ondent: | ☐ Patient ☐ Informant/Caregiver ☐ Patient and Informant |
| Patier | nt's motor state: | □ On □ Off |
| Δ.,, | rada Eraduana | SCORING |
| 0: | Never | y / Duration: (percentages denote days per week or hours per waking day) |
| 1: | Rarely | (≤ 10% of time) |
| 2: | Sometimes | (11-25% of time) |
| 3: | Frequently | (26-50% of time) |
| 4: | | e (≥ 51% of time) |
| Ave | rage Severity: | |
| 0: | Not present | (only if frequency = 0) |
| 1: | Minimal | (no distress or disturbance to patient or caregiver) |
| 2: | Mild | (minor distress or disturbance to patient or caregiver) |
| 3: | Moderate | (considerable distress or disturbance to patient or caregiver) |
| 4: | Severe | (major distress or disturbance to patient or caregiver) |
| Calc | culations: | |
| Item | Total | = Frequency multiplied by severity |
| | scale Total | = Sum of all Item totals for that Subscale |
| | | core = Sum of totals for Subscales A-M |

### International Parkinson and Movement Disorder Society -Non-Motor Rating Scale (MDS-NMS) RATER-ADMINISTERED VERSION Rate symptoms over past 4 weeks Frequency Severity Frequency (0-4)(0-4)x severity A. Depression: 1. Felt sad or depressed? ..... Had difficulty experiencing pleasure?..... 3. Felt hopeless? 4. Had negative thoughts about yourself?..... 5. Felt that life is not worth living? ..... Subscale A Total B. Anxiety: 1. Felt worried? 2. Felt nervous?..... 3. Had panic or anxiety attacks?..... 4. Been worried about being in public or in social situations?..... Subscale B Total C. Apathy: 1. Had a reduced motivation to start day-to-day activities? ..... 2. Had a reduced interest in talking to people? ..... 3. Had a reduction in experiencing emotions?..... Subscale C Total D. Psychosis: 1. Sensed things or people in margins of your visual field? (passage or presence phenomena)..... Visually misinterpreted an actual object? (illusions) ...... 3. Seen, heard, felt, tasted, or smelled things that other people did not? (hallucinations)..... 4. Believed things to be true that others did not? (e.g., delusions of persecution, jealousy, or misidentification) ........ Subscale D Total E. Impulse Control and Related Disorders: 1. Had an increase in gambling, sexual, buying, or eating behaviors? 2. Had an increase in other behaviors (e.g., internet use, hobbies, artistic activities, writing, hoarding)?..... 3. Repeatedly handled objects without any purpose? (punding) .......... 4. Routinely taken more anti-parkinsonian medications than prescribed? (dopamine dysregulation syndrome)..... Subscale E Total Copyright © 2019 International Parkinson and Movement Disorder Society. All rights reserved. | Version 1.0

# International Parkinson and Movement Disorder Society – Non-Motor Rating Scale (MDS-NMS)

| | Frequency | - | |
|---|---|---|---|
| F. Cognition: | (0-4) | (0-4) | x severity |
| Had difficulty remembering things? | | | |
| 2. Had difficulty learning new things? | | | |
| 3. Had difficulty keeping focus or paying attention? | | | |
| 4. Had difficulty finding words or expressing ideas? | 🗀 | | |
| Had difficulty planning or carrying out complex tasks, not due to motor problems? (executive abilities) | | | |
| 6. Had difficulty judging the position of things? (visuospatial | | | |
| abilities) | Subscale | F Total | |
| G. Orthostatic Hypotension: | | | |
| Felt lightheaded or fainted when changing position? | | | |
| Had dizziness or weakness upon standing? | | | |
| | Subscale | G Total | |
| H. Urinary: | | | |
| Had an urgent need to empty bladder? (urinary urgency) | | | |
| 2. Had to empty bladder more than every 2 hours? | | | |
| (urinary frequency) | | | |
| Had to empty bladder more than twice overnight? (nocturia) | Subscale | H Total | |
| I. Sexual: | | | |
| Had decreased sexual drive or interest in sex? | | | |
| Had difficulty with sexual arousal (e.g., erectile dysfunction or | | | |
| vaginal dryness) or sexual performance not related to motor | | | |
| problems (e.g., not related to Parkinson's rigidity)? | Subscale | LTotal | |
| | 000 | | |
| J. Gastrointestinal: | | | |
| 1. Had any drooling of saliva? | | | |
| 2. Had difficulty swallowing? | | | |
| Had nausea or felt sick in the stomach? | | | |
| 4. Had constipation? (defined as < 3 bowel movements/week) | Subscale | <b>↓</b> | |

# International Parkinson and Movement Disorder Society – Non-Motor Rating Scale (MDS-NMS)

| | , | | |
|---|---|---|---|
| RATER-ADMINISTERED VERSION | ON | | |
| Rate symptoms over past 4 we | eks | | |
| Rate symptoms over past 4 we C. Sleep and Wakefulness: Had difficulty falling asleep or staying asleep? (insomnia) | Frequency (0-4) | (0-4) | Frequency x severity |
| Section 9 | | le K Total | |
| Pain: | | | |
| . Had muscle, joint, or back pain? | | | |
| . Had a deep or dull aching pain within the body? | | | |
| . Had pain due to abnormal twisting movements of arms or legs or body, often present in the early morning period? (dystonia) | | | |
| . Had other types of pain? (e.g., nocturnal pain, orofacial pain) | | | |
| 1. Other: | Subsca | le L Total | |
| . Had an unintentional weight loss? (rate frequency as either not present (0) or present (4); for severity rate 0 (only if frequency = 0), 1 (minimal), 2 (mild), 3 (moderate), or 4 (severe)) | | | |
| 3 (moderate), or 4 (severe)) | . | | |
| . Felt excessively physically tired? (physical fatigue) | | $\vdash$ | |
| . Felt excessively mentally tired? (mental fatigue) | | | |
| . Had excessive sweating not related to temperature? | <b>I</b> | le M Total | |
| MDS-NMS TOTAL SCORE | | | |
| pyright © 2019 International Parkinson and Movement Disorder Society. All rights reserved. | Version 1.0 | | 4 |

#### International Parkinson and Movement Disorder Society -Non-Motor Rating Scale (MDS-NMS) RATER-ADMINISTERED VERSION Rate symptoms over past 4 weeks MDS-NMS Non-Motor Fluctuations (NMF) Subscale Do you / Does the patient experience changes in non-motor symptoms (as listed below) in relation to the timing of anti-parkinsonian medications (i.e., symptoms occurring or worsening during "Off" period)? Yes □ No If no, MDS-NMS NMF Total Score (below) = 0 If yes, please complete the following section: **SCORING** Typical degree of change from "On" to "Off" period: No change Minimal 1: Small 3: Medium Large Subscore "Change" = Sum of all "Degree of change" items MDS-NMS NMF Total Score = Subscore "Change" multiplied by Subscore "Time" Degree of change (0-4) Depression (as listed in Subscale A)..... 3. Thinking or cognitive abilities (as listed in Subscale F)..... Bladder symptoms (as listed Subscale H)...... 5. Restlessness (as listed in Subscale K, item 4)..... 6. Pain (as listed in Subscale L)..... 7. Fatigue (as listed in Subscale M, items 3 and 4)..... 8. Excessive sweating (as listed in Subscale M, item 5)..... MDS-NMS NMF Time spent in non-motor "Off" state: Subscore "Change" Rarely (≤ 10% of waking day) 2: Sometimes (11-25% of waking day) MDS-NMS NMF Subscore "Time" Frequently (26-50% of waking day) Majority of time (≥ 51% of waking day) MDS-NMS NMF Total Score (Subscore "Change" x "Time") Copyright © 2019 International Parkinson and Movement Disorder Society. All rights reserved. | Version 1.0

| | ore Sheet | | |
|---|---|---|---|
| RATER-ADMINISTE | RED VERSION | | |
| Item Total = Frequency r | | | |
| Subscale Total = Sum of all Ite | | | |
| MDS-NMS Total Score = Sum | of Lotals for Su | oscales A-M | |
| Respondent: | ant/Caregiver | ☐ Patient and | I Informant |
| Patient's motor state: On Off | J | | |
| A. Depression | Frequency | Severity | Total |
| 1. Sad or depressed | | | |
| 2. Experiencing pleasure | | | |
| 3. Hopelessness | | | |
| 4. Negative thoughts | | | |
| 5. Life not worth living | | | |
| Depression Subscale Total | | | |
| • | | | |
| B. Anxiety | Frequency | Severity | Total |
| 1. Worried | | , | |
| 2. Nervous | | | |
| Panic or anxiety attacks | | | |
| 4. Social phobia | | | |
| Anxiety Subscale Total | | | |
| Anxiety Subscale Total | Fraguanay | Soverity | Total |
| Anxiety Subscale Total C. Apathy | Frequency | Severity | Total |
| Anxiety Subscale Total C. Apathy 1. Interest activities | Frequency | Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking | Frequency | Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions | Frequency | Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking | Frequency | Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total | | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis | Frequency | Severity Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena | | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions | | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations | | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations 4. Delusions | | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations | | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations 4. Delusions | | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations 4. Delusions | Frequency | | |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations 4. Delusions Psychosis Subscale Total | Frequency | Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations 4. Delusions Psychosis Subscale Total E. Impulse Control and Related Disorders | Frequency | Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations 4. Delusions Psychosis Subscale Total E. Impulse Control and Related Disorders 1. Impulse control disorders 2. Other compulsive behaviors | Frequency | Severity | Total |
| C. Apathy 1. Interest activities 2. Interest talking 3. Emotions Apathy Subscale Total D. Psychosis 1. Passage or presence phenomena 2. Illusions 3. Hallucinations 4. Delusions Psychosis Subscale Total E. Impulse Control and Related Disorders 1. Impulse control disorders | Frequency | Severity | Total |

| atient Name/Identifier: | Date: | | |
|----------------------------------|------------|----------|-------|
| F. Cognition | Frequency | Severity | Total |
| 1. Remembering | , | , | |
| Learning new information | | | |
| Focus or attention | | | |
| 4. Find words or express ideas | | | |
| 5. Executive abilities | | | |
| 6. Visuospatial abilities | | | |
| Cognition Subscale Total | | | |
| Cognition Cabboald Total | | | |
| G. Orthostatic Hypotension | Frequency | Severity | Total |
| Lightheaded or fainted | rrequericy | Severity | Total |
| 2. Dizziness or weakness | | | |
| Orthostatic Hypotension Subscale | Total | | |
| Orthostatic hypotension Subscale | lotai | | |
| H. Urinary | Frequency | Severity | Total |
| 1. Urinary urgency | , | | |
| 2. Urinary frequency | | | |
| 3. Nocturia | | | |
| Urinary Subscale Total | | | |
| I. Sexual | Frequency | Severity | Total |
| Sex drive or interest | | • | |
| 2. Sexual arousal or performance | | | |
| Sexual Subscale Total | | | |
| J. Gastrointestinal | Frequency | Severity | Total |
| 1. Drooling | | | |
| 2. Swallowing | | | |
| 3. Nausea or sick in stomach | | | |
| 4. Constipation | | | |
| Gastrointestinal Subscale Total | • | | |
| K. Sleep and Wakefulness | Frequency | Severity | Total |
| 1. Insomnia | | | |
| 2. REM sleep behavior | | | |
| Dozing off | | | |
| Dozing off Restlessness | | | |
| 4. Restlessness | | | |

| ttient Name/Identifier: | Date: | | |
|---|---|---|---|
| L. Pain | Frequency | Severity | Total |
| 1. Muscle, joint, back pain | | • | |
| 2. Deep or dull pain | | | |
| 3. Dystonia | | | |
| . Other pain | | | |
| ain Subscale Total | | | |
| Л. Other | Fraguanay | Coverity | Total |
| | Frequency | Severity | Total |
| Weight loss Decreased smell | | | |
| 3. Physical fatigue | | | |
| 4. Mental fatigue | | | |
| 5. Excessive sweating | | | |
| Other Subscale Total | | | |
| IDS-NMS TOTAL SCORE | | | |
| MDS-NMS Score St | heet – Non Motor Fluc | tuations | |
| Subscore "Change" = S | me spent in non-motor | ange" items<br>"Off" state | pre "Time" |
| Subscore "Change" = S<br>Subscore "Time" = Ti | Sum of all "degree of cha<br>ime spent in non-motor | ange" items<br>"Off" state | egree of<br>m "On" to |
| Subscore "Change" = S<br>Subscore "Time" = Ti<br>MDS-NMS NMF Total Score = Sub<br>NON-MOTOR FLUCTUATIONS<br>optional) | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression 2. Anxiety | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression 2. Anxiety 3. Thinking or cognitive abilities 4. Bladder symptoms | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression 2. Anxiety 3. Thinking or cognitive abilities | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression 2. Anxiety 3. Thinking or cognitive abilities 4. Bladder symptoms 5. Restlessness 6. Pain 7. Fatigue | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression 2. Anxiety 3. Thinking or cognitive abilities 4. Bladder symptoms 5. Restlessness 6. Pain 7. Fatigue | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression 2. Anxiety 3. Thinking or cognitive abilities 4. Bladder symptoms 5. Restlessness 6. Pain | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |
| Subscore "Change" = S Subscore "Time" = Ti MDS-NMS NMF Total Score = Sub NON-MOTOR FLUCTUATIONS (optional) 1. Depression 2. Anxiety 3. Thinking or cognitive abilities 4. Bladder symptoms 5. Restlessness 6. Pain 7. Fatigue 8. Excessive sweating | Sum of all "degree of cha<br>ime spent in non-motor | ange" items "Off" state ied by Subsco Typical de change from | egree of<br>m "On" to |

# International Parkinson and Movement Disorder Society – Non-Motor Rating Scale (MDS-NMS)

#### **Glossary of Terms**

- A. Depression: a mood disorder characterized by sustained change in emotions (sadness, decreased interest or pleasure), cognition (negative thoughts about life or self, such as hopelessness, helplessness, indecisiveness, or death or suicide ideation) or behavior (isolative, withdrawn, sleep disturbances, appetite disturbances)
- **B.** Anxiety: an affective disorder characterized by sustained excessive worrying which can be (1) generalized and include symptoms such as restlessness, being easily fatigued, mind going blank or trouble concentrating, irritability, and muscle tension; (2) specific anxiety or panic attacks; (3) fear of being in public (agoraphobia); or (4) fear of being in social situations (social phobia)
  - Anxiety or panic attack: an abrupt surge of intense fear or intense discomfort, can include shortness of breath, heart beating fast, upset stomach, sweating, dizziness or faintness, sensation of chill or heat, or sense something bad is going to happen or even a sense of dying
- C. Apathy: a disorder characterized by decreased motor activity (less initiation of motor activity not due to parkinsonism), emotional expression (less emotional engagement separate from decreased facial expression due to parkinsonism), or speech (less likely to initiate or engage in conversation)
- D. Psychosis: a disorder characterized by changes in perception (passage or presence phenomena, illusions, or hallucinations) or thought (delusions)

Passage phenomenon: visual sensation of something moving in periphery of visual field Presence phenomenon: visual sensation of person being in periphery of visual field Illusions: visual misinterpretation of an actual object

Hallucinations: a sensory (visual, auditory, taste, smell, or feeling) experience that is not real or experienced by other people

**Delusions**: a belief that something is true for which there is no objective evidence and which other persons do not hold true

- E. Impulse control disorders: a failure to resist an impulse or drive that leads to repeated engagement in activities that become harmful to self or others; compared with pre-PD behavior Hoarding: the needless collection of objects and an inability to get rid of them Punding: the needless or purposeless repetition of a simple motor activity Dopamine dysregulation syndrome: taking an excess (beyond what is prescribed) of
  - **Dopamine dysregulation syndrome**: taking an excess (beyond what is prescribed) of Parkinson's disease medications for their motor or psychological effects, often with significant mood changes during "on" (irritability, hypomania) or "off" (dysphoria) states
- F. Cognition: the activities of thinking, understanding, learning, and remembering Attention: concentrating on one part of the environment while ignoring other things Executive abilities: cognitive processes involved in maintaining multiple pieces of information in the mind at the same time, reasoning, task flexibility, problem solving, and task planning and execution.

Visuospatial abilities: ability relating to visual perception of spatial relationships among objects

Copyright @ 2019 International Parkinson and Movement Disorder Society. All rights reserved. | Version 1.0

# International Parkinson and Movement Disorder Society – Non-Motor Rating Scale (MDS-NMS)

G. Orthostatic hypotension: a drop in blood pressure severe enough to cause symptoms when changing from sitting to standing position or from lying to sitting position

#### H. Urinary

Nocturia: excessive urination at night, defined as more than 2 times overnight

#### Sexual

**Erectile dysfunction**: inability of a man to maintain an erection sufficient for satisfying sexual activity

J. Gastrointestinal: relating to the stomach and intestines

Saliva: watery liquid secreted into the mouth by glands, providing lubrication for chewing and swallowing, and aiding digestion

Swallowing: difficulty swallowing including liquids and solids, as well as choking while swallowing

Nausea: a feeling of sickness with a tendency to vomit

**Constipation**: infrequent bowel movements (usually less than three bowel movements per week) or difficult passage of stools

#### K. Sleep and wakefulness

Insomnia: difficultly falling asleep or staying asleep

Rapid eye movement (REM) sleep: a stage in the normal sleep cycle during which dreams occur and the body undergoes marked changes including rapid eye movement, loss of reflexes, and increased pulse rate and brain activity

#### L. Pain

**Dystonia**: a state of abnormal muscle tone resulting in muscular spasm and abnormal posture **Nocturnal pain**: pain overnight

Orofacial pain: pain which is felt in the mouth, jaws, or face

#### M. Other

Olfaction: the action or capacity of smelling

Fatigue (physical): state of excessive physical weariness or exhaustion (after physical exertion), different from sleepiness

Fatigue (mental): state of excessive mental weariness or exhaustion, different from sleepiness

Copyright © 2019 International Parkinson and Movement Disorder Society. All rights reserved. | Version 1.0

## 4 MODIFIED GIDS-PD

# The Gastrointenstinal Dysfunction Scale for Parkinson's Disease modified\*

The following version of GIDS-PD has been modified by permission and license from MDS for use in the N-DOSE trial. The modifications in this version is that the timeframe for all questions has been reduced from six months to one month. Part 1b has also been omitted from the scale.



# GIDS-PD modified\*

The Gastrointestinal Dysfunction Scale for Parkinson's Disease

\*by permission and license from MDS for use in the N-DOSE trial.

Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

Modified by: Haakon Berven NeuroSysMed, Haukeland University Hospital Bergen, Norway Authored by: Marta Camacho Julia C. Greenland Caroline H. Williams-Gray

Tel +1 (414) 276-2145 Fax +1 (414) 276-3349 555 E. Wells Street, Suite 1100 Milwaukee, WI 53202-3823 www.movementdisorders.org ratingscales@movementdisorders.org

Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

# GIDS-PD modified\*

# THE GASTROINTESTINAL DYSFUNCTION SCALE IN PARKINSON'S DISEASE

\*by permission and license from MDS for use in the N-DOSE trial.

Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

#### INSTRUCTIONS

Some patients with Parkinson's disease experience changes in their digestive system. This questionnaire assesses whether you have experienced any gut problems. Tick the statement that best describes your symptoms over the <code>past month</code> . Be sure to read all the statements in each item.

If you have had the problem in the past but have not experienced the problem in the past month , please tick 'No'.

If you have used medication in the past month related to any of the following problems, answer about your experience while taking the medication.

Please answer every question. If you are uncertain about how to answer a question tick the statement that best describes your symptoms.

Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

| NAME (CTUDY CODE. | T/ | DD AVIIC DATE: | CEV. | 4.05: |
|---|---|---|---|---|
| NAME/STUDY CODE: | 10 | DDAY'S DATE: | SEX: | AGE: |
| | | | OF OM | |
| 1. Over the past month, how often, | , on average, did you pass | stool? | | |
| Frequency: | | | | |
| Occasionally: 3 times a week or less | S. | | | |
| Often: 4 to 7 times a week. | | | | |
| Frequently: 8 or more times a week | τ. | | | |
| Severity: | | | | |
| Mild: frequency of stool passing lea | ds to little or no discomfort ( | or distress. | | |
| Moderate: frequency of stool passin to manage it are needed. | ng leads to discomfort or is d | lisruptive, but r | no extra effor | ts |
| Severe: frequency of stool passing causing pain or anxiety or efforts to | | | | on). |
| 1a. Over the past (month, have you tak | en specific measures to have | e more bowel | movements? | |
| Yes No | | | | |
| If Yes, tick all that apply: | | | | |
| I have eaten more fibre (for exampl or consumed probiotics. | e, eating more prunes, cereal | ls, fibrous soup | ) | |
| I have used laxatives occasionally (to a compare to the compa | twice a week or less). | | | |
| I have used laxatives regularly (mor | e than twice a week but not | every day). | | |
| I have used laxatives daily. | | | | |
| • | | | | |

| 2. Ov | ver the past month, have you experienced straining (difficulty passing stool, finding it |
|---|---|
| pa | inful to pass stool)? |
| | Yes No |
| If Ye | uency: |
| $\bigcirc$ | Occasionally: once every 10 times I go to the toilet, or less. |
| 0 | Often: on average, once every 4 times I go to the toilet. |
| $\bigcirc$ | Frequently: at least one in every 2 times I go to the toilet. |
| Seve | erity: |
| 0 | Mild: straining is present but leads to little or no discomfort or distress. |
| | <b>Moderate:</b> straining leads to discomfort or is disruptive (for example, it delays stool passing, takes increased effort to pass stool, or you have piles because of straining). |
| 0 | Severe: straining leads to severe discomfort, distress or is very disruptive, causing pain or anxiety or efforts to manage it have to be employed (for example, you had to press on or around your |
| 3 Ov | bottom, remove stool with your hands, or have enemas). |
| | bottom, remove stool with your hands, or have enemas). Ver the past month , have you experienced hard stools? Yes No |
| If Ye | ver the past month , have you experienced hard stools? Yes No |
| If Ye | ver the past month , have you experienced hard stools? Yes No |
| If Ye | ver the past month , have you experienced hard stools? Yes No |
| If Ye | Yes No No No Occasionally: once every 10 times I go to the toilet, or less. |
| If Ye Fred | Yes No No No Occasionally: once every 10 times I go to the toilet, or less. Often: on average, once every 4 times I go to the toilet. |
| If Ye Fred | Ver the past month , have you experienced hard stools? Yes No No No Occasionally: once every 10 times I go to the toilet, or less. Often: on average, once every 4 times I go to the toilet. Frequently: at least once in every 2 times I go to the toilet. |
| If Ye Fred | Ver the past month , have you experienced hard stools? Yes No No No Occasionally: once every 10 times I go to the toilet, or less. Often: on average, once every 4 times I go to the toilet. Frequently: at least once in every 2 times I go to the toilet. erity: |
| If Ye Fred | Yes No |

GIDS-PD\* | THE GASTROINTESTINAL DYSFUNCTION SCALE IN PARKINSON'S DISEASE \*modified 4. Over the past month, have you experienced a sensation of incomplete evacuation? Yes No If Yes, Frequency: Occasionally: once every 10 times I go to the toilet, or less. Often: on average, once every 4 times I go to the toilet. Frequently: at least once in every 2 times I go to the toilet. Severity: Mild: sensation of incomplete evacuation is present but leads to little or no discomfort or distress. Moderate: sensation of incomplete evacuation leads to discomfort or is disruptive (delaying passing of stool). Severe: sensation of incomplete evacuation leads to severe discomfort, distress or is very disruptive, causing pain or anxiety or efforts to manage it have to be employed (for example, prompting several attempts to pass stool on that day). 5. Over the past month, have you experienced abdominal pain? Yes No If Yes. Frequency: Occasionally: less than once a week. Often: on average, once a week. Frequently: at least twice a week. Severity: Mild: abdominal pain is present but leads to little or no discomfort or distress. Moderate: abdominal pain leads to discomfort or is disruptive. Severe: abdominal pain leads to severe discomfort, distress or is very disruptive and stops you from doing your activities. PLEASE CHECK THAT YOU ANSWERED ALL THE QUESTIONS CONTINUE TO NEXT PAGE > Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

04/09 GIDS-PD\*| THE GASTROINTESTINAL DYSFUNCTION SCALE IN PARKINSON'S DISEASE 6. Over the past month, have you experienced days in which you have had an abnormal increase in stool passing? If you experienced constipation on some days but you also experienced increased frequency of stool passing, please tick yes. Yes No If Yes. Frequency: Occasionally: less than once a week, I have needed to pass a stool more often than usual. Often: on average, once a week, I have needed to pass a stool more often than usual. Frequently: at least twice a week, I have needed to pass a stool more often than usual. Severity: Mild: increased frequency of stool passing is present but leads to little or no discomfort or distress. Moderate: increased frequency of stool passing leads to discomfort or is disruptive. Severe: increased frequency of stool passing leads to severe discomfort, distress or is very disruptive and stops you from doing your activities (for example, faecal incontinence). 7. Over the past month, have you experienced abdominal fullness, pressure, or a sensation of trapped gas, feeling bloated or distension (visible increase in abdominal girth)? If Yes, Frequency: Occasionally: less than once a week Often: on average, once a week. Frequently: at least twice a week. Severity: Mild: recurrent abdominal fullness is present but leads to little or no discomfort or distress. Moderate: recurrent abdominal fullness leads to discomfort or is disruptive (for example, feeling excessively full after regular-sized meals). Severe: recurrent abdominal fullness leads to severe discomfort, distress or is very disruptive and stops you from doing your activities or eating plentiful meals. PLEASE CHECK THAT YOU ANSWERED ALL THE QUESTIONS CONTINUE TO NEXT PAGE Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

| *n | $\overset{ullet}{D}$ THE GASTROINTESTINAL DYSFUNCTION SCALE IN PARKINSON'S DISEASE modified |
|---|---|
| Even if yo | he past month, have you experienced involuntary weight loss? but have lost weight over the course of several months and maintained this loss over month, please tick yes. |
| Yes | ○ No |
| If Yes,<br>Quantity: | |
| Less | s than 10% of my body weight. |
| On a | average, 10% of my body weight. |
| O Mor | re than 10% of my body weight. |
| Severity: | |
| Mild | d: weight loss is present but leads to little or no discomfort or distress. |
| O Mod | derate: weight loss leads to discomfort or is disruptive. |
| Sev | ere: weight loss leads to severe discomfort, distress or is very disruptive (for example, you |
| | e to take nutritional supplements or appetite stimulants to manage it, or it causes frailty). the past month, have you experienced difficulty swallowing or did food or drinks |
| 9. Over th | |
| 9. Over th | he past month, have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? |
| 9. Over the get stuck Yes If Yes, Frequence | he past month, have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? |
| 9. Over the get stuck Yes If Yes, Frequence | he past month, have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? No |
| 9. Over the get stuck Yes If Yes, Frequence Occo | the past month, have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? No No Residually: less than once a week. |
| 9. Over the get stuck Yes If Yes, Frequence Occo | the past month , have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? No No Ey: casionally: less than once a week. en: on average, once a week. quently: at least twice a week. |
| 9. Over the get stuck Yes If Yes, Frequence Occo Ofte Free Severity: | the past month , have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? No No Ey: casionally: less than once a week. en: on average, once a week. quently: at least twice a week. |
| 9. Over the get stuck Yes If Yes, Frequence Occo Office Free Severity: Mild | the past month , have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? No No Residually: less than once a week. Pen: on average, once a week. Requently: at least twice a week. |
| 9. Over the get stuck Yes If Yes, Frequence Occo Ofte Free Severity: Mild Moc food Severity | the past month , have you experienced difficulty swallowing or did food or drinks in your throat after swallowing or go down slowly through your chest? No No Ry: Rasionally: less than once a week. Ren: on average, once a week. Rquently: at least twice a week. Rd: difficulty swallowing is present but leads to little or no discomfort or distress. Release: difficulty swallowing leads to discomfort or is disruptive (for example, you cut your |

GIDS-PD\*| THE GASTROINTESTINAL DYSFUNCTION SCALE IN PARKINSON'S DISEASE \*modified 10. Over the past month, have you experienced excessive saliva? Yes No If Yes, Frequency: Occasionally: less than once a week. Often: on average, once a week. Frequently: at least twice a week. Severity: Mild: excessive saliva is present but leads to little or no discomfort or distress. Moderate: excessive saliva leads to discomfort or is disruptive (for example, it causes drooling). Severe: excessive saliva leads to severe discomfort, distress or is very disruptive (for example, you have to take medication to manage it, you have to keep cleaning yourself or it causes embarrassment). 11. Over the past month, have you experienced heartburn? If Yes, Frequency: Occasionally: less than once a week. Often: on average, once a week. Frequently: at least twice a week. Mild: heartburn is present but leads to little or no discomfort or distress. Moderate: heartburn leads to discomfort or is disruptive (for example, you need to take medication to manage it). Severe: heartburn leads to severe discomfort, distress or is very disruptive (for example, you have trouble doing things or falling asleep). PLEASE CHECK THAT YOU ANSWERED ALL THE QUESTIONS Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

| | the past month, have you experienced nausea? |
|---|---|
| O Yes | ○ No |
| If Yes,<br>Frequency | :y: |
| Occa | casionally: less than once a week. |
| Ofte | en: on average, once a week. |
| Freq | quently: at least twice a week. |
| Severity: | |
| Mild | d: nausea is present but leads to little or no discomfort or distress. |
| ( ) | derate: nausea leads to discomfort or is disruptive (for example, you need to take anti-sickness dication to manage it or it affects your appetite). |
| | ere: nausea leads to severe discomfort, distress or is very disruptive (for example, it keeps you m doing things or it makes you vomit). |

# GIDS-PD\*| THE GASTROINTESTINAL DYSFUNCTION SCALE IN PARKINSON'S DISEASE

We would also like to ask you some important questions about your lifestyle that may contribute

| OVE | R THE <u>LAST MONTH</u> : |
|---|---|
| A. V | hich diet best represents most of your meals? |
| $\bigcirc$ | Western Diet (rich in meat and roasted potatoes/vegetables) |
| $\bigcirc$ | Mediterranean Diet (rich in meat, fish, fresh vegetables and fresh fruits) |
| $\bigcirc$ | Asian Diet (rich in noodles, rice and cooked vegetables) |
| $\bigcirc$ | Indian Diet (rich in curry, grains and lentils) |
| $\bigcirc$ | Vegetarian/Vegan (excluding meat or animal derived products from meals) |
| $\bigcirc$ | Mixed diet (you do not follow a particular diet pattern, or your diet is a mixture of some of the above) |
| в. о | n average, how many glasses of water or non-fizzy juice did you drink per day? |
| | Less than 1 glass a day (a few per week) |
| | 1-3 glasses a day |
| $\bigcirc$ | More than 3 glasses a day |
| C. H | ow many caffeinated drinks (for example, coffee, tea and energy drinks) did you have per day? |
| 0 | Less than 1 glass a day (a few per week) |
| | 1-3 glasses a day |
| | More than 3 glasses a day |
| | ow many times did you exercise for more than 30 minutes (for example, fitness classes, c walking or cycling for at least 30 minutes)? |
| $\bigcirc$ | Less than once a week |
| $\bigcirc$ | 1 to 3 exercise sessions a week |
| $\bigcirc$ | More than 3 exercise sessions a week |
| | PLEASE CHECK THAT YOU ANSWERED ALL THE QUESTIONS |

| I have never smoked I am an ex-smoker I currently smoke (daily or occasionally) F. Have you EVER been diagnosed with any of the following gastrointestinal disorders by a medical doctor? | |
|---|---|
| I currently smoke (daily or occasionally) F. Have you EVER been diagnosed with any of the following gastrointestinal disorders by | |
| F. Have you EVER been diagnosed with any of the following gastrointestinal disorders by | |
| DISORDER YES NO IF YES, CURRENTLY TO MEDICATION F | |
| Constipation Yes | ) N |
| Irritable bowel syndrome (IBS) | ) No |
| Crohn's Disease Yes | ) No |
| Gastroesophageal reflux (also known as Heartburn) | ) No |
| Ulcerative Colitis Yes | ) No |
| Diverticular Disease Yes | ) No |
| Colon Cancer Yes | ) No |
| Other: | ) No |

APPENDIX I SCORING INSTRUCTIONS

 $\begin{array}{l} \textbf{GIDS-PD}^*| \text{ THE GASTROINTESTINAL DYSFUNCTION SCALE IN PARKINSON'S DISEASE} \\ ^* \text{modified} \end{array}$ 

#### SCORING INSTRUCTIONS

Items 1 through 12 are scored as follows: (except for Item 1-frequency which is inverted)

The GIDS-PD\*can be divided into 3 subscores, each constituted by a set of items:

| SEVERITY |
|-------------|
| Mild: 1 |
| Moderate: 2 |
| Severe: 3 |

| SUBSCORES | ITEMS |
|--------------------|------------------|
| Constipation | 1, 2, 3 and 4 |
| Bowel Irritability | 5, 6, 7 and 8 |
| Upper GI | 9, 10, 11 and 12 |

Items 1a, A, B, C, D, E and F provide additional information but are **not used for scoring**. The total score for each item is computed by multiplying frequency and severity scores.

The total score of the GIDS-PD\* is computed by adding the total scores of items 1 through 12, resulting in a minimum score of 1 and a maximum score of 108.

| ITEM | FREQU | JENCY S | SCORE | SEVE | RITY S | CORE | TOTAL ITEM SCORE (F X S) | |
|---|---|---|---|---|---|---|---|---|
| 1 | 3 | 2 | 1 | 1 | 2 | 3 | Z | |
| 2 | 1 | 2 | 3 | 1 | 2 | 3 | + PATIC | |
| 3 | 1 | 2 | 3 | 1 | 2 | 3 | + NSTE | CONSTIPATION<br>SUBSCORE |
| 4 | 1 | 2 | 3 | 1 | 2 | 3 | + | |
| 5 | 1 | 2 | 3 | 1 | 2 | 3 | + | BOWEL<br>IRRITABILITY<br>SUBSCORE |
| 6 | 1 | 2 | 3 | 1 | 2 | 3 | + VEL | |
| 7 | 1 | 2 | 3 | 1 | 2 | 3 | + BOV | |
| 8 | 1 | 2 | 3 | 1 | 2 | 3 | + $\overline{\alpha}_0$ | ) |
| 9 | 1 | 2 | 3 | 1 | 2 | 3 | + | |
| 10 | 1 | 2 | 3 | 1 | 2 | 3 | + + | UPPER GI<br>SUBSCORE |
| 11 | 1 | 2 | 3 | 1 | 2 | 3 | + A Page 1 | |
| 12 | 1 | 2 | 3 | 1 | 2 | 3 | + | |
| | | TOTAL ( | GIDS-PD | SCORE | | | = | |

\*modified

Copyright © 2022 International Parkinson and Movement Disorder Society (MDS). All Rights Reserved. Adapted and used with permission of MDS. This derivative of the GIDS-PD has not been validated or tested for reliability.

# 5 MOCA

# **Montreal Cognitive Assessment**

MoCA tests were alternated to avoid learning effects. The sequence of versions for testing for each participant is listed in the table below:

| Visit | Version |
|-------------|--------------------------------|
| 1 (Week 0) | Version 8.3 Norwegian version |
| 2 (Week 4) | Version v8.1 Norwegian version |
| 3 (Week 8) | Version V8.2 Norwegian version |
| 4 (week 12) | Version v8.3 Norwegian version |

# MocA – Version 8.1 Norwegian version

| MONTREAL COGNITIVE ASSESSMENT (MOCA)<br>Version 8.1 Norwegian version | Utdanning | Navn:<br>(i år):<br>(jønn: | Fødselsdato:<br>DATO: | |
|---|---|---|---|---|
| S Slutt B 2 D 4 3 | Kopier<br>kube<br>(1 poeng) | (3 poeng) | e (ti over elleve) | POENG |
| © [1] | [ ] | [ ]<br>Kontur | [ ] [ ]<br>Tall Viser | |
| HUKOMMELSE Les ordene, deltageren må gjenta dem. Gjør to forsøk, selv om første forsøk gjennomføres helt riktig. Gjør gjenkalling etter 5 minutter. 1. fors 2. fors | øk | LØYEL KIRKE | TUSENFRYD RG | /3 D INGEN POENG |
| OPPMERKSOMHET Les rekken med tall (1 tall/sekund). Delt | ageren skal gjenta dem i<br>ageren skal gjenta dem i | | []21854 | 4 /2 |
| Les listen med bokstaver. På hver bokstav A skal deltageren banke på b | ordet med hånden sin. Ir | ngen poeng ved ≥ 2 fei | | /1 |
| Begynn fra 100 og trekk fra 7 flere ganger etter hverandre. [ ] 93 4 eller 5 riktige subtraksjoner: 3 poeng, SPRÅK Gjenta: Gjenta etter meg: Det eneste jeg vet | [ ] 86 | 72 [ ] 65<br>peng, 1 riktig: 1 po | | /3 |
| Katten gjemte seg alltid under sofaen når det v<br>Ordflyt: Si så mange ord du kan komme på som begynner n | | []<br>:tt <u>.</u> [] | (N ≥ 11 ord) | /2 |
| ABSTRAKSJON Likheten mellom for eksempel en banan og en | | | [ ] klokke - linjal | /2 |
| UTSATT GJENKALLING (MIS) Hukommelse- x3 indeks-skåre x2 (MIS) X1 Flere valg som stikkord ANSIKT ANSIKT [] | FLØYEL KIRKE | TUSENFRYD RØ | UIEN | /5 |
| | ]År []Uked | ag []Ste | d [ ] By | /6 |
| © Z. Nasreddine MD www.mocatest.org Administrert av: Opplæring og sertifisering er nødvendig for å sikre nøyaktigh | MIS: | /15<br>(Normal ≥ 26/30)<br>ersom ≤12 års utdanning | TOTAL CHÂDE | /30 |

133

#### MocA - Version 8.2 Norwegian version



#### MocA - Version 8.3 Norwegian version



# 6 EQ-5D-EL

The 5-level EQ-5D

**EQ-5D-5L – Page 1** 



Spørreskjema om helse

Norsk versjon, for Norge

(Norwegian version for Norway)

# EQ-5D-5L – Page 2

| GANGE | |
|---|---|
| Jeg har ingen problemer med å gå omkring | П |
| Jeg har litt problemer med å gå omkring | |
| Jeg har middels store problemer med å gå omkring | |
| Jeg har store problemer med å gå omkring | |
| Jeg er ute av stand til å gå omkring | |
| PERSONLIG STELL | |
| Jeg har ingen problemer med å vaske meg eller kle meg | |
| Jeg har litt problemer med å vaske meg eller kle meg | |
| Jeg har middels store problemer med å vaske meg eller kle meg | |
| Jeg har store problemer med å vaske meg eller kle meg | |
| Jeg er ute av stand til å vaske meg eller kle meg | |
| VANLIGE GJØREMÅL (f.eks. arbeid, studier, husarbeid, familie- el fritidsaktiviteter) | ller |
| Jeg har ingen problemer med å utføre mine vanlige gjøremål | |
| Jeg har litt problemer med å utføre mine vanlige gjøremål | |
| Jeg har middels store problemer med å utføre mine vanlige gjøremå | ål 🗖 |
| Jeg har store problemer med å utføre mine vanlige gjøremål | |
| Jeg er ute av stand til å utføre mine vanlige gjøremål | |
| SMERTER / UBEHAG | |
| Jeg har verken smerter eller ubehag | |
| Jeg har litt smerter eller ubehag | |
| Jeg har middels sterke smerter eller ubehag | |
| Jeg har sterke smerter eller ubehag | |
| Jeg har svært sterke smerter eller ubehag | |
| ANGST / DEPRESJON | |
| Jeg er verken engstelig eller deprimert | |
| Jeg er litt engstelig eller deprimert | |
| Jeg er middels engstelig eller deprimert | |
| Jeg er svært engstelig eller deprimert | |
| Jeg er ekstremt engstelig eller deprimert | |

## **EQ-5D-5L – Page 3**

- Vi vil gjerne vite hvor god eller dårlig helsen din er I DAG.
- Denne skalaen er nummerert fra 0 til 100.
- 100 betyr den <u>beste</u> helsen du kan tenke deg.
   0 betyr den <u>dårligste</u> helsen du kan tenke deg.
- Sett en X på skalaen for å angi hvordan helsen din er I DAG.
- Skriv deretter tallet du merket av på skalaen inn i boksen nedenfor.

HELSEN DIN I DAG =



3

Norway (Norwegian) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group